# STATISTICAL ANALYSIS PLAN

BHR-100-301

A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study to Investigate the Efficacy and Safety of Progesterone in Patients with Severe Traumatic Brain Injury

# Prepared for:

BHR Pharma, LLC

#### **Version and Author details:**

Version Date: 19APR2014

Version Number 2.0

Author:

# **SIGNATURES**

The undersigned have approved this Statistical Analysis Plan for use in this study.

| Date |
|------|
| Date |
| Date |



# **TABLE OF CONTENTS**

| 1 | INT | RODUCTION | 5 |
|---|---|---|---|
| | 1.1 | Changes from the protocol | 5 |
| 2 | STU | DY OBJECTIVES | 5 |
| 3 | STUI | DY DESIGN | 5 |
| | 3.1 | Sample Size Considerations | |
| | 3.2 | Randomization | |
| 4 | STUI | DY VARIABLES AND COVARIATES | 8 |
| • | 4.1 | Primary Outcome Variable | |
| | 4.2 | Secondary Outcome Variables | |
| | 4.2 | 2.1 Efficacy | |
| | | 2.2 Safety | |
| | 4.3 | Predetermined Covariates and Prognostic Factors | 8 |
| 5 | DEF: | INITIONS | 9 |
| 6 | ANA | LYSIS SETS | 13 |
| | 6.1 | Modified Intention-to-Treat | 13 |
| | 6.2 | Per Protocol | |
| | 6.3 | Safety | 14 |
| 7 | INTE | ERIM ANALYSIS | 14 |
| 8 | DAT | A REVIEW | 16 |
| • | 8.1 | Data Handling and Transfer | |
| | 8.2 | Data Screening | |
| 9 | STAT | TISTICAL METHODS | 17 |
| | 9.1 | Subject Disposition | |
| | 9.2 | Protocol Deviations and Violations | |
| | 9.3 | Treatments | |
| | 9.3 | | |
| | | 3.2 Concomitant Medications, Concomitant Procedures and Surgical Therapy | |
| | 9.4<br>9.5 | Demographic and Baseline Characteristics Efficacy Analyses | |
| | 9.5 | , , | |
| | | 0.5.1.1 Proportional Odds Model | 20 |
| | | 0.5.1.2 Alternate Primary Efficacy Analysis (Sliding Dichotomy) | |
| | | 0.5.1.3 Sensitivity Analysis (Dichotomized Model) | |
| | | 9.5.1.4 Interpretation of Statistical Significance of Primary Efficacy Analysis 9.5.1.5 Handling of Missing Data | |
| | | 9.5.1.6 Exploratory Analysis | |
| | 9.5 | | |
| | | 0.5.2.1 Mortality at Month 1, Month 6 | 27 |
| | | 0.5.2.2 GOS at Month 3 | |
| | | 0.5.2.3 GOS-E at Month 3 and Month 6 | |
| | 9.5 | - · | |
| | | 0.5.3.1 Time to Death | |





 $a_{rac{}{ ext{Version Date: 2.0 April 19, 2014}}}$ 

| 9.5.3.2 Comparison of CT scans at admission and Day 6 | 30 |
|---|---|
| 9.5.3.3 ICP | 30 |
| 9.5.3.4 CPP | |
| 9.5.3.5 TIL | |
| 9.6 Safety Analyses | |
| 9.6.1 Adverse Events | |
| 9.6.2 Neuroworsening | |
| 9.6.3 Deaths and Serious Adverse Events | |
| 9.6.4 Laboratory Data | |
| 9.6.5 Vital Signs | |
| 9.6.6 Physical Examinations, ECGs, and Other Observations Related to Safety | |
| 9.6.6.1 Arterial Blood Gases | |
| 9.6.7 Progesterone Levels | |
| 10 VALIDATION | 34 |
| 11 REFERENCES | 34 |
| APPENDIX 1 GLOSSARY OF ABBREVIATIONS | |
| APPENDIX 2 LIST OF POST-TEXT TABLES, FIGURES, LISTINGS, AND SUPPORTIVE | |
| OUTPUT APPENDICES | 38 |
| APPENDIX 3 SHELLS FOR POST-TEXT TABLES, FIGURES, AND LISTINGS | 57 |
| LISTINGS | 14 <i>/</i> |



#### 1 INTRODUCTION

This statistical analysis plan (SAP) describes the statistical methods to be used during the reporting and analysis of data collected under BHR Pharma Protocol BHR-100-301.

This SAP should be read in conjunction with the study protocol and electronic case report form (eCRF). This version of the plan has been developed using the protocol Amendment 3.0 dated November 15, 2011 and eCRF dated September 24, 2012. Changes to the SAP based on protocol and/or eCRF revisions are reflected in this final version. This version is approved prior to unblinding and analysis of the global trial

The SAP has been developed in two stages. This amendment, SAP version 2.0, is is the final version prior to the global study database lock. Versions of the SAP up to initial sponsor approval were known as SAP1. PRA and the Sponsor (BHR Pharma) have agreed on the changes from version 1.0 to enable the final programming for the Clinical Study Report (CSR) and a potential New Drug Application (NDA). This final version of the SAP, version 2.0, has been approved by PRA and the sponsor prior to database lock.

#### 1.1 Changes from the protocol

- The protocol states that the primary efficacy analysis will be conducted on all randomized subjects. BHR was advised by the Data and Safety Monitoring Board and the Steering Committee to redefine the intent-to-treat (ITT) population as all randomized subjects who received any amount of study drug treatment. This modified intent-to-treat (mITT) analysis was approved by the FDA in its Special Protocol Assessment Agreement Modification Letter dated April 4, 2013. This version of the SAP defines the mITT population, which will be used for all efficacy analyses.
- The protocol states that the Extended Glasgow Outcome Scale (GOS-E) will be analyzed using the 2-sided Wilcoxon Rank-Sum test. This version of the SAP states that the GOS-E will be analyzed similarly to the GOS, using a proportional odds model (POM) and sliding dichotomy (SD).

#### **2 STUDY OBJECTIVES**

The aim of this study is to determine the efficacy and safety of BHR-100 (intravenous (i.v.) progesterone lipid emulsion) compared to placebo infusion in the treatment of subjects with severe traumatic brain injury (TBI).

#### 3 STUDY DESIGN

This trial is a multicenter, randomized, double-blind, placebo-controlled study, conducted in approximately 140 Level I (or equivalent) trauma centers in a number of geographical areas including North America, Europe, Asia and South America, to compare the efficacy and safety of i.v. BHR-100 with placebo in the treatment of subjects following severe TBI. Severe TBI is defined as a Glasgow Coma Scale (GCS) score at randomization of 3-8 (inclusive). During their involvement in the study, subjects will be managed in accordance with standard guidelines for

the management of severe TBI (Brain Trauma Foundation, American Brain Injury Consortium, and European Brain Injury Consortium).

The planned duration of the study will be 6 months for each subject, with the study consisting of the 3 phases:

- Screening,
- Treatment, and
- Follow-up.

During the screening period, subjects will be assessed for inclusion into the study and informed consent will be obtained. Medical and medication histories, physical exam including weight and pupil response, vital signs, ECG, laboratory tests (hematology, serum chemistry, urinalysis, and coagulation) and arterial blood gases (ABG: partial pressure of oxygen in arterial blood (PaO<sub>2</sub>), partial pressure of carbon dioxide in arterial blood (PaCO<sub>2</sub>), bicarbonate (HCO<sub>3</sub>), pH, saturation of oxygen in arterial blood (SaO<sub>2</sub>), and fraction of inspired oxygen (FiO<sub>2</sub>)) will be performed prior to the initiation of study drug treatment. Intracranial pressure (ICP) and therapy intensity level (TIL) will be obtained prior to treatment initiation, if the ICP monitor is placed. Pretreatment/baseline assessment of TBI will be recorded using GCS and computed tomography (CT) scan.

Once a subject is determined to be eligible for inclusion into the study, he/she will be randomized (1:1) to receive either i.v. BHR-100 or placebo, stratified by geographic region (North America, Europe, Asia and South America) using an Interactive Web-based Randomization System (IWRS).

During the treatment period, subjects will be administered continuous i.v. infusion of BHR-100 or matching placebo for 120 hours and the GCS and neuroworsening (defined as any one of the following: a decrease in GCS motor score ≥ 2, development of pupillary abnormalities, any other neurological deterioration, or progression of lesion on CT scan leading to a change in subject management) will be assessed daily. Vital signs, ABGs, ICP, and CPP will be recorded periodically, and TIL, concomitant medications, and adverse events (AEs) will be monitored continuously.

During the follow-up period, subjects will be assessed at the following post-injury timepoints:

- Day 6,
- Day 15 (or ICU discharge),
- Day 30 (Month 1),
- Day 90 (Month 3),
- Day 180 (Month 6).

See the protocol schedule of events for further details of the efficacy and safety assessments conducted at each timepoint.

An independent Data Safety Monitoring Board (DSMB) will monitor data periodically during the course of the study and will update the sponsor. Reviews will occur at approximately



100-subject intervals. A DSMB charter and Data Monitoring and Analysis Plan (DMAP) have been written to provide further details.

There will be one interim analysis conducted when 200 subjects in each treatment group (400 subjects total) have reached a study endpoint (completed the study and been assessed for 6-month Glasgow Outcome Scale (GOS), died, or lost to follow up). At the interim analysis, stopping for efficacy will be assessed using statistical methods for group sequential testing with the O'Brien Fleming method.

Additionally, stopping the study for futility will be assessed by review of the conditional power at the interim analysis.

#### 3.1 Sample Size Considerations

The primary efficacy measurement for this study is GOS at 6 months after injury; see section 4.1.

For the purposes of the analysis and sample size calculation, the first 2 categories of the GOS (vegetative state and dead) will be combined. Based on the 6-month GOS outcome distribution from the head injury population with GCS 3-8 in the previous TBI Phase 3 trials in the International Mission for Prognosis and Analysis of Clinical Trials in TBI Project (IMPACT) Database, it is assumed that the following GOS responses will be observed at 6 months, in subjects treated with placebo: 31% good recovery, 21% moderate disability, 19% severe disability, and 29% vegetative state or dead (Lu, 2011).

A sample size of 1,180 subjects receiving study drug (590 in each treatment group) will be needed to detect a common odds ratio of 1.5, of improvement in GOS at 6 months in BHR-100 compared to placebo, at 90% power and a significance level of 0.01 (2-sided). This calculation used the sample size equation for comparing 2 groups of ordinal data using the technique of ordinal logistic regression proposed by Whitehead (1997).

# 3.2 Randomization

Subjects will be randomized to either BHR-100 or placebo on a 1:1 ratio, using an IWRS. The randomization will be stratified by geographic region of the site locations in order to avoid imbalance in the distribution of treatment groups within regions.

The following countries are planned to be involved in the study: Argentina, Austria, Belgium, China, Czech Republic, Finland, France, Germany, Hungary, Israel, Italy, Malaysia, Netherlands, Romania, Russia, Singapore, Spain, Taiwan, Thailand, United Kingdom, and United States. Additional countries may be considered.

These countries will be grouped into the following regions: North America (US), Europe (Austria, Belgium, Czech Republic, Finland, France, Germany, Hungary, Israel, Italy, Netherlands, Romania, Russia, Spain and UK), Asia (China, Malaysia, Singapore, Taiwan, and Thailand) and South America (Argentina).

#### 4 STUDY VARIABLES AND COVARIATES

#### 4.1 Primary Outcome Variable

The primary efficacy variable is the GOS at Month 6, post-injury assessment. The GOS is a 5-point scale used to assess the mortality and disability in TBI subjects and consists of the following 5 categories:

- Dead,
- Vegetative state,
- Severe disability,
- Moderate disability, and
- Good recovery.

For this study the first 2 categories of the GOS (dead and vegetative state) will be combined.

# 4.2 <u>Secondary Outcome Variables</u>

#### 4.2.1 Efficacy

The secondary efficacy parameters for this study will be as follows:

- Mortality at Months 1 and 6,
- GOS at Month 3,
- Extended Glasgow Outcome Scale (GOS-E) at Months 3 and 6,
- Quality of Life Short Form-36 Health Survey (SF-36) at Months 3 and 6.

The exploratory efficacy parameters for this study will be as follows:

- Changes in intracranial pathology as assessed by admission and Day 6 (+/- 1 day) CT scans,
- Changes in ICP, CPP, and TIL.

#### **4.2.2 Safety**

In order to determine if i.v. BHR-100 is safe and well-tolerated, the following safety variables will be summarized:

- AEs,
- Vital signs,
- Laboratory data,
- Physical examinations,
- Electrocardiogram (ECG),
- ABG, and
- Neuroworsening.

#### 4.3 <u>Predetermined Covariates and Prognostic Factors</u>

A number of predetermined prognostic covariates have been defined for consideration within this study:

- Age,
- Motor response component of GCS (1-2, 3, 4, or 5-6) used to determine eligibility,
- Pupillary response (bilateral, unilateral/no reactive pupils/not testable) used to determine eligibility,
- Presence of hypoxia (yes/suspected, no/unknown) any time prior to randomization,
- Presence of hypotension (yes/suspected, no/unknown) any time prior to randomization,
- CT result at baseline (Marshall's CT Classification I/II, III, IV, or evacuated/non-evacuated mass lesion),
- Presence of traumatic subarachnoid hemorrhage (yes, no), and
- Region (North America, Europe, Asia, South America).

All covariates will be measured at baseline, prior to randomization.

Randomization is expected to balance covariates amongst the treatment groups; consequently, no formal testing of baseline comparability will be conducted.

#### **5 DEFINITIONS**

# Baseline and Change from Baseline, Repeated Observations

The baseline value for each assessment is defined as the last measurement taken prior to randomization.

For any parameter at a specific visit, change from baseline is calculated as the value of that parameter at that visit minus the baseline value of that parameter, as defined above.

For data with repeated observations at a given visit, for example, vital signs, the first collected value will be used in summaries, with repeat values being included in the data listings only.

#### **Endpoint Completer**

A subject is considered an endpoint completer if they provide a GOS assessment at Month 6 or die before Month 6.

#### Study Completer

A subject is considered a study completer if they complete a 6 month assessment.

#### Duration of study drug exposure (in hours)

The duration of study drug exposure (in hours) = date:hour of last study medication administered – date:hour of first study medication administered – sum of recorded durations of infusion rate interruptions.

Please note, date:hour is used since both the date and time of medication administration is recorded in the CRF. Only interruptions greater than 30 minutes are recorded on the eCRF and will be accounted for in the duration of study drug exposure derivation.

#### Total Dose (in mg/kg)

The total dose in mg for each study drug administration record will be calculated as:

Infusion rate from eCRF (ml/hr) \* total duration of study drug administration record (hr) \* 2 (mg/ml).

The total dose in mg will be summed across all study drug administration records for a subject and then divided by the weight in kg (from IWRS).

#### Relative Dose

The relative dose for a subject will be the total dose received in mg/kg divided by the total protocol expected dose of 60.21 mg/kg. Relative dose will only be summarized for subjects who receive study drug for 120 hours +/- 5%, i.e. 114-126 hours.

# Study Medication Compliance (%)

The study medication percent compliance will be calculated as:

Number of hours of medication taken, as outlined in the protocol x 100 120 (intended duration of medication intake)

Primary Endpoint: GOS at Month 6 assessment (6 months after injury), missing data imputation

When the primary efficacy endpoint is missing, the last observation carried forward (LOCF) principle will be used to populate the primary endpoint, i.e. the Month 3 GOS assessment will be carried forward. In the event that a subject is lost to follow-up and has neither the 3 nor the 6-month GOS, the missing values will be imputed based upon the primary proportional odds model (POM).

To obtain values for the missing responses using the POM the predicted response probabilities will be used. Specifying the PREDICTED option on the OUTPUT statement of PROC LOGISTIC, 3 (number of categories in response variable -1) predicted probabilities will be provided for each subject; these are the ordered cumulative probability of each response category, i.e.

Probability( $Y \le 1$ )=P(Y=1)=Probability GOS=1  $P(Y \le 2)$ =Probability that GOS is 1 or 2  $P(Y \le 3)$ =Probability that GOS is 1, 2 or 3

Therefore, to obtain the predicted probability of each individual response, for example, the probability that the response was GOS=2, the following calculation is performed:

$$P(Y=2)=P(Y\leq 2)-P(Y=1)$$
  
Similarly,

 $P(Y=3)=P(Y\le 3)-P(Y\le 2)$ 

and finally,

 $P(Y=4)=1-[P(Y\le3)]$ 

since the individual probabilities must sum to one.

Protocol No. BHR-100-301

The missing GOS response will then be set to the most probable category, i.e. the response with the largest predicted probability.

It is anticipated that there will be minimal missing data, however sensitivity analyses will be carried out to confirm that the imputation method(s) did not have an impact on the primary efficacy analysis results. Therefore, the primary efficacy analyses will also be conducted on observed values only, without any imputation.

#### Covariates, missing data imputation

For the primary efficacy analyses, missing data for the following covariates will be imputed as the most commonly occurring value over subjects with non-missing data: motor response component of GCS, pupillary response, presence of hypoxia, presence of hypoxia, CT classification, and presence of traumatic subarachnoid hemorrhage.

#### GOS assessment – Dead responses

Subjects without a GOS response assessment at Month 6 but who have a death date from the Death Report eCRF within 6 months + 28 days of their randomization date (calculated as death date - randomization date + 1  $\leq$  208) will be assigned a Month 6 GOS response of Dead. Similarly, subjects without a GOS response assessment at Month 3 but who have a death date from the Death Report eCRF within 3 months + 28 days of their randomization date (calculated as death date - randomization date + 1  $\leq$  118) will be assigned a Month 3 GOS response of Dead.

## Secondary Endpoint: Mortality at Month 1

Survival status from the date of injury (Day 1 of the study) until Day 30 (Month 1) will be monitored and recorded as lost to follow-up, consent withdrawn, alive, dead or other. Only subjects with a mortality assessment post-injury of alive or dead will be used in the assessment of mortality.

#### Secondary Endpoint: Mortality at Month 6

Survival status from the date of injury (Day 1 of the study) until Day 180 (Month 6) will be monitored and recorded as lost to follow-up, consent withdrawn, alive, dead or other. Only subjects with a mortality assessment post-injury of alive or dead will be used in the assessment of mortality.

#### Time to death

The time to death (in days) will be defined as:

Date of death - date of TBI + 1

If a subject does not die during the conduct of the study, they will be censored at the earliest (minimum) of their Month 6 GOS assessment date and end of study date, and censor time (in days) will be defined as:

Minimum(month 6 GOS assessment date, end of study date) – date of TBI + 1

Since subjects were not followed for death after their Month 6 GOS assessment, subjects who have a death recorded after the assessment will be censored on the date of their Month 6 assessment.



#### **Exploratory Endpoint: CPP**

The following formulae are used to derive CPP:

Mean Arterial Pressure (MAP) = 2/3 diastolic BP + 1/3 systolic BP;

$$CPP = MAP - ICP$$
.

MAP will be recorded as missing if either systolic BP and/or diastolic BP measurements are not recorded. CPP will be calculated where MAP and ICP have both been recorded; if either is missing the CPP will be recorded as missing.

#### Exploratory Endpoint: TIL

TIL will be monitored during Study Days 1 - 6 (inclusive). The administration of each of the following unique treatments will have a score of 1 and the maximum score (sum of the individual items) per assessment period (study day) is 10:

- Surgical decompression,
- Barbiturate induced coma,
- Hypothermia for ICP reduction,
- Hyperventilation (pCO<sub>2</sub> < 30),
- Pressor administration,
- Hypertonic saline,
- Mannitol,
- Ventricular drainage,
- Paralysis induction,
- Sedation.

# Neuroworsening

Neuroworsening will be defined as the occurrence of any one of the following:

- A decrease in GCS motor score  $\geq 2$ ,
- Development of pupillary abnormalities,
- Any other neurological deterioration or progression of lesion on CT scan leading to a change in subject management.

# Pupillary Response

Pupillary response will come from the assessment of right and left pupil reactivity as follows:

- If both right and left pupils react, pupillary response = bilateral,
- If only one of the right or left pupil reacts, pupillary response = unilateral, and
- If neither right nor left pupil reacts = no reactive pupils, or
- If the eyes are closed and reactivity is untestable = not testable.

#### <u>Treatment-Emergent Adverse Events</u>

Treatment-emergent adverse events (TEAEs) are defined as events that start on or after the first dose of study medication. For this study it is intended that AEs will be collected for 15 days

after the initiation of study treatment; serious adverse events (SAEs) will be collected from the time of infusion start throughout the course of the subject's participation in the study (6 months).

All AE tables will be presented for TEAEs only, listings will present all AEs (including those not deemed to be TE).

#### **6 ANALYSIS SETS**

The following analysis populations will be defined for this study:

- Modified Intention-to-treat (mITT),
- Per Protocol (PP), and
- Safety.

The assignment of subjects to the study populations will occur at the blinded review meeting which will encompass discussion of major protocol violations.

#### 6.1 Modified Intention-to-Treat

The mITT population will include all randomized subjects in whom treatment with i.v. study drug was initiated. Following the ITT principle, subjects will be analyzed according to the treatment they were assigned at randomization regardless of any randomization errors or amount of study drug infusion administered.

The mITT population will be the primary efficacy population, and all efficacy analyses and summaries will be performed using this population. All demographic and baseline summaries will also be summarized using the mITT population.

#### 6.2 Per Protocol

The PP population will include all subjects in the mITT population who meet all the inclusion/exclusion criteria, received at least 96 hours over the course of 120 hours of study treatment (however, not excluding those subjects who die or are discontinued for an AE prior to receiving the full dose of 120 hours), and have a non-missing 6-month GOS score that was assessed at least 152 days from randomization. Subjects who initiate study drug infusion > 8 hours from time of injury but within 9 hours will be included in the PP population. The rationale for this is that the best available time of injury to the nearest hour is used at randomization, however a different time of injury may be determined later.

Study drug administration errors will be handled according to the following table when determining inclusion in the PP population:

# Table 1 Handling of Study Drug Administration Errors in the Per Protocol Analysis

| <b>Medication Error Scenar</b> | | |
|---|---|---|
| Randomized to | Study Drug of Erroneously<br>Received Bottle | Inclusion in PP Population |
| Placebo | Placebo | Included in placebo arm |
| Placebo | BHR-100 | Not included |
| BHR-100 | BHR-100 | Included in BHR-100 arm |
| BHR-100 | Placebo received as first administration of study drug or 2 or more bottles of placebo received at any time | Not included |
| BHR-100 | 1 placebo bottle received at any<br>time except the first<br>administration of study drug | Included in BHR-100 arm |

Subjects at any site that is removed from the study for noncompliance with ABIC/EBIC/ Brain Trauma Foundation guidelines will be excluded from the PP population.

No imputation of the 6-month GOS score will occur in the PP analysis, but missing covariates will be imputed as described in Section 5.

The PP population will be used to perform confirmatory analyses of the primary efficacy evaluation.

#### 6.3 Safety

The safety population will include all subjects who received any study drug. Subjects will be analyzed according to treatment received regardless of the randomization schedule. If a subject received *any* amount of BHR-100, they will be summarized according to treatment BHR-100 for the safety population.

The safety population will be used for all summaries of safety data and treatment exposure data.

#### 7 INTERIM ANALYSIS

A formal interim analysis will be performed once the first 200 subjects in each treatment arm (total of 400 subjects) have reached a study endpoint (death, lost to follow up, or completed the study and assessed for the 6-month GOS). The database used for the interim analysis will only contain these 400 subjects.

At the planned interim analysis, the test statistic based on the effect size (common odds ratio) will be compared to the critical value shown below. If the test statistic exceeds the critical value, the unblinded study statisticians will discuss the continuation of the trial with the DSMB and the DSMB will inform the Sponsor. In order to stop the trial at the interim analysis, the significance level will need to be less than the critical p-value (i.e. p < 0.0003).


At the planned interim analysis, a 2-sided test will be performed to detect either an increase or decrease in the common odds ratio, as described in the section of this document on primary end point analysis, section 9.5.1. In order to preserve the over-all type I error rate at 1%, the critical value for the test statistic will be inflated above 2.575, the value that would be used if no repeated testing were used. The actual critical values and p-values will be computed using statistical methods for group sequential testing with the O'Brien Fleming method.

If the p-value from the test of the null hypothesis of no treatment difference is less than 0.0003 at the interim analysis, the study may be stopped for efficacy. Table 2 indicates the critical values, p-values and cumulative type I error for this study:

Table 2
Critical Values and p-Values of Interim and Final Analyses

| Interim and final analyses | Total sample | Critical Value | p-value | Cumulative<br>Type I Error |
|---|---|---|---|---|
| Interim (1) | 400 | 3.65 | 0.0003 | 0.0003 |
| Final (2) | 1180 | 2.58 | 0.0098 | 0.0101 |

No formal stopping rule for futility will be established for this study. An assessment of conditional power at the interim analysis will be provided to the DSMB for consideration with the safety summaries in the evaluation of the overall risk/benefit of the study treatment.

Under the condition that the proportional odds model assumption holds, the statistical power to reject the null hypothesis of equal six-month GOS is shown below under a variety of scenarios (Table 3).

Conditional power is the estimate of the power to observe a difference in treatment groups different from that observed at the interim analysis. The conditional power is calculated based upon the observed critical value and measure of the completion of the trial. Methods for this calculation have been proposed by Lan, DeMets and Halperin and Lan, Simon and Halperin.

Table 3
Futility Analysis: Power to Reject Null hypothesis under Various Scenarios

| Common odds ratio <sup>1</sup> | | Power at interim and final analysis | |
|---|---|---|---|
| Placebo | BHR-100 | Interim analysis <sup>2</sup> | Final analysis <sup>3</sup> |
| 1.0 | 1.27 | 1.54% | 39.36% |
| 1.0 | 1.50 | 10.93% | 90.66% |
| 1.0 | 2.33 | 88.49% | 99.99% |

A common odds ratio of 1.27, 1.5 and 2.33 is equivalent to a 5%, 10% and 20% effect size respectively.

<sup>&</sup>lt;sup>2</sup> Interim analysis is based on the assessment of 400 completed subjects (200 in each arm).

Final analysis is based on total study recruitment at 1180 treated subjects with 590 in each arm. This sample size is calculated based on the defined baseline outcome distribution (31% Good Recovery, 21% Moderate Disability, 19% Severe Disability and 29% Vegetative State/Death) to detect a common odds ratio of 1.5 of improvement in outcome with 90% power and 1% significance level (2-sided).

In the event that the *final* primary efficacy analysis does not show statistical significance at the study-wise 1% significance level (i.e. the final analysis p-value is not less than 0.0098) a final adjusted p-value will be calculated and the result considered statistically significant at the 5% level if the adjusted p-value is less than 0.05. The adjusted p-value will be calculated using EAST (Cytel Statistical Software, Cambridge, MA) or other appropriate statistical software package to adjust for the interim analysis.

#### **8 DATA REVIEW**

#### 8.1 Data Handling and Transfer

For this study PRA International provides full Data Management services, including the development of the Data Management Plan (DMP) which outlines all Data Management activities to be undertaken. The DMP is a living document that evolves over the course of a trial and consists of the following documents:

- Data Management Process Summary,
- Annotated CRF,
- Data Management Quality Control Plan,
- Critical Variable List,
- Data Edit Specifications,
- Dictionary Coding Conventions,
- SAE/AE Reconciliation Plan,
- Electronic Clinical Data Handling Instructions, and
- Database Conversion Specifications.

For this study, PRA International defines and maintains the study database. The database will be provided to the PRA International Analysis and Reporting group in SAS dataset format.

Assessments will be conducted at the central bioanalytical laboratory for blood levels of progesterone.

# 8.2 <u>Data Screening</u>

Beyond the data screening built into the PRA DMP, programming of analysis datasets, tables, figures, and listings will be ongoing during the data management of the study. During this process potential data issues will be communicated to Data Management. Before the data are considered clean (as defined by PRA Data Management processes), blinded tables, figures, and listings will be run (using a dummy randomization) and distributed to the study team for review. Any data values requiring investigation or correction will be identified at that point, and protocol deviations will be reviewed and documented. Once all data issues have been resolved, the database will be locked, treatment codes unblinded, and the final run of outputs will take place.

Furthermore, during the conduct of the study, an independent DSMB will meet to conduct safety reviews of the data, at approximately 100-subject intervals. The duties, operational procedures, and frequency of meetings/teleconferences are described in the DSMB Charter. At each meeting, the DSMB can recommend early trial termination or study modification in response to safety concerns.

The DSMB can request additional, unplanned, unblinded analysis of primary outcome data in case of major safety issues from the safety analysis. Therefore, the DSMB will be able to monitor the study in its completeness by analyzing the overall risk/benefit of the trial results as necessitated by safety concerns that may arise.

#### 9 STATISTICAL METHODS

All analyses and reporting of study results will be conducted using SAS V9.1.3 In addition EAST will be used to adjust for the interim analysis.

All variables will be presented using appropriate descriptive statistics according to the variable nature:

- Continuous variables: number of non-missing observations, mean, standard deviation, minimum, first quartile (Q1), median, third quartile (Q3), maximum,
- Categorical variables: number of non-missing observations, absolute and relative frequency (n and percentages (%)),
- Time-to-event variables: number of non-missing observations, number and percentage of censored observations, first quartile, median (and 95% CI), third quartile, and Kaplan-Meier survival curves.

The behavior over time of continuous variables will be analyzed by presenting descriptive statistics for each time point and the difference compared to baseline (actual values and change from baseline). The behavior over time of categorical data will be analyzed by presenting the descriptive statistics for each time point and the shift compared to baseline.

The decimal places for summary statistics and percentages will be as follows:

- Precision of data + 2 decimal places (dp) for standard deviations,
- Precision of data + 1 dp for means, medians and quartiles,
- Same precision as data for minimum and maximum,
- 1 dp for percentages except when the percentage is 100% in which case no dp would be presented, and

The primary and confirmatory efficacy analyses will be 2-sided and conducted at a 1% significance level. All secondary efficacy tests will be 2-sided and conducted at a 5% significance level.

The randomization will be stratified by region. This variable will be included as a covariate in the primary and secondary GOS efficacy analyses.

Secondary efficacy analyses will be conducted in ranked order as listed in Section 9.5.2 with the understanding that no confirmatory claims can be based on variables that have a rank lower than or equal to that variable whose null hypothesis was the first that could not be rejected at the p<0.05 significance level.

All exploratory analyses will be considered supportive in nature, and therefore no adjustment will be made for multiple testing of exploratory variables.

All data will be included in subject data listings for all subjects in the mITT population.



# 9.1 Subject Disposition

An enrollment summary will be presented overall and by site, showing the first date of consent, the date of the last subject randomized, duration (in days) (calculated as end date – start date +1), and number of subjects randomized and completed endpoint.

The number and percentage of subjects randomized in total, by site, by country and by region will be summarized for each treatment group and overall for the mITT population.

The number and percentage of subjects in each study population (mITT (randomized and treated with i.v. study drug), randomized but not treated, PP, Safety, Study Completers, Endpoint Completers (includes deaths prior to Month 6), and Early Terminations) and the reasons for early termination will be summarized by treatment group and overall for mITT subjects.

Subjects remaining in the study by time will also be summarized.

These details will also be listed.

# 9.2 Protocol Deviations and Violations

Subjects with protocol violations that result in exclusion from the PP population will be listed.

## 9.3 <u>Treatments</u>

#### 9.3.1 Extent of Study Drug Exposure

The number of subjects in each of the following categories will be summarized for each treatment group and overall for the safety population:

- Who initiated study drug within 8 hours of injury,
- Who were treated for at least 96 hours,
- Who prematurely discontinued study drug (with the corresponding reason for discontinuation).

Duration of study drug exposure and total dose will also be summarized for the safety population. The duration of study drug exposure (in hours) will be summarized as both a continuous and categorical variable by treatment group and overall. Total dose (in mg/kg) will also be summarized as a continuous variable. Total dose received in milligrams will be adjusted by a subject's weight entered into IWRS at the time of randomization.

Continuous and categorical summaries of time since injury to study drug initiation will be presented.

Counts and percentages of subjects with any infusion rate modifications or interruptions, and the reasons for infusion rate modifications and interruptions, will be summarized by treatment group and overall for the safety population.

The percentage compliance with study medication will be summarized by treatment group and overall for the safety population as a continuous variable. See Section 5 for further details.


# 9.3.2 Concomitant Medications, Concomitant Procedures and Surgical Therapy

Prior medications are defined as medications with a start date before the first initiation of study medication. Concomitant medications are defined as medications which:

- Started after the initiation of study medication,
- Had a stop date on or after the first administration of study medication, or
- Are ongoing on Day 15.

It is possible for a medication to be both prior and concomitant. It should be noted that medications administered to or taken by the subject during the study will only be recorded from the time of informed consent through to Day 15 of the study.

Medications with partial start dates will be determined as prior and/or concomitant medications by using available non-missing information. Medications with completely missing start dates (i.e. missing information for medication start day, month, and year) will be assumed to be concomitant. If just the day is missing, and the month and year are the same as the month and year of study drug administration, the medication will be considered concomitant. If the day and month are missing and the year is present, and is the same as the year of study drug administration, the medication will be considered concomitant.

Medications will be coded using the WHO (World Health Organization) Drug Dictionary March 2010 version international thesaurus with no updates, adding WHO-DD preferred term for use in the relevant tabulation. Counts and percentages for prior and concomitant medications will be summarized by preferred term, treatment group and overall for the mITT population.

The number and percentage of subjects with intracranial and extracranial surgery will be summarized by surgery type, actual surgical procedure (for example, craniofacial surgery), treatment group and overall for the mITT Population.

# 9.4 <u>Demographic and Baseline Characteristics</u>

Demographic variables (age, sex, ethnicity and race), pregnancy testing, and baseline characteristics (geographical region, GCS motor score, pupillary response, presence of hypoxia, presence of hypotension, classification of CT scan, presence of traumatic subarachnoid hemorrhage) will be summarized for each treatment group and overall.

The cause of TBI and type of injuries (face, chest, abdomen, extremities, spine, head injury alone) will be summarized by treatment group and overall.

Medical histories will be coded using Medical Dictionary for Regulatory Activities (MedDRA) version 13.0 with no updates. The number and percentage of subjects reporting any medical history will be displayed together with the number and percentage of subjects having at least one medical history within each system organ class (SOC) and preferred term.

#### 9.5 <u>Efficacy Analyses</u>

#### 9.5.1 Primary Efficacy Analysis

The primary efficacy variable is GOS evaluated at 6 months post injury. The primary analysis will be based on imputation of missing data as described in Section 5.

#### 9.5.1.1 Proportional Odds Model

The primary efficacy variable of GOS at 6 months post injury will be compared between treatment groups using a POM. For the purposes of this analysis the first two categories of the GOS will be combined (vegetative state and dead). A POM will be fitted including the effect of treatment, geographic region (North America, Europe, Asia, and South America), age, GCS motor score, pupil response, and CT classification. With 4 categories in the response variable, GOS at 6 months following injury, the POM simultaneously fits 3 (number of categories – 1) binary logistic regression models as follows.

If Y = response = GOS at 6 months following injury.

#### Model 1

 $Y_1 = 0$  (not event), if Y =vegetative state or dead

 $Y_1 = 1$  (event), if Y = severe disability, moderate disability, good recovery

#### Model 2

 $Y_2 = 0$  (not event), if Y =vegetative state or dead, severe disability

 $Y_2 = 1$  (event), if Y = moderate disability, good recovery

#### Model 3

 $Y_3 = 0$  (not event), if Y = vegetative state or dead, severe disability, moderate disability

 $Y_3 = 1$  (event), if Y = good recovery

The dichotomous logistic regression models for  $Y_J$  (J=1, 2, 3) can be expressed as follows:

$$\ln (P_J/(1-P_J)) = \alpha_J + \beta_1 X_1 + \beta_2 X_2 + \beta_3 X_3 + \beta_4 X_4 + \beta_5 X_5 + \beta_6 X_6,$$

#### where

- In is the natural logarithm,
- $P_J$  = Probability of an 'event' (for example, good recovery) = Probability that  $Y_J = 1$ ,
- $P_J/(1 P_J) = odds of an 'event',$
- $X_1$  = treatment group,
- $\beta_1$  = effect of treatment,
- $X_2 = region$ ,
- $\beta_2$  = effect of region,
- $X_3 = age$ ,
- $\beta_3$  = effect of age,
- $X_4 = GCS$  motor score,
- $\beta_4$  = effect of GCS motor score,
- $X_5 = \text{pupil response}$ ,
- $\beta_5$  = effect of pupil response, and
- $X_6 = CT$  classification,
- $\beta_6$  = effect of CT classification.



With a POM, it is assumed that the effect of the explanatory variables, such as treatment, are identical for all possible dichotomies of the response variable, that is,  $\beta_1$ , etc. are the same for each model.

The fact that the effects of the explanatory variables (e.g. treatment ( $\beta_1$ ), etc.) are the same for each model is referred to as the proportional odds assumption and needs to hold for this methodology to be appropriate. This assumption will be tested using the Score Test. A non-significant result (p-value > 0.05) supports the assumption of proportional odds. As the Score Test is known to be anti-conservative, additional graphical methods will be used to assess the proportional odds assumption in greater detail, if the Score Test is statistically significant.

The proportional odds assumption for an ordinal response implies that the curves on the various cumulative logits are parallel. This assumption can be assessed visually for a given predictor (e.g. region) by plotting it against the empirical logits.

For the 4 levels of the GOS there will be 3 cumulative logits which can be expressed as:

```
Logit<sub>1</sub> = log[ p_1/(1-p_1) ] = log[ p_1/(p_2+p_3+p_4) ],

Logit<sub>2</sub> = log[ (p_1+p_2)/(1-(p_1+p_2)) ] = log[ (p_1+p_2)/(p_3+p_4) ],

Logit<sub>3</sub> = log[ (p_1+p_2+p_3)/(1-(p_1+p_2+p_3)) ] = log[ (p_1+p_2+p_3)/(p_4) ]

where p_i = P(Y=i), where Y (response, GOS at 6 months) = i and i=1, 2, 3 or 4.
```

By using the observed counts,  $y_i$ , in the study data empirical logits can be computed for use in plots as follows:

```
EmpLogit<sub>1</sub> = log[(y_1)/(y_2+y_3+y_4)]
```

where  $y_i$ =number of subjects with Y (response, GOS at 6 months) = i and i=1, 2, 3 or 4.

The empirical logits can then be calculated for each category of the predictor and plotted. If the resulting plotted lines are roughly parallel this can be considered a visual confirmation of the proportional odds assumption.

See Appendix 3 (Model Checking Figures) for plot specification details.

Provided that the proportional odds assumption is not rejected, the POM will then be used to test the null hypothesis that the odds of being "higher" or "lower" on the outcome variable, GOS at 6 months following injury, across the entire range of the outcome, adjusted for region, age, GCS motor score, pupil response, and CT classification (as defined in Section 4.3) is the same in both treatment groups, i.e.

Null Hypothesis:  $H_0: \beta_1 = 0$ Alternative Hypothesis:  $H_1: \beta_1 \neq 0$  If the p-value from the test of the null hypothesis of  $\beta_1 = 0$  is less than 0.0003 (at the interim) or 0.0098 (at the final analysis), it will be concluded that BHR-100 is statistically significantly different from placebo with respect to the GOS at 6 months following injury. The odds of some degree of improvement in the GOS at 6 months will be modeled and the corresponding common odds ratio for treatment,  $e^{\beta_1}$ , can then be interpreted to determine the direction of the treatment difference as follows. With the placebo group being considered as the reference category, if the odds ratio (OR<sub>BHR-100/placebo</sub>) is greater than 1, the odds of some improvement in the GOS at 6 months is greater in the BHR-100 treatment group compared to placebo.

In the event that the primary efficacy analysis does not show statistical significance at the study-wise 1% significance level, please refer to section 9.5.1.4 for further details on how the statistical significance of the primary efficacy analysis should be interpreted.

The POM will be fitted in SAS® using the PROC LOGISTIC procedure.

Goodness of fit of the model will be assessed using the Deviance and Pearson tests (add SCALE = NONE AGGREGATE to the MODEL statement of PROC LOGISTIC) to compare the fitted model with the saturated model. If these tests are not statistically significant it implies that the model fits the data adequately.

The score test for the proportional odds assumption and individual p-values associated with the tests of effects (treatment, geographic region, age, GCS motor score, pupil response, and CT classification) will be summarized for the POM of GOS at 6 months post injury.

The odds ratios and associated 95% CIs for the levels of the effects relative to a reference category will be presented for all factors and covariates included in the POM of GOS at 6 months post injury.

In addition to the results of the hypothesis tests from the statistical modeling, the number of non-missing observations, absolute and relative frequency (n and percentages), will be provided by treatment group for the GOS categories at 6 months post injury.

The analyses above will be repeated for the straight observed case analysis (no imputation of 6-month GOS or covariates) in the mITT population, the straight observed case analysis in the PP population (no imputation of 6-month GOS or covariates), and the analysis of imputed missing values in the mITT population for US subjects only.

In addition to the above POM for the primary analysis, the individual binary logistic regression models will be fitted for each possible dichotomization of the GOS at 6 months, as outlined above under model 1, 2 and 3. This will be done using missing value imputation for the mITT population. This will allow an assessment of the odds ratio for treatment within each possible dichotomization and a further assessment of the proportional odds assumption. If the parameter estimates obtained under each dichotomized model are similar then the proportional odds assumption would seem sensible.

A bar chart illustrating the percentage of responses in each GOS category for each treatment group will be produced for the GOS at 6 months for the mITT (observed values and missing values imputed) and PP populations (observed values).

#### 9.5.1.2 **Alternate Primary Efficacy Analysis (Sliding Dichotomy)**

If the proportional odds assumption cannot be justified, a sliding dichotomy of the GOS outcome at 6 months following injury, following categorization of subjects into different prognosis groups (worst, intermediate, and best) based on baseline prognostic factors, will be the primary efficacy analysis. The primary sliding dichotomy analysis will be based on imputation of missing data (covariates and 6-month GOS assessments).

For each subject a baseline prognostic risk score (BPRS) will be calculated as a weighted linear function of baseline prognostic factors of age, age squared, GCS motor score, Marshall CT classification, pupillary reactivity, presence of hypoxia, presence of hypotension, and presence of traumatic subarachnoid hemorrhage. The weighting of the BPRS factors will be based on the prognostic model developed in Hukkelhoven et al (2005). The BPRS will be sorted from lowest to highest, noting that higher BPRS represent a worse prognosis, and split into tertiles which will represent best, intermediate and worst prognosis.

For the cohort predicted to have the worst outcome, the outcome of severe disability or better is considered a "favorable outcome," while for the cohort predicted to have the best outcome, only the outcome of good recovery is considered a "favorable outcome." For the middle cohort there is no difference from the dichotomized model, so that the outcomes of moderate disability and good recovery are pooled to define "favorable outcome."

The hypothesis that the proportion of favorable responses observed in each treatment group is the same will be tested using the Cochran-Mantel Haenszel (CMH) Chi-Square test, adjusted for region.

Null Hypothesis:  $H_0: p_1 = p_2$ Alternative Hypothesis:  $H_1: p_1 \neq p_2$ 

where  $p_1$  = proportion of favorable responses in the BHR-100 treated group and  $p_2$  = proportion of favorable responses in the placebo treated group. The Mantel-Haenszel estimate of the common odds ratio and corresponding 95% CI will also be presented.

If the p-value from the test of the null hypothesis of  $p_1 = p_2$  is less than 0.0003 (at the interim) or 0.0098 (at the final analysis), it will be concluded that there is a statistically significantly difference in the proportion of favorable responses between the 2 treatment groups.

In addition to the formal inference testing discussed above, the difference in proportion of favorable outcomes and associated 2-sided 95% confidence interval between the BHR-100 and placebo treatment groups will be calculated.

In addition to the primary analysis that tests whether the overall proportion of favourable responses is the same in each treatment group, the CMH test results and odds ratios by baseline prognosis grouping (best, intermediate, worse) will also be presented. The Breslow-Day test will be computed to test whether the odds ratios are different across the prognostic groups. A significant test result will not affect the validity of the overall test of a difference between treatment groups, but will aid in the interpretation of the results.

The analyses above will be repeated for the straight observed case analysis (no imputation of 6-month GOS or covariates) in the mITT population, the observed case analysis in the PP population, and the analysis of imputed missing values in the mITT population for US subjects only.

#### 9.5.1.3 Sensitivity Analysis (Dichotomized Model)

The GOS at 6 months post injury will be dichotomized into Good Recovery, Moderate Disability versus Severe Disability, Vegetative Status/Dead. As a supportive analysis, the binary outcome will be analyzed using logistic regression analysis. The logistic regression model will be fitted including the effect of treatment, geographic region (North America, Europe, Asia, and South America), age, GCS motor score, pupil response, and CT classification.

If Y = response = GOS at 6 months following injury.

#### Model

 $Y_1 = 0$  (not event), if Y = vegetative state or dead, severe disability  $Y_1 = 1$  (event), if Y = moderate disability, good recovery

The dichotomous logistic regression model can be expressed as follows:

$$\ln (P/(1-P)) = \alpha_J + \beta_1 X_1 + \beta_2 X_2 + \beta_3 X_3 + \beta_4 X_4 + \beta_5 X_5 + \beta_6 X_6,$$

#### where

- In is the natural logarithm,
- P = Probability of an 'event' (moderate disability, good recovery) = Probability that Y = 1,
- P/(1-P) = odds of an 'event',
- $X_1$  = treatment group,
- $\beta_1$  = effect of treatment,
- $X_2 = region$ ,
- $\beta_2$  = effect of region,
- $X_3 = age$ ,
- $\beta_3$  = effect of age,
- $X_4 = GCS$  motor score,
- $\beta_4$  = effect of GCS motor score,
- $X_5 = \text{pupil response}$ ,
- $\beta_5$  = effect of pupil response, and
- $X_6 = CT$  classification,
- $\beta_6$  = effect of CT classification.

The logistic regression model will be used to test the null hypothesis that the odds of an 'event', i.e. observing a response of moderate disability or good recovery on the outcome variable, GOS at 6 months following injury, adjusted for region, age, GCS motor score, pupil response, and CT classification is the same in both treatment groups, i.e.


If the p-value from the test of the null hypothesis of  $\beta_1$  = 0 is less than 0.05, it will be concluded that BHR-100 is statistically significantly different from placebo with respect to the GOS at 6 months following injury. The odds of an 'event' (moderate disability or good recovery) in the GOS at 6 months will be modeled and the corresponding common odds ratio for treatment,  $e^{\beta_1}$ , can then be interpreted to determine the direction of the treatment difference as follows. With the placebo group being considered as the reference category, if the odds ratio (OR<sub>BHR-100/placebo</sub>) is greater than 1, the odds of a favorable outcome in the GOS at 6 months is greater in the BHR-100 treatment group compared to placebo.

The logistic regression analysis will be fitted in SAS® using the PROC LOGISTIC procedure.

Goodness of fit of the model will be assessed as outlined above for the Proportional Odds Model.

The individual p-values associated with the tests of effects (treatment, geographic region, age, GCS motor score, pupil response, and CT classification) will be summarized for the Logistic Regression Model of GOS at 6 months post injury.

The odds ratios and associated 95% CIs for the levels of effects relative to a reference category will be presented for all factors and covariates included in the Logistic Regression Model of GOS at 6 months post injury.

In addition to the results of the hypothesis tests from the statistical modeling, the number of non-missing observations, absolute and relative frequency (n and percentages), will be provided by treatment group for the dichotomized GOS categories at 6 months post injury.

The primary dichotomized analysis will be based on missing values of 6-month GOS and covariates imputed. It will also be repeated for the straight observed case analysis (no imputation of 6-month GOS or covariates) in the mITT population and the straight observed case analysis in the PP population.

A bar chart illustrating the percentage of responses in each of the dichotomized categories for each treatment group will be produced for the GOS at 6 months (observed values and missing values imputed) for the mITT population.

#### 9.5.1.4 Interpretation of Statistical Significance of Primary Efficacy Analysis

In the event that the primary efficacy analysis does not show statistical significance at the study-wise 1% significance level, i.e. the final analysis p-value is not less than 0.0098, a final adjusted p-value will be calculated and the result considered statistically significant at the 5% level if the adjusted p-value is less than 0.05. The adjusted p-value will be calculated using EAST (Cytel Statistical Software, Cambridge, MA) or other appropriate statistical software

package to adjust for the interim analysis using the pre-specified boundaries discussed above and in section 7.

# 9.5.1.5 Handling of Missing Data

Please refer to section 5 for further details on the handling of missing data.

#### 9.5.1.6 Exploratory Analysis

An exploratory analysis will be conducted to assess each of the following covariates of interest: treatment (BHR-100 vs. placebo), region (North America vs. Europe vs. Asia vs. South America), age, race (white vs. non-white), GCS motor score (1-2 vs. 3 vs. 4 vs. 5-6), pupil response (bilateral vs. unilateral/no reactive pupils/not testable), CT classification (I/II vs. III vs. IV vs. V/VI), presence of hypoxia (yes/suspected vs. no/unknown), presence of hypotension (yes/suspected vs. no/unknown), presence of traumatic subarachnoid hemorrhage (yes vs. no), gender (male vs. female), and time to first dose of study medication from TBI (0-4 vs. 4-6 vs. 4-8 vs. >8 hours), for inclusion into an expanded model. Each covariate, along with the corresponding interaction with treatment term, will be included in a simple model with treatment. A backward selection model will be fit beginning with all covariates. Factor by treatment interactions will be included in the backward elimination model if the p-value<0.10 in the corresponding simple model. A significance level of 0.05 may be too stringent and may exclude important variables from the model, so a significance level of 0.1 will be used for the backward selection process. If the interaction term is significant, an exploratory subgroup analysis will be performed for the corresponding covariate.

This analysis will be conducted for the POM based on imputation of missing data. Missing covariates will not be imputed for the exploratory analysis.

#### 9.5.2 Secondary Variables

Secondary efficacy parameters will be ranked as follows:

- 1) GOS-E at Month 6,
- 2) Mortality at Month 6 in mITT population (comparison of incidence of death),
- 3) GOS at Month 3,
- 4) GOS-E at Month 3,
- 5) Mortality at Month 1 in mTT population (comparison of incidence of death),
- 6) SF-36 mental composite score at Month 6,
- 7) SF-36 physical composite score at Month 6
- 8) SF-36 mental composite score at Month 3, and
- 9) SF-36 physical composite score at Month 3.

No confirmatory claims can be based on variables that have a rank lower than or equal to the variable whose null hypothesis was the first that could not be rejected at the p<0.05 significance level.



# 9.5.2.1 Mortality at Month 1, Month 6

These efficacy variables are obtained by collecting the survival status from the date of injury (Day 1 of the study) until Day 30 (Month 1) and Day 180 (Month 6) respectively as lost to follow-up, consent withdrawn, alive, dead or other. Every effort will be made to ascertain the survival status of subjects with status other than dead or alive, but in the absence of further information these observations will be omitted from the analysis. The 1-month mortality rate will be defined as the proportion of subjects at risk in the mITT population (subjects for whom the survival status at Day 30 is known) who died on or before Study Day 30. Similarly, the 6-month mortality rate will be defined as the proportion of subjects at risk in the mITT population who died on or before Study Day 180.

The hypothesis that the mortality rate observed in each treatment group is the same will be tested using the Fisher's Exact test.

Null Hypothesis:  $H_0$ :  $p_1 = p_2$ Alternative Hypothesis:  $H_1$ :  $p_1 \neq p_2$ 

where  $p_1$  = proportion of deaths in the BHR-100 treated group and  $p_2$  = proportion of deaths in the placebo treated group.

A 2-sided, 5% significance level will be used to test the null hypothesis. If rejected (p < 0.05), it will be concluded that there is a statistically significant difference in the proportion of deaths between the 2 treatment groups.

In addition to the formal inference testing discussed above, 2-sided 95% confidence intervals for the difference in the proportion of deaths between BHR-100 and placebo treatment groups will be calculated.

Summaries of mortality at Months 1 and 6 will be presented for both the mITT and PP populations.

The mortality rate for each treatment group will also be plotted on a bar chart for mortality at 1 and 6 months for the mITT population.

#### 9.5.2.2 GOS at Month 3

The GOS at Month 3 will be analyzed using the POM in the same way as the primary efficacy analysis of GOS at Month 6 outlined above for the observed values.

# 9.5.2.3 GOS-E at Month 3 and Month 6

The GOS-E at Month 3 and Month 6 will be analyzed using the POM, similar to the primary efficacy analysis of the GOS at Month 6 described above. The GOS-E is an 8-point scale with the following categories:

- Dead (D),
- Vegetative state (VS),
- Lower severe disability(SD LL),
- Upper severe disability (SD UL),
- Lower moderate disability (MD LL),



- Upper moderate disability (MD UL),
- Lower good recovery (GR LL),
- Upper good recovery (GR UL).

For the POM analysis, the first 2 categories will be combined (vegetative state and dead). With 7 categories in the response variable, the POM simultaneously fits 6 binary logistic regression models. If the proportional odds assumption cannot be justified, the GOS-E at Month 6 will be analyzed using the SD as described in Section 9.5.1.2. For each subject, a BPRS will be calculated as described in Section 9.5.1.2. Subjects will be sorted from lowest to highest based on BPRS, and split into 6 equal groups representing different prognosis groups. The first prognosis group, representing the lowest BPRS and therefore the best prognosis, will be Group 1. The definition of a favorable or unfavorable outcome for each group will be defined as in Table 4.

Table 4
Sliding Dichotomy Groupings for GOS-E

| Group | Unfavorable Outcome | Favorable Outcome |
|-----------------|---------------------|-------------------|
| 1 | D+VS+SD+MD+GR LL | GR UL |
| 2 | D+VS+SD+MD | GR |
| 3 D+VS+SD+MD LL | | MD UL+GR |
| 4 | D+VS+SD | MD+GR |
| 5 D+VS+SD LL | | SD UL+MD+GR |
| 6 | D+VS | SD+MD+GR |

D= Dead, VS=Vegetative state, SD=Severe Disability, MD=Moderate Disability, GR=Good Recovery, SD LL=Lower severe disability, SD UL=Upper severe disability, MD LL=Lower moderate disability, MD UL=Upper moderate disability, GR LL=Lower good recovery, GR UL=Upper good recovery

The hypothesis that the proportion of favorable responses observed in each treatment group is the same will be tested using the CMH test as described above.

The analyses of the GOS-E at Month 3 and Month 6 will be done for the straight observed case analysis only.

# 9.5.2.4 Quality of Life: SF-36

During the conduct of the study, the SF-36 health survey will be administered at Months 3 and 6 to assess quality of life with respect to health status. Since a baseline SF-36 is not assessed prior to study treatment, the analyses of the SF-36 will compare mean SF-36 scores at Month 3 and 6 between treatment groups.

The SF-36 consists of 36 questions that are grouped into eight scaled scores. These scores are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight.

For each scale, a simple mean imputation of missing data with a restriction to cases where the subject has completed at least 50% of the items of that scale (the "half-scale" rule) will be used.

The eight sections are as follows:

- Vitality,
- Physical functioning,
- Bodily pain,
- General health perceptions,
- Physical role functioning,
- Emotional role functioning,
- Social role functioning, and
- Mental health.

Summary statistics for the 8 scales and the physical and mental composite summary scores will be presented for each treatment group.

In addition to summarizing the data, the physical and mental composite summary scores at Month 3 and 6 will be analyzed using an analysis of covariance (ANCOVA) model including treatment group.

The null hypothesis that the mean physical and mental summary scores are the same for both treatment groups (BHR-100 and placebo) will be tested against the 2-sided alternative hypothesis that the mean physical and mental summary scores are different in each treatment group, at the 0.05 significance level.

The least square means for the treatment groups, difference in least square means between the treatment groups, effect size calculated as the absolute difference in least square means between BHR-100 and placebo divided by the root mean square, and p-value for difference between treatment groups will be presented.

A 2-sided, 5% significance level will be used to test the null hypothesis. If rejected at the 5% level (p < 0.05), it will be concluded that there is a statistically significant difference in the relevant summary score between the 2 treatment groups. The magnitude of the summary statistics will be examined to determine the direction of the treatment difference.

Diagnostic residual plots will be evaluated to test for violations of normality. If the normality assumption for the model is not met, the null hypothesis that the mean physical and mental summary scores are the same in each treatment group will be tested using the 2-sided Wilcoxon Rank-Sum test, an unstratified non-parametric test, which can be obtained from the NPAR1WAY procedure in SAS<sup>®</sup>.

#### 9.5.3 Exploratory Variables

#### **9.5.3.1** Time to Death

The actual time to death will be analyzed for the mITT population.

If a subject does not die during the conduct of the study, they will be censored at their Month 6 GOS assessment or end of study date, whichever comes first.



The LIFETEST procedure in SAS® will be used to produce Kaplan-Meier plots and estimates of 25th, 50th, and 75th quartiles and corresponding 95% confidence limits of the median time to death. The 2 treatment groups will be compared using a 2-sided log-rank test. Examination of the point estimates will indicate the direction of the treatment difference. The cumulative percent mortality based on the Kaplan-Meier survival probability estimates will be plotted for each treatment group.

The time to death (in days) will be further analyzed using a Cox proportional hazard model. The comparison of the treatment effect on the time to death will be based on the hazard ratio (HR) from the Cox regression model using the PHREG procedure in SAS<sup>®</sup>. Estimates of HR and 95% confidence limits will be presented. The model will include the same terms as the primary efficacy analysis, namely treatment, region, age, GCS motor score, pupil response, and CT classification.

The Cox proportional hazards model is a standard model used in failure time analysis. Compared to parametric analyses, its assumptions are fairly unspecified and will therefore yield robust estimates of the treatment effect. The model will be applied using the Efron approach for handling ties, since this approach is known to give a reasonable approximation of the exact likelihood in the presence of ties and is computationally faster when large amounts of data are being analyzed.

#### 9.5.3.2 Comparison of CT scans at admission and Day 6

A CT scan will be performed before randomization (Day 1) and once again at Day  $6 \pm 1$  day post-injury to assess the progression of lesion volume and brain edema. The findings by the Central Reader will be classified in accordance with the Marshall classification:

- Diffuse injury I no visible pathology (CT class I),
- Diffuse injury II (CT class II),
- Diffuse injury III swelling (CT class III),
- Diffuse injury IV shift (CT class IV),
- Evacuated mass lesion (CT class V),
- Non-evacuated mass lesion (CT class VI).

A shift summary of CT classification from Baseline to Day 6 will be presented by treatment group.

#### 9.5.3.3 ICP

Intracranial Pressure (ICP) will be collected for Days 1 - 6 of the study, at the investigators' discretion.

Descriptive summary statistics, categorical summaries (maximum daily ICP: 0 to <15,  $\geq$ 15 to <25,  $\geq$ 25 to <40 and  $\geq$ 40 mmHg and maximum daily ICP: 0 to  $\leq$ 20, >20 mmHg), and the number of subjects with maximum daily ICP  $\geq$ 25 and maximum daily ICP >20 mmHg (cutpoints of particular interest) will be presented for the maximum ICP by treatment group and study day for the mITT population.



#### 9.5.3.4 CPP

CPP is computed based upon simultaneously recorded ICP and blood pressure measurements, see Section 5 for formula. Summary statistics for the highest and lowest daily CPP values will be presented for each treatment group by Study Day.

CPP measurements in the following potentially clinically relevant categories will be presented for each treatment group: less than 50 mmHg, 50-<60 mmHg, 60-<70 mmHg and greater than or equal to 70 mmHg. The number and percentage of subjects within the various categories by Study Day will be summarized by treatment group.

Summary statistics will also be presented for the percentage of subjects with CPP measurements within the above specified categories at any time during treatment, where on-treatment will include all scheduled and unscheduled CPP measurements after the initiation of study medication.

#### 9.5.3.5 TIL

TIL will be monitored during Study Days 1 - 6 (inclusive) while ICP is being monitored (i.e. up to 6 days).

Each of the unique treatments given on a study day used for ICP management will have a score of 1, and the maximum score (sum of the individual items) per assessment period (study day) is 10. It is assumed that there will be a stepwise progression of therapy (from sedation to surgical decompression). However, in the event that the most aggressive therapies are used, i.e. the subject has barbiturate administration or surgical decompression, this will result in a TIL score of 10 regardless of which of the other therapies have been administered.

The number of non-missing observations, absolute and relative frequency (n and percentage) of the subjects having at least one occurrence of the individual therapies (surgical decompression, barbiturate induced coma, hypothermia for ICP reduction, hyperventilation, pressor administration, hypertonic saline, mannitol, ventricular drainage, paralysis induction, and sedation) will be summarized for each treatment group. The most aggressive therapy received during Days 1-6, expressed as the highest stepwise level of the TIL, will also be summarized. Furthermore, the daily TIL score will be summarized as a continuous variable by Study Day and treatment group.

#### 9.6 Safety Analyses

#### 9.6.1 Adverse Events

For this study, it is intended to limit the collection of AEs to the window in which events are considered treatment-emergent. Treatment-emergent adverse events (TEAEs) are defined as events that start on or after the first dose of study medication and up to 15 days and 6 months after the initiation of study treatment, for AEs and SAEs respectively.

Partial start dates of AEs will be imputed in order to determine whether or not the AE is TE. If just the day is missing, and any date of dose administered is within the month of the AE, the AE will be treated as TE. If the month is missing and the year is present, and any date of dose administered is within the year of the AE, the AE will be treated as TE. If the year is missing,

the AE will be treated as TE. For the imputation, the day will be set to the first date of that month, or the first dose date, if the first dose date is within that month. Alternatively, if the month is missing the month will be set to January, or the first dose date, if the first dose date is within that year.

AEs will be coded using the MedDRA international thesaurus version 13.0 with no updates, adding system organ class (SOC) and preferred term. The AE summaries will be presented for TEAEs only. The total number of subjects reporting at least one AE and the number of AEs will be summarized by treatment group. The initial summary will also provide a breakdown of events that:

- Are treatment-related,
- Are serious,
- Are treatment-related and serious,
- Resulted in the study drug being prematurely discontinued,
- Are treatment-related and resulted in the study drug being prematurely discontinued,
- Resulted in death, and
- Are treatment-related and resulted in death.

Additionally, the overall summary of AEs will be summarized by treatment group for the subgroups of interest: gender, race group (white vs. non-white vs. not allowed to obtain), and age group ( $\leq$ 45 years vs.  $\geq$ 45 years).

The number and percentage of subjects with at least one TEAE and the number of TEAEs will be presented by SOC, preferred term, and treatment group for the following summaries:

- All AEs,
- All AEs by gender,
- All AEs by race group,
- All AEs by age group,
- Treatment-related AEs,
- All AEs, by maximum severity,
- Treatment-related AEs, by maximum severity,
- All AEs, by maximum relationship,
- All AEs that resulted in the study drug being prematurely discontinued, and
- Treatment-related AEs that resulted in the study drug being prematurely discontinued.

Additionally, the following AEs of special interest will be presented by treatment group: serious thromboembolic events such as thrombotic myocardial infarction, pulmonary embolism, deep vein thrombosis, ischemic stroke; allergic reactions; marked liver function abnormalities; serious infections such as pneumonia, sepsis, meningitis. Preferred terms for each AE of special interest will be identified by medical review prior to unblinding for the primary analysis. Preferred terms related to the following events will also be grouped to ensure similar events that are coded to different terms using MedDRA are summarized together: electrolyte imbalance, anemia, infusion site reactions, thrombocyte disorders, and seizures. These events will also be listed.



#### 9.6.2 Neuroworsening

See Section 5 for definition of neuroworsening. The incidence of any episode of neuroworsening occurring  $\leq$  Day 6 and  $\leq$ Day 15 will be summarized.

Details of all neuroworsening events will also be listed.

#### 9.6.3 Deaths and Serious Adverse Events

The number and percentage of subjects with at least one SAE and the number of events will be presented by SOC, preferred term and treatment group for the following summaries:

- All SAEs, and
- Treatment-related SAEs.

The primary cause of death as recorded on the death report will be summarized by treatment group and overall for the mITT population.

#### 9.6.4 Laboratory Data

Laboratory data (coagulation, hematology, serum chemistry and urinalysis) will be collected at baseline, end of study treatment (Day 6), and Day 15 of the study.

The status of clinically significant (non AE) abnormalities (resolved, ongoing, or lost to follow-up) will be summarized for Day 15 by laboratory parameter and treatment group in the safety population.

Clinically significant (non-AE) abnormal lab results (coagulation, hematology, serum chemistry, and urinalysis) will be listed.

Coagulation, hematology, and serum chemistry laboratory assessments will also be summarized descriptively for baseline, Day 6, and Day 15. The change from baseline will be summarized for Day 6 and Day 15. All lab parameters will be summarized in standard SI units.

All lab results from Baseline, Day 6, and Day 15 will be listed.

#### 9.6.5 Vital Signs

Vital signs will be collected for Days 1 - 6 of the study.

Descriptive summary statistics will be presented for the highest and lowest measurements by study day for each vital sign parameter: pulse rate (per minute), respiration rate (per minute), systolic and diastolic blood pressure (mm Hg), and temperature (°C). A descriptive summary of weight (kg) will also be presented. These tables will include the absolute values and the change from baseline. See Section 5 for the definition of baseline.

#### 9.6.6 Physical Examinations, ECGs, and Other Observations Related to Safety

The number and percentage of subjects with normal or abnormal physical examination findings will be presented by visit, body system (e.g. skin, HEENT, etc.) and treatment group.

Post-baseline physical examination abnormalities will be listed to provide details of the noted abnormalities.

ECGs will be performed at Day 1 prior to the initiation of study treatment and at Day 6



(post-infusion).

Abnormal rhythm, conduction, and QRS complex findings will be summarized by study day and treatment group for the safety population. Subjects with abnormal and clinically significant, abnormal post-baseline results will be listed.

#### 9.6.6.1 Arterial Blood Gases

Arterial blood gases (PaO<sub>2</sub>, PaCO<sub>2</sub>, HCO<sub>3</sub>, pH, SaO<sub>2</sub> and FiO<sub>2</sub>) will be recorded before randomization (Day 1 pre-dose) and once daily during Days 1 – 6.

Descriptive summary statistic tables will be presented for the worst daily ABG parameters by treatment group and measurement day. These tables will include the absolute values and the change from baseline. The worst value will be calculated as the lowest value of the day for PaO2, HCO3, pH, SaO2, and FiO2 and the highest value of the day for PaCO2. See Section 5 for the definition of baseline and guidance on how to handle repeat observations at a given visit.

#### 9.6.7 Progesterone Levels

A descriptive summary of Day 2 progesterone levels will be presented by treatment group.

#### 10 VALIDATION

PRA Analysis and Reporting seeks to ensure the quality of the results provided for the study in the form of tables, figures, and listings (TFLs), and the derived datasets used in their creation, through the following processes:

- Derived datasets will be independently reprogrammed by a second programmer. The separate datasets produced by the two programmers must match 100%.
- Tables will be independently reprogrammed by a second programmer for numeric results. Statisticians will be involved in the process of programming and validating tables that include inferential statistical results.
- Figures will be checked for consistency against corresponding tables and listings, or independently reprogrammed if there are no corresponding tables or listings.
- Listings will be checked for consistency against corresponding tables, figures, and derived datasets.

The entire set of TFLs will be checked for completeness and consistency prior to its delivery to the sponsor by the lead analysis programmer, the lead statistician, and a senior level statistician, or above, who is not a member of the project team.

The PRA validation process will be repeated any time TFLs are redelivered using different data. Execution of this validation process will be documented through the study Table of Programs that will be provided to the sponsor at study conclusion.

#### 11 REFERENCES

Agresti A. An introduction to Categorical Data Analysis. Wiley Series. 1996.

Allison P. Logistic Regression using the SAS System. Cary, NC: SAS Institute Inc.; 1999.

CPMP/EWP/2863/99 (Points to Consider on Adjustment for Baseline Covariates).



Ellenberg SS, Fleming TR, De Mets DL. *Data Monitoring Committees in Clinical Trials A Practical Perspective*. John Wiley & Sons; 2002.

Gardner M, Altman D. *Statistics with Confidence – Confidence intervals and statistical guidelines.* London: BMJ; 1989.

Hukkelhoven CWPM, Steyerberg EW, Habbema JDF, et al. Predicting outcome after traumatic brain injury: development and validation of a prognostic score based on admission characteristics. *Journal of Neurotrauma* 2005: 22: 1025 – 1039.

ICH Guideline E9.

Lee Y J, Quan H. P-values after repeated significance testing: a simple approximation method *Statistics in Medicine* 1993: 12: 675-84.

Lu, Juan. Unpublished data from IMPACT database. 2011.

Maas AI R, Murray G, Henney H, et al. Efficacy and safety of dexanabinol in severe traumatic brain injury: results of a phase III randomised, placebo-controlled, clinical trial. *Lancet Neurol.* 2006; 5: 38-45.

Mccullagh P, Nelder JA. Generalized Linear Models. 1st ed. London: Chapman and Hall; 1983.

Proschan MA, Lan KKG, Wittes JT. *Statistical monitoring of clinical trials: a unified approach*. New York, NY: Springer; 2006.

Walker G. Common Statistical Methods for Clinical Research. Cary, NC: SAS Institute Inc.; 2002.

Whitehead J. *The Design and Analysis of Sequential Clinical Trials*. Statistics in Practice. 1997.



# APPENDIX 1 GLOSSARY OF ABBREVIATIONS

ABG Arterial Blood Gases

ABIC American Brain Injury Consortium

AE Adverse Event

ANCOVA Analysis of Covariance

BHR-100 BHR Pharma, LLC's proprietary formulation of intravenous

progesterone

BP Blood Pressure

BPRS Baseline Prognostic Risk Score

BTF Brain Trauma Foundation

CI Confidence Interval

CMH Cochran-Mantel Haenszel

CPP Cerebral Perfusion Pressure

CRF Case Report Form (paper or other media)

CSR Clinical Study Report

CT Computed Tomography

DMAP Data Monitoring and Analysis Plan

DMP Data Management Plan

DP Decimal Places

DSMB Data Safety Monitoring Board

EBIC European Brain Injury Consortium

ECG Electrocardiogram

FDA Food and Drug Administration

FiO<sub>2</sub> Fraction of Inspired Oxygen

GCS Glasgow Coma Scale

GOS Glasgow Outcome Scale

GOS-E Extended Glasgow Outcome Scale

HCO<sub>3</sub> Bicarbonate
HR Hazard Ratio

ICH International Conference on Harmonisation of Technical

Requirements for Registration of Pharmaceuticals for Human Use


ICP Intracranial Pressure
ICU Intensive Care Unit

IMPACT International Mission for Prognosis and Analysis of Clinical

Trials in TBI

ITT Intent-to-treat

i.v. Intravenous

IWRS Interactive Web-based Randomization System

LOCF Last Observation Carried Forward

MAP Mean Arterial Pressure

MedDRA Medical Dictionary for Regulatory Activities

mITT Modified Intention-to-treat

OR Odds Ratio

PaO<sub>2</sub> Partial Pressure of Oxygen

PaCO<sub>2</sub> Partial Pressure of Carbon Dioxide

POM Proportional Odds Model

PP Per Protocol
Q1 First Quartile
Q3 Third Quartile

SAE Serious Adverse Event
SAP Statistical Analysis Plan

SaO<sub>2</sub> Saturation of Oxygen, arterial blood

SD Sliding Dichotomy

SF-36 Short Form 36 Health Survey

SOC System Organ Class
TBI Traumatic Brain Injury

TEAE Treatment-Emergent Adverse Events

TFL Tables, Figures and Listings

TIL Therapy Intensity Level

WHO-DD World Health Organization-Drug Dictionary



# APPENDIX 2 LIST OF POST-TEXT TABLES, FIGURES, LISTINGS, AND SUPPORTIVE SAS OUTPUT APPENDICES

#### **Tables**

| Output | Title | Use<br>Table<br>Shell | DSMB* |
|---|---|---|---|
| Table 14.1.1.1 | Summary of Investigational Sites' Enrollment Duration (mITT Population) | | X |
| Table 14.1.1.2 | Summary of Enrollment by Region, Country and Site (mITT Population) | | X |
| Table 14.1.1.3 | Summary of Subject Disposition (Randomized Subjects) | | X |
| Table 14.1.1.4 | Summary of Subject Status by Time (mITT Population) | | |
| Table 14.1.1.5 | Country Codes per ISO | | |
| Table 14.1.2.1 | Summary of Study Drug Exposure and Time From Injury (Safety Population) | | X |
| Table 14.1.2.2 | Drug Administration Summary (Safety Population) | | |
| Table 14.1.2.3 | Summary of Study Drug Compliance Rate (Safety Population) | | |
| Table 14.1.3.1 | Prior and Concomitant Medications by WHO Drug Dictionary<br>Preferred Term (mITT Population) | | |
| Table 14.1.3.2 | Surgical Therapy (mITT Population) | | |
| Table 14.1.4.1 | Demographic Characteristics (mITT Population) | | X |
| Table 14.1.4.2 | Pregnancy Testing (mITT Population) | | X |
| Table 14.1.4.3 | Baseline Characteristics (mITT Population) | | X |
| Table 14.1.4.4 | Summary of Injury (mITT Population) | | |
| Table 14.1.5 | Summary of Medical History by System Organ Class and Preferred Term (Safety Population) | | |
| Table 14.2.1.1 | Summary of Glasgow Outcome Scale at 6 Months Post Injury – Missing Values Imputed (mITT Population) | | X |
| Table 14.2.1.2 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury – Proportional Odds Model - Missing Values Imputed (mITT Population) | | X |
| Table 14.2.1.3 | ORs and 95% CIs of Glasgow Outcome Scale at 6 Months Post<br>Injury – Proportional Odds Model - Missing Values Imputed (mITT<br>Population) | | X |
| Table 14.2.1.4 | Summary of Glasgow Outcome Scale at 6 Months Post Injury –<br>Observed Values (mITT Population) | 14.2.1.1 | X |
| Table 14.2.1.5 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury –<br>Proportional Odds Model - Observed Values (mITT Population) | 14.2.1.2 | X |





| Output | Title | Use<br>Table<br>Shell | DSMB* |
|---|---|---|---|
| Table 14.2.1.6 | ORs and 95% CIs of Glasgow Outcome Scale at 6 Months Post<br>Injury – Proportional Odds Model - Observed Values (mITT<br>Population) | 14.2.1.3 | X |
| Table 14.2.1.7 | Summary of Glasgow Outcome Scale at 6 Months Post Injury – Observed Values (PP Population) | 14.2.1.1 | |
| Table 14.2.1.8 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury –<br>Proportional Odds Model - Observed Values (PP Population) | 14.2.1.2 | |
| Table 14.2.1.9 | ORs and 95% CIs of Glasgow Outcome Scale at 6 Months Post<br>Injury – Proportional Odds Model - Observed Values (PP<br>Population) | 14.2.1.3 | |
| Table 14.2.1.10 | Summary of Glasgow Outcome Scale at 6 Months Post Injury for US<br>Only – Missing Values Imputed (mITT Population) | 14.2.1.1 | |
| Table 14.2.1.11 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury for US<br>Only – Proportional Odds Model - Missing Values Imputed (mITT<br>Population) | 14.2.1.2 | |
| Table 14.2.1.12 | ORs and 95% CIs of Glasgow Outcome Scale at 6 Months Post<br>Injury for US Only – Proportional Odds Model - Missing Values<br>Imputed (mITT Population) | 14.2.1.3 | |
| Table 14.2.1.13 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury –<br>Proportional Odds Model - Missing Values Imputed (Unadjusted<br>Analysis) (mITT Population) | 14.2.1.2 | |
| Table 14.2.1.14 | ORs and 95% CIs of Glasgow Outcome Scale at 6 Months Post<br>Injury – Proportional Odds Model - Missing Values Imputed<br>(Unadjusted Analysis) (mITT Population) | 14.2.1.3 | |
| Table 14.2.2.1 | Summary of Sliding Dichotomy (Dichotomization) – Missing Values Imputed (mITT Population) | | |
| Table 14.2.2.2 | Summary and Analysis of Sliding Dichotomy at 6 Months Post<br>Injury – Missing Values Imputed (mITT Population) | | |
| Table 14.2.2.3 | ORs and 95% CIs for Sliding Dichotomy at 6 Months Post Injury – Missing Values Imputed (mITT Population) | | |
| Table 14.2.2.4 | Summary of Sliding Dichotomy (Dichotomization) at 6 Months Post<br>Injury – Observed Values (mITT Population) | 14.2.2.1 | |
| Table 14.2.2.5 | Summary and Analysis of Sliding Dichotomy at 6 Months Post<br>Injury – Observed Values (mITT Population) | 14.2.2.2 | |
| Table 14.2.2.6 | ORs and 95% CIs for Sliding Dichotomy at 6 Months Post Injury – Observed Values (mITT Population) | 14.2.2.3 | |
| Table 14.2.2.7 | Summary of Sliding Dichotomy (Dichotomization) at 6 Months Post<br>Injury – Observed Values (PP Population) | 14.2.2.1 | |
| Table 14.2.2.8 | Summary and Analysis of Sliding Dichotomy at 6 Months Post<br>Injury – Observed Values (PP Population) | 14.2.2.2 | |
| Table 14.2.2.9 | ORs and 95% CIs for Sliding Dichotomy at 6 Months Post Injury – Observed Values (PP Population) | 14.2.2.3 | |



| Output | Title | Use<br>Table<br>Shell | DSMB* |
|---|---|---|---|
| Table 14.2.2.10 | Summary of Sliding Dichotomy (Dichotomization) at 6 Months Post<br>Injury for US Only – Missing Values Imputed (mITT Population) | 14.2.2.1 | |
| Table 14.2.2.11 | Summary and Analysis of Sliding Dichotomy at 6 Months Post<br>Injury for US Only – Missing Values Imputed (mITT Population) | 14.2.2.2 | |
| Table 14.2.2.12 | ORs and 95% CIs for Sliding Dichotomy at 6 Months Post Injury for US Only – Missing Values Imputed (mITT Population) | 14.2.2.3 | |
| Table 14.2.3.1 | Summary of Dichotomized Glasgow Outcome Scale at 6 Months<br>Post Injury – Missing Values Imputed (mITT Population) | | X |
| Table 14.2.3.2 | Analysis of Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome<br>Scale at 6 Months Post Injury – Missing Values Imputed (mITT<br>Population) | | |
| Table 14.2.3.3 | ORs and 95% CIs for Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome Scale at 6 Months Post Injury – Missing Values Imputed (mITT Population) | | |
| Table 14.2.3.4 | Summary of Dichotomized Glasgow Outcome Scale at 6 Months<br>Post Injury – Observed Values (mITT Population) | 14.2.3.1 | |
| Table 14.2.3.5 | Analysis of Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome<br>Scale at 6 Months Post Injury – Observed Values (mITT Population) | 14.2.3.2 | |
| Table 14.2.3.6 | ORs and 95% CIs for Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome Scale at 6 Months Post Injury – Observed Values (mITT Population) | 14.2.3.3 | |
| Table 14.2.3.7 | Summary of Dichotomized Glasgow Outcome Scale at 6 Months<br>Post Injury – Observed Values (PP Population) | 14.2.3.1 | |
| Table 14.2.3.8 | Analysis of Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome<br>Scale at 6 Months Post Injury – Observed Values (PP Population) | 14.2.3.2 | |
| Table 14.2.3.9 | ORs and 95% CIs for Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome Scale at 6 Months Post Injury – Observed Values (PP Population) | 14.2.3.3 | |
| Table 14.2.3.10 | Analysis of Dichotomized (GR vs. MD, SD, V/D) Glasgow Outcome<br>Scale at 6 Months Post Injury – Missing Values Imputed (mITT<br>Population) | 14.2.3.2 | |
| Table 14.2.3.11 | ORs and 95% CIs for Dichotomized (GR vs. MD, SD, V/D) Glasgow Outcome Scale at 6 Months Post Injury – Missing Values Imputed (mITT Population) | 14.2.3.3 | |
| Table 14.2.3.12 | Analysis of Dichotomized (GR, MD, SD vs. V/D) Glasgow Outcome<br>Scale at 6 Months Post Injury – Missing Values Imputed (mITT<br>Population) | 14.2.3.2 | |
| Table 14.2.3.13 | ORs and 95% CIs for Dichotomized (GR, MD, SD vs. V/D) Glasgow Outcome Scale at 6 Months Post Injury – Missing Values Imputed (mITT Population) | 14.2.3.3 | |
| Table 14.2.4.1 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury – Exploratory Analysis – Missing Values Imputed (mITT Population) | | |



| Output | Title | Use<br>Table<br>Shell | DSMB* |
|---|---|---|---|
| Table 14.2.4.2 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury by<br>Region – Exploratory Analysis – Missing Values Imputed (mITT<br>Population) | | |
| Table 14.2.4.3 | ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post<br>Injury by Region – Exploratory Analysis – Missing Values Imputed<br>(mITT Population) | | |
| Table 14.2.4.4 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury by Age<br>Group – Exploratory Analysis – Missing Values Imputed (mITT<br>Population) | | |
| Table 14.2.4.5 | ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post<br>Injury by Age Group – Exploratory Analysis – Missing Values<br>Imputed (mITT Population) | | |
| Table 14.2.4.6 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury by Race<br>Group – Exploratory Analysis – Missing Values Imputed (mITT<br>Population) | | |
| Table 14.2.4.7 | ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post<br>Injury by Race Group – Exploratory Analysis – Missing Values<br>Imputed (mITT Population) | | |
| Table 14.2.4.8 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury by GCS<br>Motor Score – Exploratory Analysis – Missing Values Imputed<br>(mITT Population) | | |
| Table 14.2.4.9 | ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post<br>Injury by GCS Motor Score – Exploratory Analysis – Missing Values<br>Imputed (mITT Population) | | |
| Table 14.2.4.10 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury by<br>Pupil Response – Exploratory Analysis – Missing Values Imputed<br>(mITT Population) | | |
| Table 14.2.4.11 | ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post<br>Injury by Pupil Response – Exploratory Analysis – Missing Values<br>Imputed (mITT Population) | | |
| Table 14.2.4.12 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury by CT<br>Classification – Exploratory Analysis – Missing Values Imputed<br>(mITT Population) | | |
| Table 14.2.4.13 | ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post<br>Injury by CT Classification – Exploratory Analysis – Missing Values<br>Imputed (mITT Population) | | |
| Table 14.2.4.14 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury by<br>Presence of Hypoxia– Exploratory Analysis – Missing Values<br>Imputed (mITT Population) | | |
| Table 14.2.4.15 | ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post<br>Injury by Presence of Hypoxia – Exploratory Analysis – Missing<br>Values Imputed (mITT Population) | | |





| Output | Title | Use<br>Table<br>Shell | DSMB* |
|---|---|---|---|
| Table 14.2.4.16 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury by<br>Presence of Hypotension– Exploratory Analysis – Missing Values<br>Imputed (mITT Population) | | |
| Table 14.2.4.17 | ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post<br>Injury by Presence of Hypotension – Exploratory Analysis – Missing<br>Values Imputed (mITT Population) | | |
| Table 14.2.4.18 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury by Presence of Traumatic Subarachnoid Hemorrhage– Exploratory Analysis – Missing Values Imputed (mITT Population) | | |
| Table 14.2.4.19 | ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post<br>Injury by Presence of Traumatic Subarachnoid Hemorrhage –<br>Exploratory Analysis – Missing Values Imputed (mITT Population) | | |
| Table 14.2.4.20 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury by<br>Gender – Exploratory Analysis – Missing Values Imputed (mITT<br>Population) | | |
| Table 14.2.4.21 | ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post<br>Injury by Gender – Exploratory Analysis – Missing Values Imputed<br>(mITT Population) | | |
| Table 14.2.4.22 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury by<br>Time to First Dose – Exploratory Analysis – Missing Values Imputed<br>(mITT Population) | | |
| Table 14.2.4.23 | ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post<br>Injury by Time to First Dose – Exploratory Analysis – Missing<br>Values Imputed (mITT Population) | | |
| Table 14.2.5.1 | Summary and Analysis of Mortality at Month 6 (mITT Population) | | X |
| Table 14.2.5.2 | Summary and Analysis of Mortality at Month 1 (mITT Population) | 14.2.5.1 | X |
| Table 14.2.5.3 | Summary and Analysis of Mortality at Month 6 (PP Population) | 14.2.5.1 | X |
| Table 14.2.5.4 | Summary and Analysis of Mortality at Month 1 (PP Population) | 14.2.5.1 | X |
| Table 14.2.5.5 | Summary and Kaplan-Meier Analysis of Time to Death (days) (mITT Population) | | |
| Table 14.2.5.6 | Summary of Cox Proportional Hazards Analysis of Time to Death (days) (mITT Population) | | |
| Table 14.2.6.1 | Summary of Glasgow Outcome Scale at 3 Months Post Injury – Observed Values (mITT Population) | 14.2.1.1 | |
| Table 14.2.6.2 | Analysis of Glasgow Outcome Scale at 3 Months Post Injury –<br>Proportional Odds Model - Observed Values (mITT Population) | 14.2.1.2 | |
| Table 14.2.6.3 | ORs and CIs of Glasgow Outcome Scale at 3 Months Post Injury – Proportional Odds Model - Observed Values (mITT Population) | 14.2.1.3 | |
| Table 14.2.7.1 | Summary of Glasgow Outcome Scale - Extended at 6 Months Post<br>Injury – Observed Values (mITT Population) | 14.2.1.1 | |





| Output | Title | Use<br>Table<br>Shell | DSMB* |
|---|---|---|---|
| Table 14.2.7.2 | Analysis of Glasgow Outcome Scale – Extended at 6 Months Post<br>Injury – Proportional Odds Model - Observed Values (mITT<br>Population) | 14.2.1.2 | |
| Table 14.2.7.3 | ORs and CIs of Glasgow Outcome Scale - Extended at 6 Months Post<br>Injury – Proportional Odds Model - Observed Values (mITT<br>Population) | 14.2.1.3 | |
| Table 14.2.7.4 | Summary of Sliding Dichotomy (Dichotomization) – Glasgow<br>Outcome Scale – Extended at 6 Months Post Injury – Observed<br>Values (mITT Population) | | |
| Table 14.2.7.5 | Summary and Analysis of Sliding Dichotomy – Glasgow Outcome<br>Scale – Extended at 6 Months Post Injury – Observed Values (mITT<br>Population) | | |
| Table 14.2.7.6 | ORs and 95% CIs for Sliding Dichotomy – Glasgow Outcome Scale – Extended at 6 Months Post Injury – Observed Values (mITT Population) | | |
| Table 14.2.7.7 | Summary of Glasgow Outcome Scale - Extended at 3 Months Post<br>Injury - Observed Values (mITT Population) | | |
| Table 14.2.7.8 | Analysis of Glasgow Outcome Scale – Extended at 3 Months Post<br>Injury – Proportional Odds Model - Observed Values (mITT<br>Population) | | |
| Table 14.2.7.9 | ORs and CIs of Glasgow Outcome Scale - Extended at 3 Months Post<br>Injury – Proportional Odds Model - Observed Values (mITT<br>Population) | | |
| Table 14.2.8.1 | Summary of SF-36 by Visit (mITT Population) | | |
| Table 14.2.8.2 | Analysis of SF-36 by Visit (mITT Population) | | |
| Table 14.2.9 | Shift Summary of CT Classification (mITT Population) | | |
| Table 14.2.10 | Summary of Maximum Intracranial Pressure by Visit (mITT Population) | | |
| Table 14.2.11.1 | Summary of Cerebral Perfusion Pressure by Visit (mITT Population) | | |
| Table 14.2.11.2 | Potentially Clinically Important On-Treatment Cerebral Perfusion<br>Pressure (mITT Population) | | |
| Table 14.2.12.1 | Summary of Therapy Intensity Level by Visit (mITT Population) | | |
| Table 14.2.12.2 | Summary of Individual TIL Therapies (mITT Population) | | |
| Table 14.2.12.3 | Summary of Maximum Therapy Intensity Level (mITT Population) | | |
| Table 14.3.1.1 | Overall Summary of Treatment Emergent Adverse Events (Safety Population) | | X |
| Table 14.3.1.2 | Overall Summary of Treatment Emergent Adverse Events by Gender (Safety Population) | | |
| Table 14.3.1.3 | Overall Summary of Treatment Emergent Adverse Events by Race<br>Group (Safety Population) | 14.3.1.2 | |



| Output | Title | Use<br>Table<br>Shell | DSMB* |
|---|---|---|---|
| Table 14.3.1.4 | Overall Summary of Treatment Emergent Adverse Events by Age<br>Group (Safety Population) | 14.3.1.2 | |
| Table 14.3.1.5 | Treatment Emergent Adverse Events by System Organ Class and<br>Preferred Term (Safety Population) | | X |
| Table 14.3.1.6 | Treatment Emergent Adverse Events by System Organ Class,<br>Preferred Term, and Gender (Safety Population) | | |
| Table 14.3.1.7 | Treatment Emergent Adverse Events by System Organ Class,<br>Preferred Term, and Race Group (Safety Population) | | |
| Table 14.3.1.8 | Treatment Emergent Adverse Events by System Organ Class,<br>Preferred Term, and Age Group (Safety Population) | | |
| Table 14.3.1.9 | Treatment-Related Treatment Emergent Adverse Events by System<br>Organ Class and Preferred Term (Safety Population) | 14.3.1.5 | X |
| Table 14.3.1.10 | Treatment Emergent Adverse Events by Maximum Severity, System Organ Class and Preferred Term (Safety Population) | | |
| Table 14.3.1.11 | Treatment-Related Treatment Emergent Adverse Events by<br>Maximum Severity, System Organ Class and Preferred Term (Safety<br>Population) | 14.3.1.9 | |
| Table 14.3.1.12 | Treatment Emergent Adverse Events by Maximum Relationship,<br>System Organ Class and Preferred Term (Safety Population) | | |
| Table 14.3.1.13 | Treatment Emergent Adverse Events Leading to Premature Discontinuation of Study Drug by System Organ Class and Preferred Term (Safety Population) | 14.3.1.5 | |
| Table 14.3.1.14 | Treatment-Related Treatment Emergent Adverse Events Leading to<br>Premature Discontinuation of Study Drug by System Organ Class<br>and Preferred Term (Safety Population) | 14.3.1.5 | |
| Table 14.3.1.15 | Treatment Emergent Adverse Events of Special Interest (Safety Population) | | X |
| Table 14.3.1.16 | List of Adverse Events of Special Interest (Safety Population) | | X |
| Table 14.3.2.1 | Serious Adverse Events by System Organ Class and Preferred Term (Safety Population) | 14.3.1.5 | X |
| Table 14.3.2.2 | Treatment-Related Serious Adverse Events by System Organ Class and Preferred Term (Safety Population) | 14.3.1.5 | X |
| Table 14.3.2.3 | Primary Cause of Death (mITT Population) | | X |
| Table 14.3.4.1 | Post-Baseline Abnormal, Clinically Significant (non-AE) Laboratory<br>Test Results: Coagulation (Safety Population) | | X |
| Table 14.3.4.2 | Post-Baseline Abnormal, Clinically Significant (non-AE) Laboratory<br>Test Results: Hematology (Safety Population) | 14.3.4.1 | X |
| Table 14.3.4.3 | Post-Baseline Abnormal, Clinically Significant (non-AE) Laboratory<br>Test Results: Serum Chemistry (Safety Population) | 14.3.4.1 | |



| Output | Title | Use<br>Table<br>Shell | DSMB* |
|---|---|---|---|
| Table 14.3.4.4 | Post-Baseline Abnormal, Clinically Significant (non-AE) Laboratory<br>Test Results: Urinalysis (Safety Population) | | |
| Table 14.3.4.5 | List of Post-Baseline Abnormal, Clinically Significant (non-AE)<br>Laboratory Test Results: Coagulation (Safety Population) | 14.3.4.9 | X |
| Table 14.3.4.6 | List of Post-Baseline Abnormal, Clinically Significant (non-AE)<br>Laboratory Test Results: Hematology (Safety Population) | | X |
| Table 14.3.4.7 | List of Post-Baseline Abnormal, Clinically Significant (non-AE)<br>Laboratory Test Results: Serum Chemistry (Safety Population) | 14.3.4.9 | X |
| Table 14.3.4.8 | List of Post-Baseline Abnormal, Clinically Significant (non-AE)<br>Laboratory Test Results: Urinalysis (Safety Population) | 14.3.4.9 | X |
| Table 14.3.4.9 | Summary of Coagulation Laboratory Test Results (Safety Population) | | |
| Table 14.3.4.10 | Summary of Hematology Laboratory Test Results (Safety Population) | 14.3.4.12 | |
| Table 14.3.4.11 | Summary of Serum Chemistry Laboratory Test Results (Safety Population) | 14.3.4.12 | |
| Table 14.3.5 | Summary of Incidence of Neuroworsening (Safety Population) | | |
| Table 14.3.6.1 | Summary of Vital Signs Corresponding to Lowest Measurement (Safety Population) | | X |
| Table 14.3.6.2 | Summary of Vital Signs Corresponding to Highest Measurement (Safety Population) | 14.3.5.1 | X |
| Table 14.3.6.3 | Summary of Vital Signs by Visit – Weight (kg) (Safety Population) | | |
| Table 14.3.7.1 | Summary of Physical Examination by Visit (Safety Population) | | |
| Table 14.3.7.2 | List of Physical Examination Abnormalities Post-Baseline (Safety Population) | | |
| Table 14.3.8.1 | Post-Baseline Abnormal ECG Results (Safety Population) | | X |
| Table 14.3.8.2 | List of Post-Baseline Abnormal ECG Results – Part 1 and Part 2 (Safety Population) | | X |
| Table 14.3.9 | Summary of Worst Arterial Blood Gas (ABG) Results by Visit (Safety Population) | | X |
| 14.3.10 | Summary of Day 2 Progesterone Levels (Safety Population) | | |

# \* Tables produced for DSMB

## **Figures**

| Figure | Title | DSMB* |
|---|---|---|
| Figure 14.2.1.1 | Glasgow Outcome Scale distribution at 6 Months Post Injury – Missing Values Imputed (mITT Population) | X |

 $a_{\scriptscriptstyle \overline{ ext{Version Date: 2.0 April 19, 2014}}}$ 

| Figure | Title | DSMB* |
|---|---|---|
| Figure 14.2.1.2 | Glasgow Outcome Scale distribution at 6 Months Post Injury – Observed Values (mITT Population) | X |
| Figure 14.2.1.3 | Glasgow Outcome Scale distribution at 6 Months Post Injury – Observed Values (PP Population) | |
| Figure 14.2.2.1 | Dichotomized Glasgow Outcome Scale at 6 Months Post Injury – Missing Values Imputed (mITT Population) | |
| Figure 14.2.2.2 | Dichotomized Glasgow Outcome Scale at 6 Months Post Injury – Observed Values (mITT Population) | |
| Figure 14.2.3.1 | Mortality at 6 Months (mITT Population) | X |
| Figure 14.2.3.2 | Mortality at 1 Month (mITT Population) | X |
| Figure 14.2.3.3 | Time to Death (mITT Population) | |

# \* Figures produced for DSMB

## **Data Listings**

| Listing | Title | DSMB* |
|---|---|---|
| Listing 16.2.1.1 | Study Completion/Discontinuation Details | |
| Listing 16.2.1.2 | Eligibility/Randomization | |
| Listing 16.2.1.3 | Exclusions from Per Protocol Population | |
| Listing 16.2.3.1 | Subject General Information | X |
| Listing 16.2.3.2 | Informed Consent | |
| Listing 16.2.4.1 | Demographic Characteristics | X |
| Listing 16.2.4.2 | Baseline Characteristics | X |
| Listing 16.2.4.3 | Pre-injury Narrative – Baseline Status – Parts 1, 2 and 3 | |
| Listing 16.2.4.4 | Glasgow Coma Scale | |
| Listing 16.2.4.5 | Medical History | |
| Listing 16.2.4.6 | Prior, and Concomitant Medications | |
| Listing 16.2.4.7 | Concomitant Procedures | |
| Listing 16.2.4.8 | Surgical Therapy | |
| Listing 16.2.4.9 | Study Admission | |
| Listing 16.2.4.10 | Subject Transfer | |
| Listing 16.2.4.11 | Facility Transfer | |
| Listing 16.2.4.12 | Intubation | |
| Listing 16.2.4.13 | Daily Fluid | |
| Listing 16.2.5.1 | Study Drug Administration Parts 1 and 2 | X |
| Listing 16.2.5.2 | End of Treatment | X |



Listing Title DSMB\* Listing 16.2.6.1.1 X Glasgow Outcome Scale, Questions Listing 16.2.6.1.2 Glasgow Outcome Scale, Explanation of Categories X Glasgow Outcome Scale – Extended, Explanation of Categories Listing 16.2.6.1.3 Listing 16.2.6.1.4 Glasgow Outcome Scale - Part 1 X Listing 16.2.6.1.5 Glasgow Outcome Scale, Glasgow Outcome Scale-Extended Narrative – Parts 1-6 Listing 16.2.6.1.6 Primary Efficacy, Covariates, and Subgroup Variables (Observed Values) X X Primary Efficacy, Covariates, and Subgroup Variables (Missing Values Listing 16.2.6.1.7 Imputed) Listing 16.2.6.2 Sliding Dichotomy Listing 16.2.6.3 Mortality X SF-36, Explanation of Categories Listing 16.2.6.4.1 SF-36 (Individual Questions) - Parts 1, 2 and 3 Listing 16.2.6.4.2 Listing 16.2.6.4.3 SF-36 (Scales and Summary Scores) - Parts 1 and 2 CT Scan and Classification - Parts 1, 2 and 3 Listing 16.2.6.5.1 CT Scan Comparison - Parts 1, 2 and 3 Listing 16.2.6.5.2 Intracranial Pressure Listing 16.2.6.6.1 Listing 16.2.6.6.2 **Intracranial Pressure Monitoring** Cerebral Perfusion Pressure Listing 16.2.6.7 Listing 16.2.6.8.1 Therapy Intensity Level Parts 1 and 2 Listing 16.2.7 Adverse Events X Listing 16.2.8.1.1 Laboratory (Coagulation) Results Listing 16.2.8.1.2 Laboratory (Hematology) Results Listing 16.2.8.1.3 Laboratory (Serum Chemistry) Results Listing 16.2.8.1.4 Laboratory (Urinalysis) Results Laboratory (Pregnancy Test) Results Listing 16.2.8.1.5 Listing 16.2.8.2 Vital Signs X Listing 16.2.8.3 Physical Examinations Listing 16.2.8.4 12-Lead Electrocardiogram (ECG) Parts 1 and 2

### \* Listings produced for DSMB

Listing 16.2.8.5
Listing 16.2.8.6

Note: Listings generated for all mITT subjects.

Arterial Blood Gas

Neuroworsening Parts 1 and 2

X



## **Statistical Output**

| Appendix | Title |
|---|---|
| Appendix 14.2.1.2 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury – Missing Values Imputed (mITT Population)* |
| The above appendix will in ORs and CIs). | clude the SAS output details relating to Table 14.2.1.2 and 14.2.1.3 (Analysis, |
| Appendix 14.2.1.5 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury – Observed Values (mITT Population) |
| The above appendix will in ORs and CIs). | clude the SAS output details relating to Table 14.2.1.5 and 14.2.1.6 (Analysis, |
| Appendix 14.2.1.8 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury – Observed Values (PP Population) |
| The above appendix will in ORs and CIs). | clude the SAS output details relating to Table 14.2.1.8 and 14.2.1.9 (Analysis, |
| Appendix 14.2.1.11 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury for US Only – Missing Values Imputed (mITT Population) |
| The above appendix will in ORs and CIs). | include the SAS output details relating to Table 14.2.1.11 and 14.2.1.12 (Analysis, |
| Appendix 14.2.1.13 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury– Missing Values Imputed (Unadjusted Analysis) (mITT Population) |
| The above appendix will in ORs and CIs). | clude the SAS output details relating to Table 14.2.1.13 and 14.2.1.14 (Analysis, |
| Appendix 14.2.2.2 | Summary and Analysis of Sliding Dichotomy at 6 Months Post Injury – Missing Values Imputed (mITT Population) |
| Appendix 14.2.2.5 | Summary and Analysis of Sliding Dichotomy at 6 Months Post Injury – Observed Values (mITT Population) |
| Appendix 14.2.2.8 | Summary and Analysis of Sliding Dichotomy at 6 Months Post Injury – Observed Values (PP Population) |
| Appendix 14.2.2.11 | Summary and Analysis of Sliding Dichotomy at 6 Months Post Injury for US Only – Missing Values Imputed (mITT Population) |
| Appendix 14.2.3.2 | Analysis of Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome Scale at 6<br>Months Post Injury – Missing Values Imputed (mITT Population) |
| The above appendix will in ORs and CIs). | clude the SAS output details relating to Table 14.2.3.2 and 14.2.3.3 (Analysis, |
| Appendix 14.2.3.5 | Analysis of Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome Scale at 6<br>Months Post Injury – Observed Values (mITT Population) |
| The above appendix will in ORs and CIs). | clude the SAS output details relating to Table 14.2.3.5 and 14.2.3.6 (Analysis, |
| Appendix 14.2.3.8 | Analysis of Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome Scale at 6<br>Months Post Injury – Observed Values (PP Population) |
| The above appendix will in ORs and CIs). | clude the SAS output details relating to Table 14.2.3.8 and 14.2.3.9 (Analysis, |



| Appendix | Title |
|---|---|
| Appendix 14.2.3.10 | Analysis of Dichotomized (GR vs. MD, SD, V/D) Glasgow Outcome Scale at 6<br>Months Post Injury – Missing Values Imputed (mITT Population) |
| The above appendix will ORs and CIs). | ll include the SAS output details relating to Table 14.2.3.10 and 14.2.3.11 (Analysis, |
| Appendix 14.2.3.12 | Analysis of Dichotomized (GR, MD, SD vs. V/D) Glasgow Outcome Scale at 6<br>Months Post Injury – Observed Values (mITT Population) |
| The above appendix will ORs and CIs). | ll include the SAS output details relating to Table 14.2.3.12 and 14.2.3.13 (Analysis, |
| Appendix 14.2.4.1 | Analysis of Glasgow Outcome Scale at 6 Months Post Injury – Exploratory Analysis – Missing Values Imputed (mITT Population) |
| The above appendix wi | ll include the SAS output details relating to Table 14.2.4.1 (Analysis, ORs and CIs). |
| Appendix 14.2.5.1 | Summary and Analysis of Mortality at Month 6 (mITT Population) |
| Appendix 14.2.5.2 | Summary and Analysis of Mortality at Month 1 (mITT Population) |
| Appendix 14.2.5.3 | Summary and Analysis of Mortality at Month 6 (PP Population) |
| Appendix 14.2.5.4 | Summary and Analysis of Mortality at Month 1 (PP Population) |
| Appendix 14.2.5.5 | Summary and Kaplan-Meier Analysis of Time to Death (days) (mITT Population) |
| Appendix 14.2.5.6 | Summary and Cox Proportional Hazards Analysis of Time to Death (days) (mITT Population) |
| Appendix 14.2.6.2 | Analysis of Glasgow Outcome Scale at 3 months post injury – Observed Values (mITT Population) |
| The above appendix will ORs and CIs). | ll include the SAS output details relating to Table 14.2.6.2 and 14.2.6.3 (Analysis, |
| Appendix 14.2.7.2 | Analysis of Glasgow Outcome Scale - Extended at 6 Months Post Injury – Observed Values (mITT Population) |
| The above appendix will ORs and CIs). | ll include the SAS output details relating to Table 14.2.7.2 and 14.2.7.3 (Analysis, |
| Appendix 14.2.7.5 | Summary and Analysis of Sliding Dichotomy – Glasgow Outcome Scale – Extended at 6 Months Post Injury – Observed Values (mITT Population) |
| Appendix 14.2.7.8 | Analysis of Glasgow Outcome Scale - Extended at 3 Months Post Injury – Observed Values (mITT Population) |
| Appendix 14.2.8.2 | Analysis of SF-36 by Visit (mITT Population) |



#### **Model Checking Figures**

| Figure 14.2.1.1.1 | Graphical Assessment of Proportional Odds Assumption for Proportional Odds Model of Glasgow Outcome Scale at 6 months [Treatment Group] – Missing Values Imputed (mITT Population) |
|---|---|
| Figure 14.2.1.1.2 | Graphical Assessment of Proportional Odds Assumption for Proportional Odds Model of Glasgow Outcome Scale at 6 months [Region] – Missing Values Imputed (mITT Population) |
| Figure 14.2.1.1.3 | Graphical Assessment of Proportional Odds Assumption for Proportional Odds Model of Glasgow Outcome Scale at 6 months [Age] – Missing Values Imputed (mITT Population) |
| Figure 14.2.1.1.4 | Graphical Assessment of Proportional Odds Assumption for Proportional Odds Model of Glasgow Outcome Scale at 6 months [GCS Motor Score] – Missing Values Imputed (mITT Population) |
| Figure 14.2.1.1.5 | Graphical Assessment of Proportional Odds Assumption for Proportional Odds Model of Glasgow Outcome Scale at 6 months [Pupil Response] – Missing Values Imputed (mITT Population) |
| Figure 14.2.1.1.6 | Graphical Assessment of Proportional Odds Assumption for Proportional Odds Model of Glasgow Outcome Scale at 6 months [CT Classification] – Missing Values Imputed (mITT Population) |



| Figure | 14.2.1.1.1 |
|---|---|
| Title 1 | Graphical Assessment of Proportional Odds Assumption for Proportional Odds Model of Glasgow Outcome Scale at 6 months – Missing Values Imputed [Treatment Group] (mITT Population) |
| Title 2 | Predictor = Treatment Group |
| Type of graph | Line graph |
| y-axis | Empirical Cumulative Logit |
| y-axis (label) | Empirical Cumulative Logit |
| x-axis | Treatment Group |
| x-axis (label) | Treatment Group |
| Legend (if applicable) | A legend should be included to identify each empirical cumulative logit $1 = \text{EmpLogit}_1 = \log[(y_1)/(y_2 + y_3 + y_4)]$ , $2 = \text{EmpLogit}_2 = \log[(y_1 + y_2)/(y_3 + y_4)]$ and $3 = \text{EmpLogit}_3 = \log[(y_1 + y_2 + y_3)/(y_4)]$ And treatment group: BHR-100 and Placebo |
| Footnote 1 | Program: xxxxxxx.sas, Output: xxxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x |
| Additional information | Corresponds to table 14.2.1.1. |

| Figure | 14.2.1.1.2 |
|---|---|
| Title 1 | Graphical Assessment of Proportional Odds Assumption for Proportional Odds Model of Glasgow Outcome Scale at 6 months Missing Values Imputed [Region] (mITT Population) |
| Title 2 | Predictor = Region |
| Type of graph | Line graph |
| y-axis | Empirical Cumulative Logit |
| y-axis (label) | Empirical Cumulative Logit |
| x-axis | Region |
| x-axis (label) | Region |
| Legend (if applicable) | A legend should be included to identify each empirical cumulative logit $1 = \text{EmpLogit}_1 = \log[(y_1)/(y_2 + y_3 + y_4)]$ , $2 = \text{EmpLogit}_2 = \log[(y_1 + y_2)/(y_3 + y_4)]$ and $3 = \text{EmpLogit}_3 = \log[(y_1 + y_2 + y_3)/(y_4)]$ And region: North America, Europe, Asia and South America |
| Footnote 1 | Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x |
| Additional information | Corresponds to table 14.2.1.1. |

| Figure | 14.2.1.1.3 |
|---|---|
| Title 1 | Graphical Assessment of Proportional Odds Assumption for Proportional Odds Model of Glasgow Outcome Scale at 6 months Missing Values Imputed [Age] (mITT Population) |
| Title 2 | Predictor = Age |
| Type of graph | Line graph |
| y-axis | Empirical Cumulative Logit |
| y-axis (label) | Empirical Cumulative Logit |
| x-axis | Age |
| x-axis (label) | Age |
| Legend (if applicable) | A legend should be included to identify each empirical cumulative logit $1 = \text{EmpLogit}_1 = \log[(y_1)/(y_2 + y_3 + y_4)]$ , $2 = \text{EmpLogit}_2 = \log[(y_1 + y_2)/(y_3 + y_4)]$ and $3 = \text{EmpLogit}_3 = \log[(y_1 + y_2 + y_3)/(y_4)]$ |
| Footnote 1 | Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x |
| Additional information | Corresponds to table 14.2.1.1. |

| Figure | 14.2.1.1.4 |
|---|---|
| Title 1 | Graphical Assessment of Proportional Odds Assumption for Proportional Odds Model of Glasgow Outcome Scale at 6 months Missing Values Imputed [GCS Motor Score] (mITT Population) |
| Title 2 | Predictor = GCS motor score |
| Type of graph | Line graph |
| y-axis | Empirical Cumulative Logit |
| y-axis (label) | Empirical Cumulative Logit |
| x-axis | GCS motor score |
| x-axis (label) | GCS motor score |
| Legend (if applicable) | A legend should be included to identify each empirical cumulative logit $1 = \text{EmpLogit}_1 = \log[(y_1)/(y_2 + y_3 + y_4)]$ , $2 = \text{EmpLogit}_2 = \log[(y_1 + y_2)/(y_3 + y_4)]$ and $3 = \text{EmpLogit}_3 = \log[(y_1 + y_2 + y_3)/(y_4)]$ And GCS motor score: $\leq 2 \text{ versus } > 2$ . |
| Footnote 1 | Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x |
| Additional information | Corresponds to table 14.2.1.1. |

| Figure | 14.2.1.1.5 |
|---|---|
| Title 1 | Graphical Assessment of Proportional Odds Assumption for Proportional Odds Model of Glasgow Outcome Scale at 6 months Missing Values Imputed [Pupil Response] (mITT Population) |
| Title 2 | Predictor = Pupil Response |
| Type of graph | Line graph |
| y-axis | Empirical Cumulative Logit |
| y-axis (label) | Empirical Cumulative Logit |
| x-axis | Pupil Response |
| x-axis (label) | Pupil Response |
| Legend (if applicable) | A legend should be included to identify each empirical cumulative logit $1 = \text{EmpLogit}_1 = \log[(y_1)/(y_2 + y_3 + y_4)]$ , $2 = \text{EmpLogit}_2 = \log[(y_1 + y_2)/(y_3 + y_4)]$ and $3 = \text{EmpLogit}_3 = \log[(y_1 + y_2 + y_3)/(y_4)]$ And Pupil Response: bilateral, unilateral, no reactive pupils, or not testable |
| Footnote 1 | Program: xxxxxxx.sas, Output: xxxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x |
| Additional information | Corresponds to table 14.2.1.1. |

| Figure | 14.2.1.1.6 |
|---|---|
| Title 1 | Graphical Assessment of Proportional Odds Assumption for Proportional Odds Model of Glasgow Outcome Scale at 6 months Missing Values Imputed [CT Classification] (mITT Population) |
| Title 2 | Predictor = CT Classification |
| Type of graph | Line graph |
| y-axis | Empirical Cumulative Logit |
| y-axis (label) | Empirical Cumulative Logit |
| x-axis | CT Classification |
| x-axis (label) | CT Classification |
| Legend (if applicable) | A legend should be included to identify each empirical cumulative logit $1 = \text{EmpLogit}_1 = \log[(y_1)/(y_2 + y_3 + y_4)]$ , $2 = \text{EmpLogit}_2 = \log[(y_1 + y_2)/(y_3 + y_4)]$ and $3 = \text{EmpLogit}_3 = \log[(y_1 + y_2 + y_3)/(y_4)]$ And CT Classification: Marshall's CT Classification II, III, IV, evacuated and non-evacuated mass lesion |
| Footnote 1 | Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x |
| Additional information | Corresponds to table 14.2.1.1. |


## APPENDIX 3 SHELLS FOR POST-TEXT TABLES, FIGURES, AND LISTINGS



Table 14.1.1.1 Summary of Investigational Sites' Enrollment Duration (mITT Population)

| | | Study | | | Number of Subjects | |
|---|---|---|---|---|---|---|
| Region/Country <sup>1</sup> /<br>Site | Principal<br>Investigator | Start Date <sup>2</sup> | End Date <sup>2</sup> | Duration<br>(days) <sup>3</sup> | Randomized | Completed<br>Endpoint <sup>4</sup> |
| All Sites (N=xxx) | | DDMONYYYY | DDMONYYYY | XX | XX | XX |
| Region 1/Country AR/ | | | | | | |
| 01 | xxxxxxxxxx | DDMONYYYY | DDMONYYYY | XX | XX | XX |
| 02 | xxxxxxxxxx | DDMONYYYY | DDMONYYYY | XX | XX | XX |
| 03 | xxxxxxxxxxx | DDMONYYYY | DDMONYYYY | XX | xx | XX |

Source: Listing 16.2.3.1.

 $<sup>^{1}</sup>$  See Table 14.1.1.6 for 2-letter country codes.  $^{2}$  Start Date and End Date are the date of the first consent and the last subject randomization at a specific site, respectively.

 $<sup>^3</sup>$  Duration (days) = End Date - Start Date + 1.  $^4$  Subjects are endpoint completers if they provide a GOS assessment at Month 6 or die before Month 6.

Table 14.1.1.2 Summary of Enrollment by Region, Country, and Site (mITT Population)

| | | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) |
| Region <sup>1</sup> /Country <sup>2</sup> /Site | <del>Statistic</del> | n (%) | n (%) | n (%) |
| All Sites | — n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Region | | | | |
| North America | <del>- n (%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Europe | <u> n (%) </u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Asia | <u> n (%) </u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| South America | <del>- n (%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Country | | | | |
| AR | <del>n (%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| AU | — n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| BE | — n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Region/Site | | | | |
| North America | <del>- n (%)</del> | | | |
| 01 | <u> n ( </u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| 02 | <u> n ( </u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | <u> n ( </u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Europe | | | | |
| 01 | | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| 02 | | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

<sup>&</sup>lt;sup>1</sup> North America=United States, Europe=Austria, Belgium, Czech Republic, Finland, France, Germany, Hungary, Israel, Italy, Netherlands, Romania, Russia, Spain, and United Kingdom, Asia=China, Malaysia, Singapore, Taiwan, and Thailand, South America=Argentina.

Note: Percentages are based on the number of subjects in each treatment group and overall in the population of interest.

Source: Listing 16.2.4.1.

<sup>&</sup>lt;sup>2</sup> See Table 14.1.1.6 for 2-letter country codes.

Table 14.1.1.3 Summary of Subject Disposition (Randomized Subjects)

| | | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Subjects Who Were | | | | |
| Randomized but Not Treated | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Modified Intention-to-Treat <sup>1</sup> | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Safety Population <sup>2</sup> | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Per Protocol <sup>3</sup> | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Study Completers <sup>4</sup> | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Endpoint Completers <sup>5</sup> | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Early Termination | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Reason for Early Termination | | | | |
| Death | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Adverse Event(s) | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Withdrawal of Consent | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Protocol Violation | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Lost to Follow-up | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Discretion of the Investigator | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Discretion of the Sponsor | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Other | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

<sup>&</sup>lt;sup>1</sup> Modified Intention-to-Treat (mITT) Population includes all subjects who were randomized and in whom treatment with i.v. study drug was initiated (analyzed according to randomized treatment).

Note: Percentages are based on the number of subjects in each treatment group and overall in the population of interest.

Source: Listings 16.2.1.1, 16.2.1.2, 16.2.3.1

<sup>&</sup>lt;sup>2</sup> Safety Population includes all subjects who received any study medication (analyzed according to actual treatment received).

<sup>&</sup>lt;sup>3</sup> Per Protocol Population includes all subjects in the mITT population who meet all inclusion/exclusion criteria, received at least 96 hours of study medication treatment, and have a non-missing 6-month GOS score.

<sup>4</sup> Subjects are completers if they complete 6 months involvement in the study.

 $<sup>^{5}</sup>$  Subjects who provide a GOS at 6 months, including deaths carried forward to 6 months.

 $\mathcal{U}_{\overline{\mathsf{Version}}\,\mathsf{Date}:\,2.0\,\,\mathsf{April}\,\,\mathsf{19},\,\mathsf{2014}}$ 

Table 14.1.1.4 Summary of Subject Status by Time (mITT Population)

| | | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| | Statistic | (N=XX) | (N=xx) | (N=xx) |
| Study Completers | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Early Termination | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Subjects Remaining in Study | | | | |
| Day 1 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Day 2 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Day 3 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Day 4 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Day 5 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Day 6 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Day 15 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Day 30 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Day 90 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Day 180 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: Subjects are completers if they completed a Month 6 visit. Early terminations include deaths.

Note: Percentages are based on the number of subjects in each treatment group and overall in the population of interest.

Source: Listing 16.2.1.1.



Table 14.1.1.5 Country Codes per ISO

| Code | Country |
|------|----------------|
| AR | Argentina |
| AT | Austria |
| BE | Belgium |
| CN | China |
| CZ | Czech Republic |
| DE | Germany |
| ES | Spain |
| FI | Finland |
| FR | France |
| GB | United Kingdom |
| HU | Hungary |
| IL | Israel |
| IT | Italy |
| MY | Malaysia |
| NL | Netherlands |
| RO | Romania |
| RU | Russia |
| SG | Singapore |
| TH | Thailand |
| TW | Taiwan |
| US | United States |

Note: ISO=International Organization for Standardization.

Table 14.1.2.1 Summary of Study Drug Exposure and Time from Injury (Safety Population)

| | | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Trt <sup>1</sup> Initiated Within 8 Hours of Injury | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Treated for at Least 96 Hours | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Reason for Incomplete Drug | | | | |
| Administration | | | | |
| Adverse Event | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Death | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| PI Decision | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Sponsor Decision | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Consent Withdrawn | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Other | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Length of Exposure (hours) | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | xx.x | XX.X |
| | Q1, Q3 | xx.x , xx.x | xx.x , xx.x | XX.X , XX.X |
| | Min, Max | XX , XX | XX , XX | xx , xx |
| Length of Exposure: Categorized (hours) | | | | |
| >0-<=24 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| >24-<=48 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| >48-<=72 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| >72-<=96 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| >96-<=120 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| >120 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: Length of Exposure (in hours) = last dose date/time - first dose date/time - (sum of recorded durations of infusion rate interruptions).

Note: Percentages are based on the number of subjects in each treatment group and overall in the population of interest.

Source: Listing 16.2.5.2.

 $<sup>^2</sup>$  Relative Dose is summarized for the subset of subjects who received drug for 114 to 126 hours (120 +/- 5%).

Table 14.1.2.1 Summary of Study Drug Exposure and Time from Injury (Safety Population)

| | | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Total Dose (mg/kg) | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X , XX.X | XX.X , XX.X | xx.x , xx.x |
| | Min, Max | xx , xx | xx , xx | xx , xx |
| Relative Dose <sup>2</sup> | | | | |
| 0 < Relative Dose <=80% | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| 80% < Relative Dose <=100% | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| 100% < Relative Dose <=120% | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Relative Dose > 120% | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Time Since Injury to Study Drug (ho | urs) | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x |
| | Min, Max | XX , XX | XX , XX | xx , xx |
| Time Since Injury to Study Drug: | | | | |
| Categorized (hours) | | | | |
| 0-<=4 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| >4-<=6 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| >6-<=8 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| >8-<=9 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| >9 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: Length of Exposure (in hours) = last dose date/time - first dose date/time - (sum of recorded durations of infusion rate interruptions).

Note: Percentages are based on the number of subjects in each treatment group and overall in the population of interest.

Source: Listing 16.2.5.2.

<sup>&</sup>lt;sup>1</sup> Trt = Treatment.

 $<sup>^2</sup>$  Relative Dose is summarized for the subset of subjects who received drug for 114 to 126 hours (120 +/- 5%).



 $a = \frac{1}{\text{Version Date: 2.0 April 19, 2014}}$ 

Table 14.1.2.2 Drug Administration Summary (Safety Population)

| Question | Response | Statistic | BHR-100<br>(N=xx) | Placebo<br>(N=xx) | Total (N=xx) |
|---|---|---|---|---|---|
| | | | n (%) | n (%) | n (%) |
| Infusion Rate Modified on Any Day | Yes | | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | No | | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Reason for Modification | Adverse Event | <del>n (%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | IV Access Problem | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Subcutaneous Infusion | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Inappropriate/Non-Consistent<br>Infusion Rate | <del>n (%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Other | n (೪) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Infusion Interrupted >30 Minutes on Any Day | Yes | | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| - | No | | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Reason for Modification | Adverse Event | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | IV Access Problem | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Subcutaneous Infusion | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Inappropriate/Non-Consistent<br>Infusion Rate | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Other | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |

Note: Percentages are based on the number of subjects in each treatment group and overall in the population of interest.

Source: Listing 16.2.5.1.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Include loading dose and maintenance doses in same table.]


Table 14.1.2.3 Summary of Study Drug Compliance Rate (Safety Population)

| | | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Overall Compliance (%) | n | XX | XX | XX |
| <del>-</del> | Mean (SD) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| | Median | XX.XX | XX.XX | xx.xx |
| | Q1, Q3 | xx.xx , xx.xx | xx.xx , xx.xx | xx.xx , xx.xx |
| | Min, Max | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x |

Note: Compliance rate is calculated by dividing the hours of study medication taken by the number of hours that should have been taken during the treatment period multiplied by 100.

Source: Listing 16.2.5.1 and 16.2.5.2.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Programmer Note: See section 5 and 9.3.1 for details about compliance calculation]



Table 14.1.3.1 Prior and Concomitant Medications by WHO Drug Dictionary Preferred Term (mITT Population)

| | | BHR-100<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| Any Prior or Concomitant<br>Medication | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 2 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 3 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 4 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 5 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: Percentages are based on the number of subjects in each treatment group and total in the population of interest.

Note: Subjects could have received more than one prior medication.

Note: Prior medications are defined as medications with a stop date before the first administration of study medication. Concomitant medications are defined as medications with a start or stop date after the first administration of study medication or ongoing on Day 15.

Source: Listing 16.2.4.6.



 $a \pm \alpha$  Version Date: 2.0 April 19, 2014

Table 14.1.3.2 Surgical Therapy (mITT Population)

| | | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| Characteristic | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Type of Surgery | N | xx | XX | xx |
| Intracranial | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Extracranial | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Intracracranial Surgery Type | N | XX | XX | xx |
| Aneurysm (non trauma) | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Acute Subdural Hematoma | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Contusion | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Craniofacial Surgery | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| CSF Shunt | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Chronic Subdural Hematoma | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Decompressive Craniectomy Injuries | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Depressed Skull Fracture | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Epidural Hematoma | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Intracerebral Hematoma | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Infection | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Optic Nerve Decompression | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Posterior Fossa Surgery | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Skull Base Fracture | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Ventriculostomy for CSG Drainage | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Debridement - Minimal for Penetrating Injuries | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Debridement - Extensive for Penetrating Injuries | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Foreign Body Removal | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Bone Flap Replacement | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Other | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: Percentages are based on the number of subjects with data in each treatment group and total in the population of interest.

Source: Listing 16.2.4.8.



 $a rac{}{}$  Version Date: 2.0 April 19, 2014

Table 14.1.3.2 Surgical Therapy (mITT Population)

| | · | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| Characteristic | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Extracranial Surgery Type | N | xx | xx | xx |
| Maxillofacial | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Extremity Fracture Lower Limb (Internal Fixation) | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Extremity Fracture Lower Limb (External Fixation) | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Extremity Fracture Upper Limb (Internal Fixation) | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Extremity Fracture Upper Limb (External Fixation) | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Fasciotomy | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Laparotomy (Abdomen) | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Pelvic Fracture (Internal Fixation) | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Pelvic Fracture (External Fixation) | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Placement of Chest Tube | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Placement of Gastric Tube (PEG) | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Spinal Stabilization/Thoracic | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Spinal Stabilization/Lumbal | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Thoracotomy | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Tracheostomy | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Urinary Catheter | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Vascular (Operative) | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Vascular (Endovascular Treatment) | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Wound Closure Graft | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Other | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: Percentages are based on the number of subjects with data in each treatment group and total in the population of interest.

Source: Listing 16.2.4.8.



 $a ag{Version Date: 2.0 April 19, 2014}$ 

Table 14.1.4.1 Demographic Characteristics (mITT Population)

| | | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| Characteristic | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Age (years) | n | XX | XX | XX |
| inge (years) | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X , XX.X | XX.X , XX.X | XX.X , XX.X |
| | Min, Max | xx , xx | XX , XX | XX , XX |
| Sex | N | XX | XX | XX |
| Male | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Female | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Ethnicity | N | XX | XX | XX |
| Hispanic or Latino | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Not Hispanic or Latino | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Not Allowed to Obtain | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Race | N | XX | XX | XX |
| White | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Black, African American or of African heritage | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Native Hawaiian or other Pacific Islander | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Asian | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| American Indian or Alaska Native | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Not Allowed to Obtain | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Other | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: Percentages are based on the number of subjects with data in each treatment group and total in the population of interest.

Note: Age (years) = (date of informed consent - date of birth + 1)/365.25.

Source: Listing 16.2.4.1.

Table 14.1.4.2 Pregnancy Testing (mITT Population)

| | | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| Characteristic | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Female <sup>1</sup> | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Female of Child-Bearing Potential <sup>2</sup> | N | xx | XX | xx |
| Yes | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| No | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Missing | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Sample Collected for Pregnancy Test <sup>3</sup> | N | xx | XX | xx |
| Yes | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| No | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Missing | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Pregnancy Test Result <sup>4</sup> | N | xx | XX | xx |
| Positive | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Negative | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Missing | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

<sup>&</sup>lt;sup>1</sup> Percentages are calculated using the number of subjects with data as the numerator and the number of subjects in the mITT population as the denominator.

Source: Listing 16.2.8.1.5.

 $<sup>^{\</sup>frac{1}{2}}$  Percentages are calculated using the number of subjects with data as the numerator and the number of female subjects as the denominator.

<sup>&</sup>lt;sup>3</sup> Percentages are calculated using the number of subjects with data as the numerator and the number of female subjects of child-bearing potential as the denominator.

<sup>&</sup>lt;sup>4</sup> Percentages are calculated using the number of subjects with data as the numerator and the number of samples collected for pregnancy testing as the denominator.

Table 14.1.4.3 Baseline Characteristics (mITT Population)

| | | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) |
| Characteristic | -Statistic | n (%) | n (%) | n (%) |
| Region | | | | |
| North America | <u> n (%)</u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Europe | <del>− n (%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Asia | <del>n_(%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| South America | <u> n (%)</u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| GCS Motor score | | | | |
| 1-2 | <del>− n (%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| 3 | <del>− n (%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| 4 | <u> n (%)</u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| 5-6 | <u> n (%)</u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Pupillary Response | | | | |
| Bilateral | <del>− n (%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Unilateral | <del>− n (%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| No Reactive Pupils | <del>n_(%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Not Testable | <u> n (%)</u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Hypoxia <sup>1</sup> | | | | |
| Yes | <u> n (%)</u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| No | <del>_ n_(%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Suspected | <del>_ n_(%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Unknown | <del>− n (%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: GCS=Glasgow Coma Score.

Note: Percentages are based on the number of subjects with baseline data in each treatment group and overall.

Source: Listing 16.2.6.1.6.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: The GCS motor score will come from the screening GCS, presence of hypoxia/hypotension comes from resuscitation CRF page, CT classification and presence of subarachnoid hemorrhage will come from the screening CT scan. Pupillary response will come from the assessment of right and left pupil reactivity. If both right and left pupils react = bilateral, if either right or left pupil reacts = unilateral, if neither pupil reacts = no reactivel pupils, or the eyes are closed (i.e. untestable) = not testable.]

<sup>&</sup>lt;sup>1</sup> Hypoxia is defined as  $PaO_2 < 60$  mmHg.

 $<sup>^{2}</sup>$  Hypotension is defined as systolic blood pressure < 90 mmHg.


Table 14.1.4.3 Baseline Characteristics (mITT Population)

| | | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| | | (N=xx) | (N=xx) | (N=xx) |
| Characteristic | -Statistic | n (%) | n (%) | n (%) |
| Hypotension <sup>2</sup> | | | | |
| Yes | — n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| No | - n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Suspected | - n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Unknown | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Olikilowii | 11 (0) | AA (AA.A 0) | AA (AA.A 0) | AA (AA.A 0) |
| Marshall CT Classification | | | | |
| I | | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| II | <del>n (%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| III | <u> n (%) </u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| IV | <del>− n (%)</del> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Evacuated/Non-Evacuated Mass Lesion | <u> n (%)</u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Traumatic Subarachnoid Hemorrhage | | | | |
| Yes | - n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| No | <u>n (%)</u> | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: GCS=Glasgow Coma Score.

Note: Percentages are based on the number of subjects with baseline data in each treatment group and overall.

Source: Listing 16.2.6.1.6.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: The GCS motor score will come from the screening GCS, presence of hypoxia/hypotension comes from resuscitation CRF page, CT classification and presence of subarachnoid hemorrhage will come from the screening CT scan. Pupillary response will come from the assessment of right and left pupil reactivity. If both right and left pupils react = bilateral, if either right or left pupil reacts = unilateral, if neither pupil reacts = no reactivel pupils, or the eyes are closed (i.e. untestable) = not testable.]

<sup>&</sup>lt;sup>1</sup> Hypoxia is defined as  $PaO_2 < 60$  mmHg.

 $<sup>^{2}</sup>$  Hypotension is defined as systolic blood pressure < 90 mmHg.



Table 14.1.4.4 Summary of Injury (mITT Population)

| | | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| Characteristic | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Construction Production | | | | |
| Cause of Traumatic Brain Injury | n | XX | XX | XX |
| Motor Vehicle | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Motorcycle | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Fall | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Sports/Recreation | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Pedestrian | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Diving | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Assault | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Other | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: Percentages are based on the number of subjects in each treatment group and total in the population of interest.

Source: Listing 16.2.4.2.



Table 14.1.4.4 Summary of Injury (mITT Population)

| | | BHR-100 | Placebo | Total |
|-------------------|-----------|-------------|-------------|-------------|
| Characteristic | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Head Injury Alone | n (웅) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Face | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Chest | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Abdomen | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Extremities | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Spine | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: Percentages are based on the number of subjects in each treatment group and total in the population of interest.

Source: Listing 16.2.4.2.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: The summaries of Face, Chest, Abdomen, Extremities, and Spine injuries will include subjects who had a severe or critical exam result for the given injury. Head injury alone summary will include subjects who did not have a severe or critical injury to one of the other body parts.]



 $a_{ ext{Version Date: 2.0 April 19, 2014}}$ 

Table 14.1.5 Summary of Medical History by System Organ Class and Preferred Term (Safety Population)

| System Organ Class | | BHR-100 | Placebo | Total |
|----------------------|-----------|-------------|-------------|-------------|
| Preferred Term | Statistic | (N=xx) | (N=XX) | (N=xx) |
| Any Medical History | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| System Organ Class 1 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 2 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 3 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 4 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 5 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| System Organ Class 2 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 1 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 2 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 3 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 4 | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Preferred Term 5 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: Percentages are based on the number of subjects in each treatment group and total in the population of interest.

Source: Listing 16.2.4.5.

Table 14.2.1.1 Summary of Glasgow Outcome Scale at 6 Months Post Injury - Missing Values Imputed (mITT Population)

| | | BHR-100 | Placebo |
|-----------------------|-----------|-------------|-------------|
| Glasgow Outcome Scale | Statistic | (N=xx) | (N=xx) |
| Good Recovery | n (%) | xx (xx.x %) | xx (xx.x %) |
| Moderate Disability | n (%) | xx (xx.x %) | xx (xx.x %) |
| Severe Disability | n (%) | xx (xx.x %) | xx (xx.x %) |
| Vegetative State/Dead | n (%) | xx (xx.x %) | xx (xx.x %) |

Note: Missing values are first imputed by carrying forward the Month 3 GOS assessment. If a subject has neither the 3 nor the 6 month GOS, the missing value is imputed based upon the primary proportional odds model. Percentages are based on the number of non-missing GOS at the month 6 assessment in each treatment group in the population of interest.

Source: Listing 16.2.6.1.4.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: For the "Observed Values" summaries, please add a Missing category to the table.]



Table 14.2.1.2 Analysis of Glasgow Outcome Scale<sup>1</sup> at 6 Months Post Injury - Proportional Odds Model - Missing Values Imputed (mITT Population)

| Characteristic | ${ m DF}^2$ | Chi-Square <sup>3</sup> | P-Value <sup>3</sup> |
|---|---|---|---|
| Score Test for Proportional Odds Assumption <sup>4</sup> | xx | xx.xxx | x.xxx |
| Treatment | XX | xx.xxx | x.xxx |
| Region | xx | xx.xxx | x.xxx |
| Age | XX | xx.xxx | x.xxx |
| GCS Motor Score | xx | xx.xxx | x.xxx |
| Pupil Response | XX | xx.xxx | x.xxx |
| CT Classification | XX | xx.xxx | x.xxx |

Note: Missing values are first imputed by carrying forward the Month 3 GOS assessment. If a subject has neither the 3 nor the 6 month GOS, the missing value is imputed based upon the primary proportional odds model. Missing covariates are imputed as the most common level over all subjects.

Source: Listing 16.2.6.1.4 and 16.2.6.1.6.

<sup>&</sup>lt;sup>1</sup> Response variable Glasgow Outcome Scale at 6 months post injury has 4 values (Good Recovery, Moderate Disability, Severe Disability and Vegetative State/Dead).

<sup>&</sup>lt;sup>2</sup> DF=Degrees of Freedom.

<sup>&</sup>lt;sup>3</sup> The score test is based on the Chi-Square test and the Type 3 analysis of effects are based on the Wald Chi-Square test from a Logistic Regression analysis (Proportional Odds Model). The POM will model the odds of a favorable outcome/higher GOS category and will be fitted including treatment, geographic region (North America, Europe, Asia, and South America), age, GCS motor score (1-2, 3, 4, 5-6), pupil response (unilateral, bilateral, no reactive pupils/not testable), and CT classification (I/II, III, IV, V/VI).

<sup>&</sup>lt;sup>4</sup> A non-significant result supports the proportional odds assumption.

Table 14.2.1.3 ORs<sup>1</sup> and 95% CIs<sup>2</sup> for Glasgow Outcome Scale at 6 Months Post Injury - Proportional Odds Model - Missing Values Imputed (mITT Population)

| Effect <sup>3</sup> | Odds Ratio | 95% CI <sup>2</sup> |
|---|---|---|
| Treatment (BHR-100 vs. Placebo) | x.xx | (x.xx, x.xx) |
| Region (North America vs. Europe) | x.xx | (x.xx, x.xx) |
| Region (Asia vs. Europe) | X.XX | (x.xx, x.xx) |
| Region (South America vs. Europe) | x.xx | (x.xx, x.xx) |
| Age | x.xx | (x.xx, x.xx) |
| GCS Motor Score (3 vs. 1/2) | x.xx | (x.xx, x.xx) |
| GCS Motor Score (4 vs. 1/2) | X.XX | (x.xx, x.xx) |
| GCS Motor Score (5/6 vs. 1/2) | x.xx | (x.xx, x.xx) |
| Pupil Response (Bilateral vs. Unilateral/No Reactive Pupils/Not Testable) | x.xx | (x.xx, x.xx) |
| CT Classification (I/II vs. V/VI) | x.xx | (x.xx, x.xx) |
| CT Classification (III vs. V/VI) | X.XX | (x.xx, x.xx) |
| CT Classification (IV vs. V/VI) | X.XX | (x.xx, x.xx) |

Note: Missing values are first imputed by carrying forward the Month 3 GOS assessment. If a subject has neither the 3 nor the 6 month GOS, the missing value is imputed based upon the primary proportional odds model. Missing covariates are imputed as the most common level over all subjects.

Source: Listing 16.2.6.1.4 and 16.2.6.1.6.

<sup>1</sup> OR=Odds Ratio.

<sup>&</sup>lt;sup>2</sup> CI=Confidence Interval.

<sup>&</sup>lt;sup>3</sup> The OR and CIs come from a Logistic Regression analysis (Proportional Odds Model). The POM will model the odds of a favorable outcome/higher GOS category and will be fitted including treatment, geographic region (North America, Europe, Asia, and South America), age, GCS motor score (1-2, 3, 4, 5-6), pupil response (unilateral, bilateral, no reactive pupils/not testable), and CT classification (I/II, III, IV, V/VI). For factors, the last level is taken as the reference level. For example, CT classification with 5 levels (II-V/VI), level V/VI is taken as the reference level. Marshall CT Score classification was used.




Table 14.2.1.4 Summary of Glasgow Outcome Scale at 6 Months Post Injury - Observed Values (mITT Population)

Table 14.2.1.5 Analysis of Glasgow Outcome Scale at 6 Months Post Injury - Proportional Odds Model - Observed Values (mITT Population)

Table 14.2.1.6 ORs<sup>1</sup> and 95% CIs<sup>2</sup> for Glasgow Outcome Scale at 6 Months Post Injury - Proportional Odds Model - Observed Values (mITT Population)

Table 14.2.1.7 Summary of Glasgow Outcome Scale at 6 Months Post Injury - Observed Values (PP Population)

Table 14.2.1.8 Analysis of Glasgow Outcome Scale at 6 Months Post Injury - Proportional Odds Model - Observed Values (PP Population)

Table 14.2.1.9 ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post Injury - Proportional Odds Model - Observed Values (PP Population)

Table 14.2.1.10 Summary of Glasgow Outcome Scale at 6 Months Post Injury for US Only - Missing Values Imputed (mITT Population)

Table 14.2.1.11 Analysis of Glasgow Outcome Scale at 6 Months Post Injury for US Only - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.1.12 ORs<sup>1</sup> and 95% CIs<sup>2</sup> for Glasgow Outcome Scale at 6 Months Post Injury for US Only - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.1.13 Analysis of Glasgow Outcome Scale at 6 Months Post Injury - Proportional Odds Model - Missing Values Imputed (Unadjusted Analysis) (mITT Population)

Table 14.2.1.14 ORs<sup>1</sup> and 95% CIs<sup>2</sup> for Glasgow Outcome Scale at 6 Months Post Injury - Proportional Odds Model - Missing Values Imputed (Unadjusted Analysis) (mITT Population)

Note: Tables 14.2.1.13 and 14.2.1.14 will only have a row for Treatment, as other covariates will not be included in the model.



Table 14.2.2.1 Summary of Sliding Dichotomy (Dichotomization) at 6 Months Post Injury - Missing Values Imputed (mITT Population)

| | | | BHR-100 | Placebo | Overall |
|---|---|---|---|---|---|
| Prognosis | Characteristic | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Best | n | n | XX | xx | xx |
| | Good Recovery | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Moderate Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Severe Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Vegetative State/Dead | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Intermediate | n | n | XX | xx | xx |
| | Good Recovery | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Moderate Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Severe Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Vegetative State/Dead | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Worst | n | n | XX | XX | xx |
| | Good Recovery | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Moderate Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Severe Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Vegetative State/Dead | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Overall | n | n | XX | XX | xx |
| | Good Recovery | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Moderate Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Severe Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Vegetative State/Dead | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: Missing values are first imputed by carrying forward the Month 3 GOS assessment. If a subject has neither the 3 nor the 6 month GOS, the missing value is imputed based upon the primary proportional odds model. Missing covariates are imputed as the most common level over all subjects.

Percentages are based on the number of subjects in each treatment group in the population of interest.

Source: Listing 16.2.6.2.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Is there a way to indicate with a different font or making the font bold the Glasgow Outcome Scale outcomes that respond to a favorable outcome, i.e. split the overall column into approximately 50:50 within each prognosis group?]



Table 14.2.2.2 Summary and Analysis of Sliding Dichotomy at 6 Months Post Injury - Missing Values Imputed (mITT Population)

| Prognosis | Characteristic | Statistic | BHR-100<br>(N=xx) | Placebo<br>(N=xx) | P-Value <sup>1</sup><br>BHR-100 vs. Placebo | Difference (95% CI) <sup>2</sup><br>BHR-100 - Placebo |
|---|---|---|---|---|---|---|
| Overall | n | n | XX | XX | 0.xxx | xx.x (xx.x, xx.x) |
| | Favorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| | Unfavorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| Best | n | n | XX | xx | 0.xxx | xx.x (xx.x, xx.x) |
| | Favorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| | Unfavorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| Intermediate | n | n | XX | xx | 0.xxx | xx.x (xx.x, xx.x) |
| | Favorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| | Unfavorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| Worst | n | n | XX | xx | 0.xxx | xx.x (xx.x, xx.x) |
| | Favorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| | Unfavorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |

Note: Missing values are first imputed by carrying forward the Month 3 GOS assessment. If a subject has neither the 3 nor the 6 month GOS, the missing value is imputed based upon the primary proportional odds model. Missing covariates are imputed as the most common level over all subjects. Percentages are based on the number of subjects in each treatment group in the population of interest.

1 P-value is based on Cochran-Mantel Haenszel Chi-Square test adjusted for region.

Source: Listing 16.2.6.2.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

Table 14.2.2.4 Summary of Sliding Dichotomy (Dichotomization) at 6 Months Post Injury - Observed Values (mITT Population)

Table 14.2.2.5 Summary and Analysis of Sliding Dichotomy at 6 Months Post Injury - Observed Values (mITT Population)

Table 14.2.2.6 ORs and 95% CIs for Sliding Dichotomy at 6 Months Post Injury - Observed Values (mITT Population)

Table 14.2.2.7 Summary of Sliding Dichotomy (Dichotomization) at 6 Months Post Injury - Observed Values (PP Population)

Table 14.2.2.8 Summary and Analysis of Sliding Dichotomy at 6 Months Post Injury - Observed Values (PP Population)

Table 14.2.2.9 ORs and 95% CIs for Sliding Dichotomy at 6 Months Post Injury - Observed Values (PP Population)

<sup>&</sup>lt;sup>2</sup> Difference is in proportion of favourable outcomes. The confidence interval for the difference is the standard Wald asymptotic confidence interval based on the normal approximation to the binomial distribution.




Table 14.2.2.10 Summary of Sliding Dichotomy (Dichotomization) at 6 Months Post Injury for US Only - Missing Values Imputed (mITT Population)

Table 14.2.2.11 Summary and Analysis of Sliding Dichotomy at 6 Months Post Injury for US Only - Missing Values Imputed (mITT Population)

Table 14.2.2.12 ORs and 95% CIs for Sliding Dichotomy at 6 Months Post Injury for US Only - Missing Values Imputed (mITT Population)


Table 14.2.2.3  $ORs^1$  and 95%  $CIs^2$  for Sliding Dichotomy at 6 Months Post Injury - Missing Values Imputed (mITT Population)

| Characteristic | Prognosis | p-value | OR <sup>3</sup> (95% CI) |
|---|---|---|---|
| Breslow-Day Test for Homogeneity o | f Odds Ratios | x.xxx | |
| Prognosis | Overall | | x.xx (xx.x, xx.x) |
| | Best | | x.xx (xx.x, xx.x) |
| | Intermediate | | x.xx ( $xx.x$ , $xx.x$ ) |
| | Wost | | x.xx ( $xx.x$ , $xx.x$ ) |

Note: Missing values are first imputed by carrying forward the Month 3 GOS assessment. If a subject has neither the 3 nor the 6 month GOS, the missing value is imputed based upon the primary proportional odds model. Missing covariates are imputed as the most common level over all subjects.

Source: Listing 16.2.6.2.

<sup>1</sup> OR=Odds Ratio.

<sup>&</sup>lt;sup>2</sup> CI=Confidence Interval.

 $<sup>^3</sup>$  OR for BHR-100 vs. Placebo is based on Cochran-Mantel Haenszel Chi-Square test adjusted for region.


Table 14.2.3.1 Summary of Dichotomized Glasgow Outcome Scale at 6 Months Post Injury - Missing Values Imputed (mITT Population)

| | | | Placebo |
|---|---|---|---|
| Glasgow Outcome Scale <sup>1</sup> | Statistic | (N=xx) | (N=xx) |
| N | n | XX | XX |
| GR | n (응) | xx (xx.x %) | xx (xx.x %) |
| MD, SD, V/D | n (%) | xx (xx.x %) | xx (xx.x %) |
| N | n | XX | XX |
| GR, MD | n (%) | xx (xx.x %) | xx (xx.x %) |
| SD, V/D | n (%) | xx (xx.x %) | xx (xx.x %) |
| N | n | xx | xx |
| GR, MD, SD | n (%) | xx (xx.x %) | xx (xx.x %) |
| V/D | n (%) | xx (xx.x %) | xx (xx.x %) |

Note: Missing values are first imputed by carrying forward the Month 3 GOS assessment. If a subject has neither the 3 nor the 6 month GOS, the missing value is imputed based upon the primary proportional odds model. Missing covariates are imputed as the most common level over all subjects. Percentages are based on the number of subjects with data at the month 6 assessment in each treatment group in the population of interest.

Source: Listing 16.2.6.1.4.

<sup>&</sup>lt;sup>1</sup> GR=Good Recovery, MD=Moderate Disability, SD=Severe Disability, V/D=Vegetative State/Dead. Vegetative state and dead categories are combined for analysis.

Table 14.2.3.2 Analysis of Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome Scale<sup>1</sup> at 6 Months Post Injury - Missing Values Imputed (mITT Population)

| Variable | ${\sf DF}^2$ | Chi-Square <sup>3</sup> | P-Value <sup>3</sup> |
|---|---|---|---|
| Treatment | xx | xx.xx | x.xxx |
| Region | XX | xx.xxx | X.XXX |
| Age | XX | xx.xxx | X.XXX |
| GCS Motor Score | XX | xx.xxx | x.xxx |
| Pupil Response | XX | xx.xxx | x.xxx |
| CT Classification | XX | XX.XXX | X.XXX |

Note: Missing values are first imputed by carrying forward the Month 3 GOS assessment. If a subject has neither the 3 nor the 6 month GOS, the missing value is imputed based upon the primary proportional odds model. Missing covariates are imputed as the most common level over all subjects.

Source: Listing 16.2.6.1.4 and 16.2.6.1.6.

<sup>&</sup>lt;sup>1</sup> Response variable Glasgow Outcome Scale at 6 months post injury has 2 values (Good Recovery, Moderate Disability vs. Severe Disability, Vegetative State/Dead).

<sup>&</sup>lt;sup>2</sup> DF=Degrees of Freedom.

<sup>&</sup>lt;sup>3</sup> The Type 3 analysis of effects are based on the Wald Chi-Square test from a Logistic Regression analysis. The odds of a favorable outcome (GR, MD) will be modeled and will be fitted including treatment, geographic region (North America, Europe, Asia, and South America), age, GCS motor score (1-2, 3, 4, 5-6), pupil response (unilateral, bilateral, no reactive pupils/not testable), and CT classification (I/II, III, IV, V/VI).<sup>4</sup>



Table  $14.2.3.3~\mathrm{ORs}^1$  and  $95\%~\mathrm{CIs}^2$  for Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome Scale at 6 Months Post Injury - Missing Values Imputed (mITT Population)

| Effect <sup>3</sup> | Odds Ratio | 95% CI <sup>2</sup> |
|---|---|---|
| Treatment (BHR-100 vs. Placebo) | x.xx | (x.xx, x.xx) |
| Region (North America vs. Europe) | x.xx | (x.xx, x.xx) |
| Region (Asia vs. Europe) | X.XX | (x.xx, x.xx) |
| Region (South America vs. Europe) | x.xx | (x.xx, x.xx) |
| Age | x.xx | (x.xx, x.xx) |
| GCS Motor Score (3 vs. 1/2) | x.xx | (x.xx, x.xx) |
| GCS Motor Score (4 vs. 1/2) | X.XX | (x.xx, x.xx) |
| GCS Motor Score (5/6 vs. 1/2) | x.xx | (x.xx, x.xx) |
| Pupil Response (Bilateral vs. Unilateral/No Reactive Pupils/Not Testable) | x.xx | (x.xx, x.xx) |
| CT Classification (I/II vs. V/VI) | x.xx | (x.xx, x.xx) |
| CT Classification (III vs. V/VI) | X.XX | (x.xx, x.xx) |
| CT Classification (IV vs. V/VI) | X.XX | (x.xx, x.xx) |

Note: Missing values are first imputed by carrying forward the Month 3 GOS assessment. If a subject has neither the 3 nor the 6 month GOS, the missing value is imputed based upon the primary proportional odds model. Missing covariates are imputed as the most common level over all subjects.

For factors, the last level is taken as the reference level. For example, CT classification with 4 levels (II-V/VI), level V/VI is taken as the reference level. Marshall CT classification was used.

Source: Listing 16.2.6.1.4 and 16.2.6.1.6.

<sup>1</sup> OR=Odds Ratio.

<sup>&</sup>lt;sup>2</sup> CI=Confidence Interval.

<sup>&</sup>lt;sup>3</sup> The OR and CIs come from a Logistic Regression analysis. The odds of a favorable outcome (GR, MD) will be modeled and will be fitted including treatment, geographic region (North America, Europe, Asia, and South America), age, GCS motor score (1-2, 3, 4, 5-6), pupil response (unilateral, bilateral, no reactive pupils/not testable), and CT classification (I/II, III, IV, V/VI).



Table 14.2.3.4 Summary of Dichotomized Glasgow Outcome Scale at 6 Months Post Injury - Observed Values (mITT Population)

| | | BHR-100 | Placebo |
|------------------------------------|-----------|-------------|-------------|
| Glasgow Outcome Scale <sup>1</sup> | Statistic | (N=xx) | (N=xx) |
| n | n | XX | XX |
| GR, MD | n (%) | xx (xx.x %) | xx (xx.x %) |
| GR, MD<br>SD, V/D | n (%) | xx (xx.x %) | xx (xx.x %) |

<sup>&</sup>lt;sup>1</sup> GR=Good Recovery, MD=Moderate Disability, SD=Severe Disability, V/D=Vegetative/Dead. Vegetative state and dead categories are combined.

Note: Percentages are based on the number of subjects in each treatment group in the population of interest.

Source: Listing 16.2.6.1.4.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

Note to Programmer: Missing value imputation ONLY done for GR, MD vs. SD, V/D dichotomization.


Table 14.2.3.5 Analysis of Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome Scale at 6 Months Post Injury - Observed Values (mITT Population)

Table 14.2.3.6 ORs and 95% CIs for Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome Scale at 6 Months Post Injury - Observed Values (mITT Population)

Table 14.2.3.7 Summary of Dichotomized Glasgow Outcome Scale at 6 Months Post Injury - Observed Values (PP Population)
Table 14.2.3.8 Analysis of Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome Scale at 6 Months Post Injury - Observed Values (PP

Population)

Table 14.2.3.9 ORs1 and 95% CIs2 for Dichotomized (GR, MD vs. SD, V/D) Glasgow Outcome Scale at 6 Months Post Injury - Observed Values (PP Population)

Table 14.2.3.10 Analysis of Dichotomized (GR vs. MD, SD, V/D) Glasgow Outcome Scale<sup>1</sup> at 6 Months Post Injury - Missing Values Imputed (mITT Population)

Table 14.2.3.11 ORs<sup>1</sup> and 95% CIs<sup>2</sup> for Dichotomized (GR vs. MD, SD, V/D) Glasgow Outcome Scale at 6 Months Post Injury -Missing Values Imputed (mITT Population)

Table 14.2.3.12 Analysis of Dichotomized (GR, MD, SD vs. V/D) Glasgow Outcome Scale<sup>1</sup> at 6 Months Post Injury - Missing Values Imputed (mITT Population)

Table 14.2.3.13 ORs¹ and 95% CIs² for Dichotomized (GR, MD, SD vs. V/D) Glasgow Outcome Scale at 6 Months Post Injury - Missing Values Imputed (mITT Population)

Table 14.2.4.1 Analysis of Glasgow Outcome Scale at 6 Months Post Injury - Exploratory Analysis - Missing Values Imputed (mITT Population) - EXAMPLE SHELL\*

| Effort | $DF^4$ | Wald<br>Chi-Square⁵ | P-Value <sup>5</sup> | Interaction Wald<br>Chi-Square <sup>5</sup> | Interaction with<br>Treatment P-value |
|---|---|---|---|---|---|
| Effect | Dr | Cni-square | r-value | Cni-square | Treatment P-value |
| Simple Model <sup>2</sup> | | | | | |
| Treatment | XX | xx.xxx | x.xxx | xx.xxx | |
| Region | XX | xx.xxx | x.xxx | xx.xxx | x.xxx |
| Age | XX | xx.xxx | x.xxx | xx.xxx | x.xxx |
| Race | XX | xx.xxx | x.xxx | xx.xxx | x.xxx |
| GCS Motor Score | XX | XX.XXX | x.xxx | XX.XXX | x.xxx |
| Pupil Response | XX | xx.xxx | x.xxx | xx.xxx | x.xxx |
| CT Classification | XX | xx.xxx | x.xxx | xx.xxx | x.xxx |
| Hypoxia | XX | xx.xxx | x.xxx | xx.xxx | x.xxx |
| Hypotension | XX | xx.xx | X.XXX | XX.XXX | x.xxx |
| Subarachnoid Hemorrhage | XX | xx.xx | X.XXX | XX.XXX | x.xxx |
| Gender | XX | xx.xxx | x.xxx | xx.xxx | x.xxx |
| Time to first dose | XX | XX.XXX | X.XXX | xx.xxx | X.XXX |
| Backward Elimination Model <sup>3</sup> | | | | | |
| Treatment | XX | XX.XXX | x.xxx | | |
| Region | XX | xx.xxx | x.xxx | | |
| Age | XX | XX.XXX | x.xxx | | |

<sup>1</sup> Response variable Glasgow Outcome Scale at 6 months post injury has 4 values (Good Recovery, Moderate Disability, Severe Disability and Vegetative State/Dead).

Source: Listing 16.2.6.1.4 and 16.2.6.1.6.

<sup>&</sup>lt;sup>2</sup> Each factor is included in a model with treatment and the factor by treatment interaction and run individually.

 $<sup>^3</sup>$  The backward elimination model begins with all factors in the model. Factor by treatment interactions with p<0.10 in the simple model are included in the Backward Elimination Model. Factors must have a significance level of p<0.10 to remain in the model. Only the final model is shown.

<sup>&</sup>lt;sup>4</sup> DF=Degrees of Freedom.

<sup>&</sup>lt;sup>5</sup> The Type 3 analysis of effects are based on the Wald Chi-Square test.



[\* The above template is an example. ONLY the final exploratory model will be presented, so not all the terms indicated above may be included.]

If any of the interaction terms in the exploratory analysis are significant, the following subgroup analyses will be presented:

Table 14.2.4.2 Analysis of Glasgow Outcome Scale at 6 Months Post Injury by Region - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table  $14.2.4.3 \, \mathrm{ORs}^1$  and  $95\% \, \mathrm{CIs}^2$  for Glasgow Outcome Scale at 6 Months Post Injury by Region - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.4 Analysis of Glasgow Outcome Scale at 6 Months Post Injury by Age Group - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table  $14.2.4.5 \text{ ORs}^1$  and  $95\% \text{ CIs}^2$  for Glasgow Outcome Scale at 6 Months Post Injury by Age Group - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.6 Analysis of Glasgow Outcome Scale<sup>1</sup> at 6 Months Post Injury by Race Group - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.7 ORs<sup>1</sup> and 95% CIs<sup>2</sup> for Glasgow Outcome Scale at 6 Months Post Injury by Race Group - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.8 Analysis of Glasgow Outcome Scale<sup>1</sup> at 6 Months Post Injury by GCS Motor Score - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.9 ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post Injury by GCS Motor Score - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.10 Analysis of Glasgow Outcome Scale<sup>1</sup> at 6 Months Post Injury by Pupil Response - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.11 ORs<sup>1</sup> and 95% CIs<sup>2</sup> for Glasgow Outcome Scale at 6 Months Post Injury by Pupil Response - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.12 Analysis of Glasgow Outcome Scale at 6 Months Post Injury by CT Classification - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.13 ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post Injury by CT Classification - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.14 Analysis of Glasgow Outcome Scale<sup>1</sup> at 6 Months Post Injury by Presence of Hypoxia - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.15 ORs<sup>1</sup> and 95% CIs<sup>2</sup> for Glasgow Outcome Scale at 6 Months Post Injury by Presence of Hypoxia - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.16 Analysis of Glasgow Outcome Scale<sup>1</sup> at 6 Months Post Injury by Presence of Hypotension - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.17 ORs<sup>1</sup> and 95% CIs<sup>2</sup> for Glasgow Outcome Scale at 6 Months Post Injury by Presence of Hypotension - Proportional Odds Model - Missing Values Imputed (mITT Population)




Table 14.2.4.18 Analysis of Glasgow Outcome Scale<sup>1</sup> at 6 Months Post Injury by Presence of Traumatic Subarachnoid Hemorrhage - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.19 ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post Injury by Traumatic Subarachnoid Hemorrhage - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.20 Analysis of Glasgow Outcome Scale at 6 Months Post Injury by Gender - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table  $14.2.4.21~\mathrm{ORs^1}$  and  $95\%~\mathrm{CIs^2}$  for Glasgow Outcome Scale at 6 Months Post Injury by Gender - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.22 Analysis of Glasgow Outcome Scale<sup>1</sup> at 6 Months Post Injury by Time to First Dose - Proportional Odds Model - Missing Values Imputed (mITT Population)

Table 14.2.4.23 ORs and 95% CIs for Glasgow Outcome Scale at 6 Months Post Injury by Time to First Dose - Proportional Odds Model - Missing Values Imputed (mITT Population)



Table 14.2.5.1 Summary and Analysis of Mortality at Month 6 (mITT Population)

| Mortality | Statistic | BHR-100<br>(N=xx) | Placebo<br>(N=xx) | P-Value <sup>1</sup><br>BHR-100 vs. Placebo | Difference (BHR-100 -<br>Placebo)<br>(95% CI²) |
|---|---|---|---|---|---|
| $N^3$ | n | XX | xx | | |
| Lost to Follow-up | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| Consent Withdrawn | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| Alive | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| Dead | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| Other | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| $N^4$ | n | XX | xx | | |
| Alive | n (%) | xx (xx.x %) | xx (xx.x %) | 0.xxx | x.xx (x.xx, x.xx) |
| Dead | n (%) | xx (xx.x %) | xx (xx.x %) | | |

<sup>1</sup> P-value is based on Fishers Exact test. Only subjects who were either alive or dead at Month 6 will be included in the analysis.

Source: Listing 16.2.6.3.1.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Add a missing category if not all mITT subjects provide details on Month 6 mortality.]

Table 14.2.5.2 Summary and Analysis of Mortality at Month 1 (mITT Population) [Update the footnotes to reflect Month 1 timepoint.]

Table 14.2.5.3 Summary and Analysis of Mortality at Month 6 (PP Population) Table 14.2.5.4 Summary and Analysis of Mortality at Month 1 (PP Population)

 $<sup>^2</sup>$  2-sided 95% confidence interval for the difference in percentage of deaths between BHR-100 and placebo.

<sup>&</sup>lt;sup>3</sup> Percentages are based on the number of subjects in the mITT population.

<sup>4</sup> Percentages are based on the number of subjects with status=alive or dead, Month 6 within the mITT Population.



Table 14.2.5.5 Summary and Kaplan-Meier Analysis of Time to Death¹ (days) (mITT Population)

| | Statistic | BHR-100<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|
| Kaplan-Meier Estimates | Total Deaths | XX | XX |
| | Total Censored | XX | XX |
| | 25 <sup>th</sup> percentile | XX | XX |
| | Median (95% CI) | xx (xx , xx) | xx (xx , xx) |
| | 75 <sup>th</sup> percentile | XX | XX |
| Treatment Difference from Placebo <sup>2</sup> | | p=0.xxx | |

 $<sup>^{1}</sup>$  Time to Death (in days) = Date of death/date of last contact (for censored records) - date of TBI + 1.  $^{2}$  P-value is based on Log-Rank test.

Source: Listing 16.2.6.3.1.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: The K-M estimates are those obtained from PROC LIFETEST.

The log-rank test is fitted in SAS using the following syntax:

PROC LIFETEST DATA=<dataset name>;

TIME WKS\*CENS(1 - censoring indicator);

STRATA TREATMENT;

RUN;



Version Date: 2.0 April 19, 2014 Protocol No. BHR-100-301

Table 14.2.5.6 Summary of Cox Proportional Hazards Analysis of Time to Death (days) (mITT Population)

| Factor/Covariate <sup>1</sup> | Hazard Ratio <sup>1</sup> | 95% Confidence Limits | P-value |
|---|---|---|---|
| Treatment Group (BHR-100 vs. Placebo) | x.xxx | (x.xxx, x.xxx) | 0.xxx |
| Region (North America vs. Europe) | X.XXX | (x.xxx, x.xxx) | 0.xxx |
| Region (Asia vs. Europe) | X.XXX | (x.xxx, x.xxx) | 0.xxx |
| Region (South America vs. Europe) | x.xxx | (x.xxx, x.xxx) | 0.xxx |
| Age | x.xxx | (x.xxx, x.xxx) | 0.xxx |
| GCS Motor Score (3 vs. 1/2) | x.xxx | (x.xxx, x.xxx) | 0.xxx |
| GCS Motor Score (4 vs. 1/2) | x.xxx | (x.xxx, x.xxx) | 0.xxx |
| GCS Motor Score (5/6 vs. 1/2) | x.xxx | (x.xxx, x.xxx) | 0.xxx |
| Pupil Response (Bilateral vs. Unilateral/No<br>Reactive Pupils/Not Testable) | x.xxx | (x.xxx, x.xxx) | 0.xxx |
| CT Classification (I/II vs. V/VI) | x.xxx | (x.xxx, x.xxx) | 0.xxx |
| CT Classification (III vs. V/VI) | x.xxx | (x.xxx, x.xxx) | 0.xxx |
| CT Classification (IV vs. V/VI) | X.XXX | (x.xxx, x.xxx) | 0.xxx |

 $<sup>^{1}</sup>$  For factors the last level is taken as the reference level. Marshall CT classification was used.

Source: Listings 16.2.6.1.6 and 16.2.6.3.1.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Indicator variables or PROC TPHREG (which has a CLASS statement) will need to be created for the factors with more than 2 levels (Region, GCS motor score, Pupil Response and CT classification).

```
proc tphreq data=<dataset>;
class treatment region gcs motor pupil ct class;
model time to death*censoring(0-censoring indicator)=treatment region age gcs motor pupil ct class/ties=efron;
proc phreg data=<dataset>;
treatment gcs motor pupil ct class;
model time to death*censoring(0-censoring indicator)=treatment region1 4 region2 4 region3 4 age gcs motor pupil1 3 pupil2 3
ct class2 6 ct class3 6 ct class4 6 ct class5 6/ties=efron; NB. Underlined terms are indicator variables.
NB. Using EFRON method for ties.]
```

Table 14.2.6.1 Summary of Glasqow Outcome Scale at 3 Months Post Injury - Observed Values (mITT Population) Table 14.2.6.2 Analysis of Glasgow Outcome Scale at 3 Months Post Injury - Proportional Odds Model - Observed Values (mITT Population)




Table 14.2.6.3 ORs and 95% CIs for Glasgow Outcome Scale at 3 Months Post Injury - Proportional Odds Model - Observed Values (mITT Population)



Table 14.2.7.1 Summary of Glasgow Outcome Scale - Extended at 6 Months Post Injury - Observed Values (mITT Population)

| | | BHR-100 | Placebo |
|--------------------------------|-----------|-------------|-------------|
| Glasgow Outcome Scale-Extended | Statistic | (N=xx) | (N=xx) |
| Dead | n (%) | xx (xx.x %) | xx (xx.x %) |
| Vegetative State | n (%) | xx (xx.x %) | xx (xx.x %) |
| Lower Severe Disability | n (%) | xx (xx.x %) | xx (xx.x %) |
| Upper Severe Disability | n (%) | xx (xx.x %) | xx (xx.x %) |
| Lower Moderate Disability | n (%) | xx (xx.x %) | xx (xx.x %) |
| Upper Moderate Disability | n (%) | xx (xx.x %) | xx (xx.x %) |
| Lower Good Recovery | n (%) | xx (xx.x %) | xx (xx.x %) |
| Upper Good Recovery | n (%) | xx (xx.x %) | xx (xx.x %) |
| Missing | n | XX | XX |

Note: Percentages are based on the number of non-missing GOS-E at the month 6 assessment in each treatment group within the population of interest.

Source: Listings 16.2.6.1.4.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

Table 14.2.7.2 Analysis of Glasgow Outcome Scale - Extended at 6 Months Post Injury - Proportional Odds Model - Observed Values (mITT Population)
[See shell for 14.2.1.2.]

Table 14.2.7.3 ORs and CIs of Glasgow Outcome Scale - Extended at 6 Months Post Injury - Proportional Odds Model - Observed Values (mITT Population)
[See shell for 14.2.1.3.]

Table 14.2.7.4 Summary of Sliding Dichotomy (Dichotomization) - Glasgow Outcome Scale - Extended at 6 Months Post Injury - Observed Values (mITT Population)

| | | | BHR-100 | Placebo | Overall |
|---|---|---|---|---|---|
| Prognosis | Characteristic | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Group 1 (Best) | n | n | XX | XX | XX |
| GIOUP I (Best) | | | | | |
| | Upper Good Recovery | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Lower Good Recovery | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Upper Moderate Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Lower Moderate Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Upper Severe Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Lower Severe Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Vegetative State/Dead | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Group 2 | n | n | XX | XX | xx |
| _ | Upper Good Recovery | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Lower Good Recovery | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Upper Moderate Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Lower Moderate Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Upper Severe Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Lower Severe Disability | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| | Vegetative State/Dead | n (응) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Group 6 (Worst)

Overall

Note: Percentages are based on the number of subjects in each treatment group in the population of interest.

Source: Listing 16.2.6.1.4.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Include all 6 prognosis groups and an overall summary. Please make the font bold for the responses in each prognosis group that correspond to a favorable outcome (see SAP text above in Section 9.5.2.3.]



Table 14.2.7.5 Summary and Analysis of Sliding Dichotomy - Glasgow Outcome Scale - Extended at 6 Months Post Injury - Observed Values (mITT Population)

| Prognosis | Characteristic | Statistic | BHR-100<br>(N=xx) | Placebo<br>(N=xx) | P-Value <sup>1</sup><br>BHR-100 vs. Placebo | Difference (95% CI) <sup>2</sup><br>BHR-100 - Placebo |
|---|---|---|---|---|---|---|
| Overall | n | n | XX | XX | 0.xxx | xx.x (xx.x, xx.x) |
| | Favorable | n (%) | xx (xx.x %) | xx (xx.x %) | | , , , |
| | Unfavorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| Group 1 (Best) | n | n | XX | xx | 0.xxx | xx.x (xx.x, xx.x) |
| | Favorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| | Unfavorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| Group 2 | n | n | XX | xx | 0.xxx | xx.x (xx.x, xx.x) |
| | Favorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| | Unfavorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| Group 3 | n | n | XX | xx | 0.xxx | xx.x (xx.x, xx.x) |
| | Favorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |
| | Unfavorable | n (%) | xx (xx.x %) | xx (xx.x %) | | |

Note: Percentages are based on the number of subjects in each treatment group in the population of interest.

 $<sup>^{1}</sup>$  P-value is based on Cochran-Mantel Haenszel Chi-Square test adjusted for region.

<sup>&</sup>lt;sup>2</sup> Difference is in proportion of favourable outcomes. The confidence interval for the difference is the standard Wald asymptotic confidence interval based on the normal approximation to the binomial distribution.

Source: Listing 16.2.6.1.4.



Table 14.2.7.6 ORs<sup>1</sup> and 95% CIs<sup>2</sup> for Sliding Dichotomy - Glasgow Outcome Scale - Extended at 6 Months Post Injury - Observed Values (mITT Population)

| Characteristic | Prognosis | p-value | OR <sup>3</sup> (95% CI) |
|---|---|---|---|
| Breslow-Day Test for Homogeneity of Odds Ratios | | x.xxx | |
| Prognosis | Overall Group 1 (Best) Group 2 Group 3 Group 4 Group 5 Group 6 (Worst) | | x.xx (xx.x, xx.x) |

<sup>1</sup> OR=Odds Ratio.

Source: Listing 16.2.6.1.4.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

Table 14.2.7.7 Summary of Glasgow Outcome Scale - Extended at 3 Months Post Injury - Observed Values (mITT Population)
Table 14.2.7.8 Analysis of Glasgow Outcome Scale - Extended at 3 Months Post Injury - Proportional Odds Model - Observed Values (mITT Population)
[See shell for 14.2.1.2.]

Table 14.2.7.9 ORs and CIs of Glasgow Outcome Scale - Extended at 3 Months Post Injury - Proportional Odds Model - Observed Values (mITT Population)

[See shell for 14.2.1.3.]

<sup>&</sup>lt;sup>2</sup> CI=Confidence Interval.

 $<sup>^3</sup>$  OR for BHR-100 vs. Placebo is based on Cochran-Mantel Haenszel Chi-Square test adjusted for region.



Table 14.2.8.1 Summary of SF-36 by Visit (mITT Population)

| Scale | | BHR-100 | Placebo |
|----------------------|----------------|--------------|--------------|
| Visit | Statistic | (N=xx) | (N=xx) |
| Vitality | | | |
| | _ | | |
| Month 3 | n<br>Mann (CD) | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X |
| | Q1, Q3 | XX.X , XX.X | XX.X , XX.X |
| | Min, Max | XX , XX | XX , XX |
| Month 6 | n | xx | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | XX.X |
| | Q1, Q3 | xx.x , xx.x | XX.X , XX.X |
| | Min, Max | xx , xx | XX , XX |
| Physical Functioning | , | • | , |
| Month 3 | n | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X |
| | Q1, Q3 | xx.x , xx.x | xx.x , xx.x |
| | Min, Max | xx , xx | xx , xx |
| Month 6 | n | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X |
| | Q1, Q3 | XX.X , XX.X | XX.X , XX.X |
| | Min, Max | XX , XX | XX , XX |

<sup>&</sup>lt;sup>1</sup> SF-36=Short Form (36) Health Survey.

Source: Listing 16.2.6.4.3.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Repeat for Month 3 and Month 6 for vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health & physical and mental composite summary scores.]



Table 14.2.8.2 Analysis of SF-36 by Visit (mITT Population)

| | | | LS M | ean | _ Difference in LS Mean | | |
|---|---|---|---|---|---|---|---|
| Summary Scores | Visit | Comparison | BHR-100 | Placebo | BHR-100 - Placebo<br>(95% CI) <sup>1</sup> | Effect<br>Size <sup>1</sup> | P-Value <sup>1</sup> |
| Physical Composite | Month 3 | BHR-100 vs.<br>Placebo | XX.X | XX.X | xx.x (xx.x, xx.x) | x.xxx | 0.xxx |
| | Month 6 | BHR-100 vs.<br>Placebo | XX.X | XX.X | xx.x (xx.x, xx.x) | X.XXX | 0.xxx |
| Mental Composite | Month 3 | BHR-100 vs.<br>Placebo | xx.x | xx.x | xx.x (xx.x, xx.x) | x.xxx | 0.xxx |
| | Month 6 | BHR-100 vs.<br>Placebo | XX.X | XX.X | xx.x (xx.x, xx.x) | x.xxx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> LS Mean, Effect Size and P-Value are based on type III sum of squares from an ANCOVA model for the SF-36 composite summary scores at Month 3 and Month 6, including treatment group.

The SF-36 scores are calculated so that a higher score indicates better health.

A positive difference in LS Mean (BHR-100 - Placebo) indicates a positive effect of BHR-100 over placebo.

Source: Listing 16.2.6.4.3.



Table 14.2.9 Shift Summary of CT1 Classification (mITT Population)

| | | | | | D | ay 6 <sup>2</sup> | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Baseline <sup>2</sup> | I | II | III | IV | Evacuated<br>Mass Lesion | Non-Evacuated<br>Mass Lesion | Missing | Dead |
| BHR-100<br>(N=xx) | I | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x<br>%) |
| (11 1111) | II | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x<br>%) |
| | III | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x<br>%) |
| | IV | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x<br>%) |
| | Evacuated<br>Mass Lesion | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x<br>%) |
| | Non-<br>Evacuated<br>Mass Lesion | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x<br>%) |
| | Missing | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x<br>%) |

<sup>&</sup>lt;sup>1</sup> CT=Computed Tomography.

Source: Listing 16.2.6.5.1.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Repeat for Placebo.]

The Baseline scan was obtained pre-randomization. The second CT was obtained post-infusion on Day 6 +/- 1 day (Post-Injury).

CT scans were assessed and compared by the Central Reader, and classified as follows: I=Diffuse Injury No Visible Pathologic Change,

II=Diffuse Injury - Cisterns present, III=Diffuse Injury with Swelling, IV=Diffuse Injury with Shift, V=Evacuated Mass Lesion and VI=Non-Evacuated Mass Lesion.

Table 14.2.10 Summary of Maximum Intracranial Pressure by Visit (mITT Population)

| • | | | BHR-100 | Placebo |
|---|---|---|---|---|
| Visit <sup>1</sup> | Characteristic <sup>2</sup> | Statistic | (N=xx) | (N=xx) |
| Baseline | Missing ICP | n | xx | xx |
| | Maximum ICP (continuous) | n | xx | XX |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | XX.X | XX.X |
| | | Q1, Q3 | xx.x , xx.x | XX.X , XX.X |
| | | Min, Max | xx , xx | xx , xx |
| | Maximum ICP (categorical) | | | |
| | 0 to < 15 mmHg | n (%) | xx (xx.x %) | xx (xx.x) |
| | >=15 to $< 25$ mmHg | n (%) | xx (xx.x %) | xx (xx.x) |
| | >=25 to $< 40$ mmHg | n (%) | xx (xx.x %) | xx (xx.x) |
| | >=40 mmHg | n (%) | xx (xx.x %) | xx (xx.x) |
| | Maximum ICP (categorical) | | | |
| | 0 to <= 20 mmHg | n (%) | xx (xx.x %) | xx (xx.x) |
| | >20 mmHg | n (%) | xx (xx.x %) | xx (xx.x) |
| | Maximum ICP >= 25mmHq | | | |
| | Yes | n (%) | xx (xx.xx %) | xx (xx.xx %) |
| | No | n (%) | xx (xx.xx %) | xx (xx.xx %) |
| | 110 | 11 (0) | m (m·m o) | M (M.M. 0) |
| | Maximum ICP > 20mmHg | | | |
| | Yes | n (%) | xx (xx.xx %) | xx (xx.xx %) |
| | No | n (%) | xx (xx.xx %) | xx (xx.xx %) |

<sup>&</sup>lt;sup>1</sup> The baseline value is defined as the last measurement taken prior to first administration of study drug.

Note: Percentages are calculated using the number of subjects with data as the numerator and the number of subjects with a non-missing ICP result as the denominator.

Source: Listing 16.2.6.6.1.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Repeat for Day 1-6 (scheduled visits only).]

<sup>&</sup>lt;sup>2</sup> ICP=Intracranial Pressure.

 $a_{rac{}{ ext{Version Date: 2.0 April 19, 2014}}$ 

Table 14.2.11.1 Summary of Cerebral Perfusion Pressure by Visit (mITT Population)

| | _ | <u> </u> | BHR-100 | Placebo |
|---|---|---|---|---|
| Visit <sup>1</sup> | Characteristic <sup>2</sup> | Statistic | (N=xx) | (N=xx) |
| Baseline | Missing CPP | n | xx | xx |
| | Lowest CPP (continuous) | n | xx | xx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | XX.X | XX.X |
| | | Q1, Q3 | xx.x , xx.x | XX.X , XX.X |
| | | Min, Max | xx , xx | xx , xx |
| | Lowest CPP (categorical) | n | xx | xx |
| | < 50mmHg | n (%) | xx (xx.x %) | xx (xx.x %) |
| | >=50 - <60mmHg | n (%) | xx (xx.x %) | xx (xx.x %) |
| | >=60 - <70mmHg | n (%) | xx (xx.x %) | xx (xx.x %) |
| | >=70mmHg | n (%) | xx (xx.x %) | xx (xx.x %) |
| | Highest CPP (continuous) | n | xx | xx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | XX.X | XX.X |
| | | Q1, Q3 | xx.x , xx.x | xx.x , xx.x |
| | | Min, Max | xx , xx | xx , xx |
| | Highest CPP (categorical) | n | xx | xx |
| | < 50mmHg | n (%) | xx (xx.x %) | xx (xx.x %) |
| | >=50 - <60mmHg | n (%) | xx (xx.x %) | xx (xx.x %) |
| | >=60 - <70mmHg | n (%) | xx (xx.x %) | xx (xx.x %) |
| | >=70mmHg | n (%) | xx (xx.x %) | xx (xx.x %) |

 $<sup>^1</sup>$  The baseline value is defined as the last measurement taken prior to first administration of study drug (Day 1).  $^2$  CPP=Cerebral Perfusion Pressure.

Source: Listing 16.2.6.7.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Repeat for Day 1-6. ]



Table 14.2.11.2 Potentially Clinically Important On-Treatment<sup>1</sup> Cerebral Perfusion Pressure (mITT Population)

| Characteristic <sup>2</sup> | Response | Statistic | BHR-100<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| Subjects with any On-treatment CPP Measurement | | n | xx | xx |
| Any CPP value < 50mmHg | Yes<br>No | n (%)<br>n (%) | xx (xx.x %)<br>xx (xx.x %) | xx (xx.x %)<br>xx (xx.x %) |
| Any CPP value >=50 - <60mmHg | Yes<br>No | n (%)<br>n (%) | xx (xx.x %)<br>xx (xx.x %) | xx (xx.x %)<br>xx (xx.x %) |
| Any CPP value >=60 - <70mmHg | Yes<br>No | n (%)<br>n (%) | xx (xx.x %)<br>xx (xx.x %) | xx (xx.x %)<br>xx (xx.x %) |
| Any CPP value >=70mmHg | Yes<br>No | n (%)<br>n (%) | xx (xx.x %)<br>xx (xx.x %) | xx (xx.x %)<br>xx (xx.x %) |

 $<sup>^1</sup>$  On-treatment includes all scheduled and unscheduled CPP measurements taken during Days 1-6 after initiation of study medication.  $^2$  CPP=Cerebral Perfusion Pressure.

Source: Listing 16.2.6.7.



Table 14.2.12.1 Summary of Therapy Intensity Level by Visit (mITT Population)

| Visit <sup>1</sup> | | | BHR-100 | Placebo |
|---|---|---|---|---|
| Characteristic <sup>2</sup> | Response | Statistic | (N=xx) | (N=xx) |
| Baseline | | n | XX | xx |
| TIL (continuous) | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | XX.X |
| | | Q1, Q3 | xx.x , xx.x | XX.X , XX.X |
| | | Min, Max | XX , XX | XX , XX |
| Day 1 | | n | xx | xx |
| TIL (continuous) | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | XX.X | XX.X |
| | | Q1, Q3 | xx.x , xx.x | XX.X , XX.X |
| | | Min, Max | xx , xx | XX , XX |

Source: Listing 16.2.6.8.1.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Repeat for Day 2-6.]

 $<sup>^{1}</sup>$  The baseline value is defined as the last measurement taken prior to first administration of study drug (Day 1).  $^{2}$  TIL=Therapy Intensity Level. TIL is recorded for up to 6 days while ICP is being monitored. Each of the listed treatments will have a score of 1 with a maximum score of 10 per subject.



 $a_{\overline{ ext{Version Date: 2.0 April 19, 2014}}}$ 

Table 14.2.12.2 Summary of Individual TIL Therapies (mITT Population)

| | BHR-100 | Placebo |
|-----------------------------------------|-------------|-------------|
| herapy | (N=xx) | (N=XX) |
| Surgical Decompression | xx (xx.x %) | xx (xx.x %) |
| Barbiturate Induced Coma | xx (xx.x %) | xx (xx.x %) |
| Hypothermia | xx (xx.x %) | xx (xx.x %) |
| Hyperventilation (pCO <sub>2</sub> <30) | xx (xx.x %) | xx (xx.x %) |
| Pressor Administration (to keep CPP>60) | xx (xx.x %) | xx (xx.x %) |
| Hypertonic Saline | xx (xx.x %) | xx (xx.x %) |
| Mannitol | xx (xx.x %) | xx (xx.x %) |
| Ventricular Drainage | xx (xx.x %) | xx (xx.x %) |
| Paralysis Induction | xx (xx.x %) | xx (xx.x %) |
| Sedation | xx (xx.x %) | xx (xx.x %) |

Subjects may have received multiple therapies, and therefore may be counted in multiple rows. Source: Listing 16.2.6.8.1.


Table 14.2.12.3 Summary of Maximum Therapy Intensity Level (mITT Population)

| Therapy | Response | Statistic | BHR-100<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| Inerapy | <del>Response</del> | <del>Statistic</del> | (N-XX) | (IV-XX) |
| Surgical Decompression | | | xx (xx.x %) | xx (xx.x %) |
| Barbiturate Induced Coma | | | xx (xx.x %) | xx (xx.x %) |
| Hypothermia | | | xx (xx.x %) | xx (xx.x %) |
| Hyperventilation (pCO <sub>2</sub> <30) | | | xx (xx.x %) | xx (xx.x %) |
| Pressor Administration (to keep CPP>60) | | | xx (xx.x %) | xx (xx.x %) |
| Hypertonic Saline | | | xx (xx.x %) | xx (xx.x %) |
| Mannitol | | | xx (xx.x %) | xx (xx.x %) |
| Ventricular Drainage | | | xx (xx.x %) | xx (xx.x %) |
| Paralysis Induction | | | xx (xx.x %) | xx (xx.x %) |
| Sedation | | | xx (xx.x %) | xx (xx.x %) |
| No Intervention | | | xx (xx.x %) | xx (xx.x %) |

Note: Subjects are summarized according to the maximum therapy received on Days 1-6.

Source: Listing 16.2.6.8.1.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x



Table 14.3.1.1 Overall Summary of Treatment Emergent Adverse Events (Safety Population)

| | | -100<br>=xx) | Placebo<br>(N=xx) | |
|---|---|---|---|---|
| dverse Event Category | # (%) Subj | # AEs | # (%) Subj | # AEs |
| ny | xx (xx.x %) | XX | xx (xx.x %) | xx |
| ny Treatment-Related AE | xx (xx.x %) | XX | xx (xx.x %) | XX |
| ny Serious AE | xx (xx.x %) | XX | xx (xx.x %) | XX |
| ny Treatment-Related Serious AE | xx (xx.x %) | XX | xx (xx.x %) | xx |
| y AE Leading to Premature Discontinuation of Study Drug | xx (xx.x %) | XX | xx (xx.x %) | xx |
| y Treatment-Related AE Leading to Premature Discontinuation of Study Drug | xx (xx.x %) | XX | xx (xx.x %) | XX |
| ny AE Which Resulted in Death | xx (xx.x %) | XX | xx (xx.x %) | xx |
| y Treatment-Related AE Which Resulted in Death | xx (xx.x %) | XX | xx (xx.x %) | xx |

Note: Treatment-emergent adverse events are defined as events that start on or after the first dose of study medication.

Note: For each category, subjects are included only once, even if they experienced multiple events in that category.

Note: Percentages are based on the number of subjects in each treatment group in the population of interest.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: An event is considered related to study medication if it has a relationship other than not related. An event is considered serious, if "Is this a serious adverse event (SAE)"=Yes, an event leads to premature discontinuation of study drug if action taken with study drug due to the AE is drug withdrawn and an event which resulted in death has "If SAE is Yes, Results in death?"=Yes.]



Table 14.3.1.2 Overall Summary of Treatment Emergent Adverse Events by Gender (Safety Population)

Gender: Male

| | | R-100<br>=xx) | Placebo<br>(N=xx) | |
|---|---|---|---|---|
| Adverse Event Category | # (%) Subj | # AEs | # (%) Subj | # AEs |
| Any | xx (xx.x %) | XX | xx (xx.x %) | XX |
| ny Treatment-Related AE | xx (xx.x %) | XX | xx (xx.x %) | xx |
| ny Serious AE | xx (xx.x %) | XX | xx (xx.x %) | xx |
| ny Treatment-Related Serious AE | xx (xx.x %) | XX | xx (xx.x %) | xx |
| ny AE Leading to Premature Discontinuation of Study Drug | xx (xx.x %) | XX | xx (xx.x %) | xx |
| ny Treatment-Related AE Leading to Premature Discontinuation of Study Drug | xx (xx.x %) | XX | xx (xx.x %) | xx |
| ny AE Which Resulted in Death | xx (xx.x %) | XX | xx (xx.x %) | XX |
| ny Treatment-Related AE Which Resulted in Death | xx (xx.x %) | XX | xx (xx.x %) | xx |

Note: Treatment-emergent adverse events are defined as events that start on or after the first dose of study medication.

Note: For each category, subjects are included only once, even if they experienced multiple events in that category.

Note: Percentages are based on the number of subjects in each treatment group in the population of interest.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: An event is considered related to study medication if it has a relationship other than not related. An event is considered serious, if "Is this a serious adverse event (SAE)"=Yes, an event leads to premature discontinuation of study drug if action taken with study drug due to the AE is drug withdrawn and an event which resulted in death has "If SAE is Yes, Results in death?"=Yes.]



Table 14.3.1.2 Overall Summary of Treatment Emergent Adverse Events by Gender (Safety Population)

Gender: Female

| | | R-100<br>=xx) | Placebo<br>(N=xx) | |
|---|---|---|---|---|
| Adverse Event Category | # (%) Subj | # AEs | # (%) Subj | # AEs |
| Any | xx (xx.x %) | xx | xx (xx.x %) | xx |
| Any Treatment-Related AE | xx (xx.x %) | XX | xx (xx.x %) | xx |
| Any Serious AE | xx (xx.x %) | xx | xx (xx.x %) | xx |
| Any Treatment-Related Serious AE | xx (xx.x %) | xx | xx (xx.x %) | xx |
| Any AE Leading to Premature Discontinuation of Study Drug | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Any Treatment-Related AE Leading to Premature Discontinuation of Study Drug | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Any AE Which Resulted in Death | xx (xx.x %) | xx | xx (xx.x %) | xx |
| Any Treatment-Related AE Which Resulted in Death | xx (xx.x %) | XX | xx (xx.x %) | XX |

Note: Treatment-emergent adverse events are defined as events that start on or after the first dose of study medication.

Note: For each category, subjects are included only once, even if they experienced multiple events in that category.

Note: Percentages are based on the number of subjects in each treatment group in the population of interest.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: An event is considered related to study medication if it has a relationship other than not related. An event is considered serious, if "Is this a serious adverse event (SAE)"=Yes, an event leads to premature discontinuation of study drug if action taken with study drug due to the AE is drug withdrawn and an event which resulted in death has "If SAE is Yes, Results in death?"=Yes.]

Table 14.3.1.3 Overall Summary of Treatment Emergent Adverse Events by Race Group(Safety Population) [Repeat the table for each Race group: white, non-white, not allowed to obtain]
Table 14.3.1.4 Overall Summary of Treatment Emergent Adverse Events by Age Group (Safety Population)
[Repeat the table for each Age group: ≤45 years, >45 years]

xx (xx.x %)

xx (xx.x %)

xx (xx.x %)

xx (xx.x %)

XX

xx

Version Date: 2.0 April 19, 2014

Preferred Term 2

Preferred Term 3

Preferred Term 4

Preferred Term 5

| | | BHR-100<br>(N=xx) | | Placebo (N=xx) |
|---|---|---|---|---|
| System Organ Class | | | | |
| Preferred Term | # (%) Subj | # AEs | # (%) Subj | # AEs |
| Any Adverse Event | xx (xx.x %) | xx | xx (xx.x %) | xx |
| System Organ Class 1 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 1 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 2 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 3 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 4 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 5 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| System Organ Class 2 | xx (xx.x %) | XX | xx (xx.x %) | xx |
| Preferred Term 1 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 2 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 3 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 4 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 5 | xx (xx.x %) | XX | xx (xx.x %) | xx |
| System Organ Class 3 | xx (xx.x %) | xx | xx (xx.x %) | XX |
| Preferred Term 1 | xx (xx.x %) | XX | xx (xx.x %) | xx |

Note: Treatment-emergent adverse events are defined as events that start on or after the first dose of study medication.

Note: Adverse events are coded by MedDRA Version 13.0.

Note: For each system organ class and preferred term, subjects are included only once, even if they experienced multiple events in that system organ class or preferred term.

XX

XX

XX

Note: Percentages are based on the number of subjects in each treatment group in the population of interest.

xx (xx.x %)

xx (xx.x %)

xx (xx.x %)

xx (xx.x %)

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Sort in decreasing order of frequency in the BHR-100 column by SOC and by preferred term within SOC.]

Table 14.3.1.9 Treatment-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) [Repeat above table for treatment-related AEs.]

Table 14.3.1.6 Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Gender (Safety Population)

| | Gender=N | | | |
|----------------------|-------------|---------|-------------|---------|
| | | BHR-100 | | Placebo |
| | | (N=xx) | | (N=XX) |
| ubgroup | | | | |
| System Organ Class | | " | | |
| Preferred Term | # (%) Subj | # AEs | # (%) Subj | # AEs |
| Any Adverse Event | xx (xx.x %) | xx | xx (xx.x %) | xx |
| System Organ Class 1 | xx (xx.x %) | xx | xx (xx.x %) | xx |
| Preferred Term 1 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 2 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 3 | xx (xx.x %) | xx | xx (xx.x %) | XX |
| Preferred Term 4 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 5 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| System Organ Class 2 | xx (xx.x %) | xx | xx (xx.x %) | xx |
| Preferred Term 1 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 2 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 3 | xx (xx.x %) | xx | xx (xx.x %) | XX |
| Preferred Term 4 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 5 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| System Organ Class 3 | xx (xx.x %) | xx | xx (xx.x %) | xx |
| Preferred Term 1 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 2 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 3 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 4 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 5 | xx (xx.x %) | xx | xx (xx.x %) | XX |

Note: Treatment-emergent adverse events are defined as events that start on or after the first dose of study medication.

Note: Adverse events are coded by MedDRA Version 13.0.

Note: For each system organ class and preferred term, subjects are included only once, even if they experienced multiple events in that system organ class or preferred term.

Note: Percentages are based on the number of subjects in each treatment group in the population of interest.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Repeat for Gender=Female. Sort in decreasing order of frequency in the BHR-100 column by SOC and by preferred term within SOC.]

Table 14.3.1.7 Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Race Group (Safety Population)
[Repeat above table for race groups White, Non-white, and Not allowed to obtain.]

Table 14.3.1.8 Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Age Group (Safety Population)




[Repeat above table for age groups ≤45 years and >45 years.]

Table 14.3.1.10 Treatment Emergent Adverse Events by Maximum Severity, System Organ Class and Preferred Term (Safety Population)

| | | BHR-100 (N=xx) | | | Placebo (N=xx) | |
|---|---|---|---|---|---|---|
| System Organ Class | Mild | Moderate | Severe | Mild | Moderate | Severe |
| Preferred Term | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| All Adverse Events | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| System Organ Class 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Preferred Term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Preferred Term 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Preferred Term 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Preferred Term 5 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| System Organ Class 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Preferred Term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Preferred Term 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Preferred Term 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Preferred Term 5 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |

Note: Treatment-Emergent adverse events are defined as events that start on or after the first dose of study medication.

Note: Adverse Events are coded by MedDRA Version 13.0.

Note: For each system organ class and preferred term, subjects are included only once, even if they experienced multiple events in that system organ class or preferred term.

Note: Percentages are based on the number of subjects in each treatment group in the population of interest.

Note: If the severity of an Adverse Event is missing, then it is considered to be severe.

Source: Listing 16.2.7.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Each subject is counted only once in the particular AE class, under the highest intensity they experienced for that class of AE.]

Table 14.3.1.11 Treatment-Related Treatment Emergent Adverse Events by Maximum Severity, System Organ Class and Preferred Term (Safety Population)

Table 14.3.1.12 Treatment Emergent Adverse Events by Maximum Relationship and System Organ Class and Preferred Term (Safety Population)

| | | BHR-100 | ) (N=xx) | | | Placebo (N=xx) | | |
|---|---|---|---|---|---|---|---|---|
| System Organ Class | Not Related | Possibly | ossibly Probably | | Not Related | Possibly | Probably | Related |
| Preferred Term | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| All Adverse Events | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |
| System Organ Class 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |
| Preferred Term 2 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |
| Preferred Term 3 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |
| Preferred Term 4 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |
| Preferred Term 5 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |
| System Organ Class 2 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |
| Preferred Term 1 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |
| Preferred Term 2 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |
| Preferred Term 3 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |
| Preferred Term 4 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |
| Preferred Term 5 | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x % |

Note: Treatment-Emergent adverse events are defined as events that start on or after the first dose of study medication.

Note: Adverse Events are coded by MedDRA Version 13.0.

Note: For each system organ class and preferred term, subjects are included only once, even if they experienced multiple events in that system organ class or preferred term.

Note: Percentages are based on the number of subjects in each treatment group in the population of interest.

Note: If the relationship of an Adverse Event is missing, then it is considered to be related to study medication.

Source: Listing 16.2.7.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Each subject is counted only once in the particular AE class, under the most related category they experienced for that class of AE. If the AE relationship to study medication is missing, then it is considered to be related.]




Table 14.3.1.13 Treatment Emergent Adverse Events Leading to Premature Discontinuation of Study Drug by System Organ Class and Preferred Term (Safety Population)

Table 14.3.1.14 Treatment-Related Treatment Emergent Adverse Events Leading to Premature Discontinuation of Study Drug by System Organ Class and Preferred Term (Safety Population)

[Use shell for Table 14.3.1.7, change footnotes accordingly.]



Table 14.3.1.15 Treatment Emergent Adverse Events of Special Interest (Safety Population)

| | | BHR-100<br>(N=xx) | | Placebo<br>(N=xx) |
|---|---|---|---|---|
| AE of Special Interest Preferred Term | # (%) Subj | # AEs | # (%) Subj | # AEs |
| Any Adverse Event of Special Interest | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Serious Thromboembolic Events | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 1 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Preferred Term 2 | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Thrombotic Myocardial Infarction | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Pulmonary Embolism | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Deep Vein Thrombosis | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Ischemic Stroke | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Allergic Reactions | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Marked Liver Function Abnormalities | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Serious Infections | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Pneumonia | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Pneumonia Streptococcal | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Sepsis | xx (xx.x %) | XX | xx (xx.x %) | XX |
| Meningitis | xx (xx.x %) | XX | xx (xx.x %) | xx |

Note: Treatment-emergent adverse events are defined as events that start on or after the first dose of study medication.

Note: Adverse events are coded by MedDRA Version 13.0.

Note: For each preferred term, subjects are included only once, even if they experienced multiple events in that preferred term.

Note: Percentages are based on the number of subjects in each treatment group in the population of interest.

Program: xxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Sort in decreasing order of frequency in the BHR-100 column by preferred term. Need to identify the MedDRA preferred terms that relate to these events of special interest (see page 28 of protocol for events of special interest details).]



## Table 14.3.1.16 List of Adverse Events of Special Interest (Safety Population)

| Treat<br>-ment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Adverse Event/<br>Preferred Term/<br>SOC | Start Date/<br>Day <sup>2</sup> | Stop Date | Length of<br>Exposure<br>(days) <sup>3</sup> | Duration <sup>4</sup> | Intensity | Relation-<br>ship/<br>Outcome | Action Taken<br>with Study<br>Drug | Serious?/<br>Treatment<br>Emergent? <sup>5</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| BHR-<br>100 | **-** | M/10/W | ***************/ ********************* | DDMONYYYY/<br>xx | DDMONYYYY | xx | жж | Mild,<br>Moderate,<br>Severe | Not<br>Related,<br>Possibly<br>Related,<br>Probably<br>Related/Re<br>covered/re<br>solved,<br>Recovering<br>/Resolving | Dose not changed, drug withdrawn, | Yes/<br>Yes |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

Events of special interest are defined as one of the following dictionary defined terms: Serious Thromboembolic Events, Thrombotic Myocardial Infarction, Pulmonary Embolism, Deep Vein Thrombosis, Ischemic Stroke, Allergic Reactions, Marked Liver Function Abnormalities, Serious Infections, Pneumonia, Pneumonia Streptococcal, Sepsis, or Meningitis.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

<sup>&</sup>lt;sup>2</sup> Day is relative to the start date of study medication, event start date - administration start date + 1 if event start date if on or after the date of the start of study medication administration or event start date - administration start date if event date if before the date of the start of study medication administration.

 $<sup>^{3}</sup>$  Length of exposure is based on administration start date and administration end date during the study (end date - start date + 1).

<sup>&</sup>lt;sup>4</sup> Duration = AE end date - AE start date + 1.

<sup>&</sup>lt;sup>5</sup> Treatment emergent adverse events are defined as events that start on or after the first dose of study medication.



 $a_{\overline{ ext{Version Date: 2.0 April 19, 2014}}}$ 


Table 14.3.2.1 Serious Adverse Events by System Organ Class and Preferred Term (Safety Population)
Table 14.3.2.2 Treatment-Related Serious Adverse Events by System Organ Class and Preferred Term (Safety Population)
[Use shell for Table 14.3.1.7, change footnotes accordingly.]



 $a_{ extstyle extstyle$ 

Table 14.3.2.3 Primary Cause of Death (mITT Population)

| | | BHR-100 | Placebo | Total |
|---|---|---|---|---|
| | Statistic | (N=xx) | (N=xx) | (N=xx) |
| ny Death | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Increased Intracranial Pressure | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Increase in Hematoma Size | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| New Hematoma/Re-accumulation | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Cerebral Edema | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Herniation | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Cerebral Infarct | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Cerebral Vasospasm | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Meningitis | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Extracranial Injury | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Myocardial Infarction | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Pulmonary Embolus | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Multiple Organ Failure | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Pneumonia | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Adult Respiratory Distress Syndrome | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Sepsis | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Unknown/Undetermined | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Other | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x



Table 14.3.4.1 Post-Baseline Abnormal, Clinically Significant (non-AE) Laboratory Test Results: Coagulation (Safety Population)

| | BHI | R-100 | | Placebo |
|---|---|---|---|---|
| | Day 6 | Day 15 | Day 6 | Day 15 |
| Outcome | n (%) | n (%) | n (%) | n (%) |
| Number of Abnormal, Clinically Significant (non-AE) lab results | xx | xx | xx | xx |
| Resolved | | xx (xx.x %) | | xx (xx.x %) |
| Ongoing | | xx (xx.x %) | | xx (xx.x %) |
| Lost to Follow-up | | xx (xx.x %) | | xx (xx.x %) |
| Missing | | xx (xx.x %) | | xx (xx.x %) |

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: If there are no results with a Missing outcome, do not include the Missing row.]



Table 14.3.4.2 Post-Baseline Abnormal, Clinically Significant (non-AE) Laboratory Test Results: Hematology (Safety Population)

| | BHI | R-100 | | Placebo |
|---|---|---|---|---|
| Parameter | Day 6 Da | | Day 6 | Day 15 |
| Outcome | n (%) | n (%) | n (%) | n (%) |
| White blood cell count | | | | |
| Number of Abnormal, Clinically Significant (non-AE) lab results | xx | xx | xx | xx |
| Resolved | | xx (xx.x %) | | xx (xx.x %) |
| Ongoing | | xx (xx.x %) | | xx (xx.x %) |
| Lost to Follow-up | | xx (xx.x %) | | xx (xx.x %) |
| Missing | | xx (xx.x %) | | xx (xx.x %) |

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Repeat for remaining hematology lab tests: Differential WBC, Red blood cell count (RBC), Hemoglobin, Hematocrit, Reticulocyte count, and Platelets. If there are no results with a Missing outcome, do not include the Missing row.]




Table 14.3.4.3 Post-Baseline Abnormal, Clinically Significant (non-AE) Laboratory Test Results: Serum Chemistry (Safety Population) (Use Table 14.3.4.2 shell, Subset off details for serum chemistry lab tests: AST, ALT, Alkaline Phosphatase, GGT, Total Protein, Total Cholesterol, Triglycerides, Glucose, Sodium, Potassium, Chloride)

Table 14.3.4.4 Post-Baseline Abnormal, Clinically Significant (non-AE) Laboratory Test Results: Urinalysis (Safety Population) (Use Table 14.3.4.2 shell, Subset off details for all urinalysis tests)

Version Date: 2.0 April 19, 2014 Protocol No. BHR-100-301

Table 14.3.4.5 List of Post-Baseline Abnormal, Clinically Significant (non-AE) Laboratory Test Results: Coagulation (Safety Population)

(Produce for INR)

[Use shell below for Table 14.3.4.6]

Table 14.3.4.6 List of Post-Baseline Abnormal, Clinically Significant (non-AE) Laboratory Test Results: Hematology (Safety Population)

| Sex | ~ / | Can / | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Sex/ Creatment Subject Age/ Group No. Race <sup>1</sup> Test Name | Test Name | <u> </u> | | Result Range<br>(Unit) Flag <sup>2</sup> | | Low | High | Outcome | Other,<br>specify | |
| -xxx M/3 | 35/W | Hemoglobin | Screening | DDMONYYYY | xx.x a/L | T. | XX.X | XX.X | Ongoing | |
| 11, 0 | 00, | 1101110 9 1 0 2 1 11 | UN | DDMONYYYY | xx.x q/L | L | XX.X | XX.X | Resolved | |
| | | | Day 6 | DDMONYYYY | xx.x g/L | L | XX.X | XX.X | Ongoing | |
| | | | Day 15 | DDMONYYYY | xx.x g/L | L | XX.X | XX.X | Other | XXXXXXXXX |
| | Ra | Race <sup>1</sup> | Race <sup>1</sup> Test Name | Race <sup>1</sup> Test Name Visit xxx M/35/W Hemoglobin Screening UN Day 6 | Race <sup>1</sup> Test Name Visit Date xxx M/35/W Hemoglobin Screening DDMONYYYY UN DDMONYYYY Day 6 DDMONYYYY | Race <sup>1</sup> Test Name Visit Date (Unit) XXX M/35/W Hemoglobin Screening DDMONYYYY XX.X g/L UN DDMONYYYY XX.X g/L Day 6 DDMONYYYY XX.X g/L | Race <sup>1</sup> Test Name Visit Date (Unit) Flag <sup>2</sup> XXX M/35/W Hemoglobin Screening DDMONYYYY xx.x g/L L UN DDMONYYYY xx.x g/L L Day 6 DDMONYYYY xx.x g/L L | Race <sup>1</sup> Test Name Visit Date (Unit) Flag <sup>2</sup> Low XXX M/35/W Hemoglobin Screening DDMONYYYY xx.x g/L L xx.x UN DDMONYYYY xx.x g/L L xx.x Day 6 DDMONYYYY xx.x g/L L xx.x | Race <sup>1</sup> Test Name Visit Date (Unit) Flag <sup>2</sup> Low High XXX M/35/W Hemoglobin Screening DDMONYYYY xx.x g/L L xx.x xx.x UN DDMONYYYY xx.x g/L L xx.x xx.x Day 6 DDMONYYYY xx.x g/L L xx.x xx.x | Race <sup>1</sup> Test Name Visit Date (Unit) Flag <sup>2</sup> Low High Outcome XXX M/35/W Hemoglobin Screening DDMONYYYY xx.x g/L L xx.x xx.x Ongoing UN DDMONYYYY xx.x g/L L xx.x xx.x Resolved Day 6 DDMONYYYY xx.x g/L L xx.x xx.x Ongoing |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

[Note to Programmer: Produce for clinically significant abnormalities only. Produce for Hemoglobin, Hematocrit, RBC, Reticulocyte Count, Platelet Count, WBC, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils.]

Table 14.3.4.7 List of Post-Baseline Abnormal, Clinically Significant (non-AE) Laboratory Tests: Serum Chemistry (Safety Population)

(Produce for Sodium, Potassium, Chloride, Total Cholesterol, Triglycerides, ALT, AST, GGT, Alkaline Phosphatase, Total Protein, Glucose.)

Table 14.3.4.8 List of Post-Baseline Abnormal, Clinically Signficant (non-AE) Laboratory Tests: Urinalysis (Safety Population) (Produce for pH, Specific Gravity, Protein, Glucose, Blood, WBC, RBC, Casts, Epithelial Cells, Bacteria.)
[Use shell for table 14.3.4.6]

<sup>&</sup>lt;sup>2</sup> N = Normal, L = Low, H = High.

UN = Unscheduled.



Table 14.3.4.9 Summary of Coagulation Laboratory Test Results (Safety Population)

| | | E | BHR-100 | I | Placebo |
|---|---|---|---|---|---|
| | | | (N=xx) | | (N=xx) |
| | | | Change from | | Change from |
| arameter/Visit | Statistic | Actual Value | Baseline | Actual Value | Baseline |
| NR (ratio) | | | | | |
| Baseline | n | XX | | XX | |
| | Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | |
| | Median | XX.X | | XX.X | |
| | Min, Max | xx , xx | | xx , xx | |
| | Q1, Q3 | XX , XX | | XX , XX | |
| Day 6 | n | XX | XX | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx , xx | xx , xx | xx , xx | xx , xx |
| | Q1, Q3 | XX , XX | xx , xx | XX , XX | xx , xx |
| Day 15 | n | XX | XX | XX | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | xx.x | XX.X | XX.X |
| | Min, Max | xx , xx | xx , xx | xx , xx | XX , XX |
| | Q1, Q3 | xx , xx | xx , xx | xx , xx | xx , xx |

Note: The baseline value is defined as the last measurement taken prior to first administration of study drug (Day 1).

Source: Listing 16.2.8.1.1.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

Table 14.3.4.10 Summary of Hematology Laboratory Test Results (Safety Population)
(Produce for Hemoglobin, Hematocrit, RBC, Reticulocyte Count, Platelets, WBC, Neutrophils, Lymphocytes, Monocytes, Eosinophils, and Basophils. Sort parameters alphabetically. Summarize parameters in standard SI units.)

Table 14.3.4.11 Summary of Serum Chemistry Laboratory Test Results (Safety Population)
(Produce for Sodium, Potassium, Chloride, Total Cholesterol, Triglycerides, ALT, AST, GGT, Alkaline phosphatase, Total Protein, Glucose. Sort parameters alphabetically. Summarize parameters in standard SI units.)



Table 14.3.5 Summary of Incidence of Neuroworsening (Safety Population)

| | Statistic | BHR-100<br>(N=xx) | Placebo<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| Subjects Experiencing Neuroworsening<br>Event ≤ Day 6 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Subjects Experiencing Neuroworsening<br>Event ≤ Day 15 | n (%) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

Note: Neuroworsening is defined as any one of the following: a decrease in GCS motor score  $\geq 2$ , development of pupillary abnormalities, any other neurological deterioration or progression of lesion on CT scan leading to a change in subject management. Note: Percentages are based on the number of subjects in each treatment group and overall in the population of interest.

Source: Listing 16.2.8.6.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x



Table 14.3.6.1 Summary of Vital Signs Corresponding to Lowest Measurement by Visit (Safety Population)

| | | | 3HR-100<br>(N=xx) | Placebo<br>(N=xx) | |
|---|---|---|---|---|---|
| | | • | Change from | | Change from |
| Variable/Visit | Statistic | Actual Value | Baseline | Actual Value | Baseline |
| Pulse (per min) | | | | | |
| Baseline | n | XX | | XX | |
| | Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | |
| | Median | XX.X | | XX.X | |
| | Min, Max | xx , xx | | xx , xx | |
| | Q1, Q3 | XX , XX | | XX , XX | |
| Day 1 | N | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | xx.x | XX.X | XX.X |
| | Min, Max | xx , xx | xx , xx | xx , xx | xx , xx |
| | Q1, Q3 | XX , XX | XX , XX | XX , XX | XX , XX |
| Day 2 | N | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | xx.x | XX.X | xx.x |
| | Min, Max | xx , xx | xx , xx | xx , xx | XX , XX |
| | Q1, Q3 | xx , xx | xx , xx | xx , xx | xx , xx |

Note: The baseline value is defined as the last measurement taken prior to first administration of study drug (Day 1).

Source: Listing 16.2.8.2.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Repeat for Day 3-6. Repeat for other vital sign parameters - respiration rate (bpm, breaths per minute), systolic pressure (mmHg), diastolic blood pressure (mmHg), and temperature (C). The vital signs are reported which correspond to the lowest and highest measurements per study day.]

Table 14.3.6.2 Summary of Vital Signs Corresponding to Highest Measurement by Visit (Safety Population)



 $a_{rac{}{ ext{Version Date: 2.0 April 19, 2014}}$ 

Table 14.3.6.3 Summary of Vital Signs by Visit - Weight (kg) (Safety Population)

| | | | BHR-100<br>(N=xx) | Placebo<br>(N=xx) | |
|---|---|---|---|---|---|
| Variable/Visit | Statistic | Actual Value | Change from<br>Baseline | Actual Value | Change from<br>Baseline |
| Weight (kg) | | | | | |
| Baseline | n | XX | | XX | |
| | Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | |
| | Median | XX.X | | XX.X | |
| | Min, Max | XX , XX | | xx , xx | |
| | Q1, Q3 | XX , XX | | XX , XX | |
| Day 6 | N | XX | XX | XX | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx , xx | xx , xx | xx , xx | xx , xx |
| | Q1, Q3 | xx , xx | xx , xx | xx , xx | xx , xx |

Note: The baseline value is defined as the last measurement taken prior to first administration of study drug (Day 1).

Source: Listing 16.2.8.2.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x



Table 14.3.7.1 Summary of Physical Examination by Visit (Safety Population)

| Body System/<br>Visit | Characteristic | Statistic | BHR-100<br>(N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|
| Skin | | N | XX | XX |
| Baseline | Normal | n (%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) |
| | Not Done | n | xx (xx.x%) | xx (xx.x%) |
| | | N | xx | xx |
| Day 6 | Normal | n (%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) |
| | Not Done | n | xx (xx.x%) | xx (xx.x%) |
| HEENT | | N | xx | xx |
| Baseline | Normal | n (%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) |
| | Not Done | n | xx (xx.x%) | xx (xx.x%) |
| | | N | xx | xx |
| Day 6 | Normal | n (%) | xx (xx.x%) | xx (xx.x%) |
| - | Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) |
| | Not Done | n | xx (xx.x%) | xx (xx.x%) |
| Respiratory | | N | xx | xx |
| Screening | Normal | n (%) | xx (xx.x%) | xx (xx.x%) |
| 3 | Abnormal | n (%) | xx (xx.x%) | xx (xx.x%) |
| | Not Done | n | xx (xx.x%) | xx (xx.x%) |

Note: The baseline value is defined as the last measurement taken prior to first administration of study drug (Day 1). For physical examination assessments this will be the screening visit.

Note: Percentages are based on the number of subjects with data at the visit within the population of interest.

Source: Listing 16.2.8.3.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Physical examination is only conducted at screening and Day 6 visit.

Repeat for all Body systems: Skin, HEENT, Respiratory, Cardiovascular, Abdomen (including liver and kidneys), Neurological,
Gastrointestinal, Genitourinary, Endocrine, Lymph Nodes.]



Table 14.3.7.2 List of Physical Examination Abnormalities Post-Baseline (Safety Population)

| Treatment Group | Subject No. | Sex/Age/<br>Race <sup>1</sup> | Body System | Baseline <sup>2</sup> | Visit <sup>3</sup> | Describe Abnormality |
|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | (Skin, HEENT, Respiratory, Cardiovascular, Abdomen (including liver and kidneys), Neurological, Gastrointestinal, Genitourinary, Endocrine, Lymph Nodes.) | Normal | (Day 6, UN) | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

•••

[Note to Programmer: Only produce for records which record the physical examination post-baseline as abnormal.]

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

 $<sup>^2</sup>$  The baseline value is defined as the last measurement taken prior to first administration of study drug (Day 1). For physical examination assessments this will be the screening visit.

<sup>3</sup> UN = Unscheduled.



 $a ag{Version Date: 2.0 April 19, 2014}$ 

14.3.8.1 Post-baseline Abnormal ECG Results (Safety Population)

| | | | BHR-100 | Placebo |
|---|---|---|---|---|
| Visit <sup>1</sup> | Characteristic <sup>2</sup> | Statistic | (N=xx) | (N=xx) |
| Baseline | Abnormal Rhythm | n | XX | xx |
| | Sinus Arrhythmia | n (%) | xx (xx.x %) | xx (xx.x %) |
| | Atrial Fibrillation | n (%) | xx (xx.x %) | xx (xx.x %) |
| | Atrial Flutter | n (%) | xx (xx.x %) | xx (xx.x %) |
| | Premature Ventricular Contraction | n (%) | xx (xx.x %) | xx (xx.x %) |
| | Other Arrhythmia | n (%) | xx (xx.x %) | xx (xx.x %) |
| | Abnormal Rhythm - Clin Sig | n | XX | xx |
| | Yes | n (%) | xx (xx.x %) | xx (xx.x %) |
| | No | n (%) | xx (xx.x %) | xx (xx.x %) |
| | Abnormal Conduction | n | XX | xx |
| | LBBB | n (%) | xx (xx.x %) | xx (xx.x %) |
| | RBBB | n (%) | xx (xx.x %) | xx (xx.x %) |
| | AV Block | n (%) | xx (xx.x %) | xx (xx.x %) |
| | QT Prolongation | n (%) | xx (xx.x %) | xx (xx.x %) |
| | Other | n (%) | xx (xx.x %) | xx (xx.x %) |
| | Abnormal Conduction - Clin Sig | n | XX | XX |
| | Yes | n (%) | xx (xx.x %) | xx (xx.x %) |
| | No | n (%) | xx (xx.x %) | xx (xx.x %) |

 $<sup>^{1}</sup>$  The baseline value is defined as the last measurement taken prior to first administration of study drug (Day 1).  $^{2}$  Clin Sig = Clinically Significant.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Repeat for Baseline and Day 6.]



 $a_{rac{}{ ext{Version Date: 2.0 April 19, 2014}}$ 

14.3.8.1 Post-baseline Abnormal ECG Results (Safety Population)

| | | | BHR-100 | Placebo |
|---|---|---|---|---|
| Visit <sup>1</sup> | Characteristic <sup>2</sup> | Statistic | (N=xx) | (N=xx) |
| Danalina | Abramal ODG Camples | _ | | |
| Baseline | Abnormal QRS Complex | n | XX | XX |
| | Non-specific ST Changes | n (%) | xx (xx.x %) | xx (xx.x %) |
| | Old MI | n (%) | xx (xx.x %) | xx (xx.x %) |
| | Myocardial Ischemia | n (응) | xx (xx.x %) | xx (xx.x %) |
| | Acute Myocardial Infarction | n (%) | xx (xx.x %) | xx (xx.x %) |
| | Other | n (%) | xx (xx.x %) | xx (xx.x %) |
| | Abnormal QRS Complex - Clin Sig | n | XX | xx |
| | Yes | n (%) | xx (xx.x %) | xx (xx.x %) |
| | No | n (%) | xx (xx.x %) | xx (xx.x %) |

 $<sup>^1</sup>$  The baseline value is defined as the last measurement taken prior to first administration of study drug (Day 1).  $^2$  Clin Sig = Clinically Significant.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Repeat for Screening and Day 6.]



Table 14.3.8.2 List of Post-Baseline Abnormal ECG Results - Part 1 (Safety Population)

| | | | | | Rhythm | | | | Conduction | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject<br>No. | Sex/Age/<br>Race <sup>1</sup> | Visit <sup>2</sup> | Result | Specify# | Clin.<br>Sig. <sup>3</sup> | Result | Specify# | QTC Prolongation (ms) | Clin.<br>Sig. <sup>3</sup> |
| BHR-100 | xx-xxx | M/35/W | Day 6 | Abnormal | Sinus Arrhythmia | No | Normal | | | |
| | | | UN | Abnormal | Other: xxxxxxxxxxxx | Yes | Abnormal | QT<br>Prolongation | xxx | No |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

[Note to Programmer: Only produce for records which record the ECG post-baseline as abnormal.]

<sup>&</sup>lt;sup>2</sup> UN = Unscheduled.

<sup>&</sup>lt;sup>3</sup> Clin. Sig. = Clinically Significant.

<sup>#</sup> If specify=other include details from the other specify comment here.



Table 14.3.8.2 List of Post-Baseline Abnormal ECG Results - Part 2 (Safety Population)

| | | | | | QRS Complex | | |
|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject<br>No. | Sex/Age/<br>Race <sup>1</sup> | Visit <sup>2</sup> | Result | Specify# | Clin.<br>Sig. <sup>3</sup> | Comments |
| BHR-100 | xx-xxx | M/35/W | Day 6 | Abnormal | Non-specific ST Changes | Yes | *********** |
| | | | UN | Normal | | | |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

[Note to Programmer: Only produce for records which record the ECG post-baseline as abnormal.]

<sup>&</sup>lt;sup>2</sup> UN = Unscheduled.

<sup>&</sup>lt;sup>3</sup> Clin. Sig. = Clinically Significant.

<sup>#</sup> If specify=other include details from the other specify comment here.



14.3.9 Summary of Worst Arterial Blood Gas (ABG) Results by Visit (Safety Population)

| | BHR-100 (N = XXX) | | Placebo (N = XXX) | |
|---|---|---|---|---|
| ABG Parameter<br>Timepoint | Change | | Change | |
| | Value | from Baseline | Value | From Baseline |
| $PaO_2$ | | | | |
| Baseline | | | | |
| n | xx | | XX | |
| Mean (std) | xx.xx (xx.xxx) | | xx.xx (xx.xxx) | |
| Median | XX.X | | XX.X | |
| Q1, Q3 | XX.X, XX.X | | XX.X, XX.X | |
| Min, Max | xx.x, xx.x | | xx.x, xx.x | |
| Day 1 | | | | |
| n | xx | xx | XX | xx |
| Mean (std) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X |
| Day 2 | | | | |
| n | xx | | XX | |
| Mean (std) | xx.xx (xx.xxx) | | xx.xx (xx.xxx) | |
| Median | XX.X | | XX.X | |
| Q1, Q3 | xx.x, xx.x | | xx.x, xx.x | |
| Min, Max | XX.X, XX.X | | XX.X, XX.X | |

Note: The baseline value is defined as the last measurement taken prior to first administration of study drug (Day 1). Worst result is calculated as lowest value of the day for  $PaO_2$ ,  $HCO_3$ , pH,  $SaO_2$ , and  $FiO_2$  and the highest value of the day for  $PaCO_2$ .

Source: Listing 16.2.8.5.

Program: xxxxxxx.sas, Output: xxxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Repeat for all ABG parameters:  $PaO_2$ ,  $PaCO_2$ ,  $HCO_3$ , pH,  $SaO_2$  (%) and  $FiO_2$  (%) and all visits (Day1-6). Values should be the worst ABG result recorded that day.]

 $a_{ extstyle extstyle$ 


Table 14.3.10 Summary of Day 2 Progesterone Levels (Safety Population)

| Parameter | Statistic | BHR-100<br>(N = XXX) | Placebo (N = XXX) |
|-----------|-----------|----------------------|-------------------|
| ay 2 | | | |
| -1 - | | | |
| Baseline | n | XXX | XXX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X |
| | Min, Max | XX , XX | xx , xx |
| | Q1, Q3 | XX , XX | xx , xx |

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

| Figure | 14.2.1.1 |
|---|---|
| Title 1 | Glasgow Outcome Scale distribution at 6 Months Post Injury – Missing Values Imputed (mITT Population) |
| Title 2 | |
| Type of graph | Bar Chart |
| y-axis | % response |
| y-axis (label) | % response |
| x-axis | Glasgow Outcome Scale response |
| x-axis (label) | Glasgow Outcome Scale response |
| Legend (if applicable) | Treatment Group: BHR-100 and Placebo. Different bar color for each treatment group. Glasgow Outcome Scale response: D/VS=Dead, Vegetative State, SD=Severe Disability, MD=Moderate Disability, GR=Good Recovery |
| Footnote 1 | Note: Percentages are based on the number of GOS at the month 6 assessment in each treatment group in the population of interest, after imputation. Missing values are first imputed by carrying forward the Month 3 GOS assessment. If a subject has neither the 3 nor the 6 month GOS, the missing value is imputed based upon the primary proportional odds model. Program: xxxxxxxx.sas, Output: xxxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x |
| Additional information | Corresponds to table 14.2.1.1. |

| Figure | 14.2.1.2 |
|---|---|
| Title 1 | Glasgow Outcome Scale distribution at 6 Months Post Injury – Observed Values (mITT Population) |
| Title 2 | |
| Type of graph | Bar Chart |
| y-axis | % response |
| y-axis (label) | % response |
| x-axis | Glasgow Outcome Scale response |
| x-axis (label) | Glasgow Outcome Scale response |
| Legend (if applicable) | Treatment Group: BHR-100 and Placebo. Different bar color for each treatment group. Glasgow Outcome Scale response: D/VS=Dead, Vegetative State, SD=Severe Disability, MD=Moderate Disability, GR=Good Recovery |
| Footnote 1 | Note: Percentages are based on the number of non-missing GOS at the month 6 assessment in each treatment group in the population of interest. Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x |
| Additional information | Corresponds to table 14.2.1.4. |


| Figure | 14.2.1.3 |
|---|---|
| Title 1 | Glasgow Outcome Scale distribution at 6 Months Post Injury – Observed Values (PP Population) |
| Title 2 | |
| Type of graph | Bar Chart |
| y-axis | % response |
| y-axis (label) | % response |
| x-axis | Glasgow Outcome Scale response |
| x-axis (label) | Glasgow Outcome Scale response |
| Legend (if applicable) | Treatment Group: BHR-100 and Placebo. Different bar color for each treatment group. Glasgow Outcome Scale response: D/VS=Dead, Vegetative State, SD=Severe Disability, MD=Moderate Disability, GR=Good Recovery |
| Footnote 1 | Note: Percentages are based on the number of non-missing GOS at the month 6 assessment in each treatment group in the population of interest. Program: xxxxxxx.sas, Output: xxxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x |
| Additional information | Corresponds to table 14.2.1.7. |

| Figure | 14.2.2.1 |
|---|---|
| Title 1 | Dichotomized Glasgow Outcome Scale at 6 Months Post Injury – Missing Values Imputed (mITT Population) |
| Title 2 | |
| Type of graph | Bar Chart |
| y-axis | % response |
| y-axis (label) | % response |
| x-axis | Dichotomized Glasgow Outcome Scale response (favorable, unfavorable) |
| x-axis (label) | Dichotomized Glasgow Outcome Scale response (favorable, unfavorable) |
| Legend (if applicable) | |
| Footnote 1 | Favorable response = GR,MD; Unfavorable response = SD, VS/D. Note: Missing values are first imputed by carrying forward the Month 3 GOS assessment. If a subject has neither the 3 nor the 6 month GOS, the missing value is imputed based upon the primary proportional odds model. |
| Additional information | Corresponds to table 14.2.3.1. |

| Figure | 14.2.2.2 |
|---|---|
| Title 1 | Dichotomized Glasgow Outcome Scale at 6 Months Post Injury – Observed Values (mITT Population) |
| Title 2 | |
| Type of graph | Bar Chart |
| y-axis | % response |
| y-axis (label) | % response |
| x-axis | Dichotomized Glasgow Outcome Scale response (favorable, unfavorable) |
| x-axis (label) | Dichotomized Glasgow Outcome Scale response (favorable, unfavorable) |
| Legend (if applicable) | |
| Footnote 1 | Favorable response = GR,MD; Unfavorable response = SD, VS/D. |
| Additional information | Corresponds to table 14.2.3.4. |

| Figure | 14.2.3.1 |
|---|---|
| Title 1 | Mortality at 6 months (mITT Population) |
| Title 2 | |
| Type of graph | Bar Chart |
| y-axis | % mortality |
| y-axis (label) | % mortality |
| x-axis | Treatment Group |
| x-axis (label) | Treatment Group |
| Legend (if applicable) | Treatment Group: BHR-100 and Placebo. Different bar color/pattern for each treatment group. |
| Footnote 1 | Note: Fishers Exact test p=0.xxx. Only subjects who were either alive or dead at Month 6 will be included in the analysis. Note: Percentages are based on the number of subjects with status=alive or dead at Month 6 within the mITT population. |
| | Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x |
| Additional information | Corresponds to table 14.2.5.1. |
| Figure | 14.2.3.2 |
|---|---|
| Title 1 | Mortality at 1 month (mITT Population) |
| Title 2 | |
| Type of graph | Bar Chart |
| y-axis | % mortality |
| y-axis (label) | % mortality |
| x-axis | Treatment Group |
| x-axis (label) | Treatment Group |
| Legend (if applicable) | Treatment Group: BHR-100 and Placebo. Different bar color/pattern for each treatment group. |
| Footnote 1 | Note: Fishers Exact test p=0.xxx. Only subjects who were either alive or dead at Month 1 will be included in the analysis. Note: Percentages are based on the number of subjects with status=alive or dead at Month 1 within the mITT population. Program: xxxxxxxx.sas, Output: xxxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x |
| Additional information | Corresponds to table 14.2.5.2. |

| Figure | 14.2.3.3 |
|---|---|
| Title 1 | Time to Death (mITT Population) |
| Title 2 | |
| Type of graph | Line graph |
| y-axis | 1 - Kaplan-Meier survival estimates x 100 |
| y-axis (label) | Cumulative Percent Dead |
| x-axis | Time (0-6/7 months) |
| x-axis (label) | Time (in months) |
| Legend (if applicable) | BHR-100, Placebo (different line type for each treatment group) |
| Footnote 1 | Time to death = (Date of death or date of last contact (if censored) – date of TBI + $1$ )/30.4. |
| | Program: xxxxxxxx.sas, Output: xxxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x |
| Additional | Censored observations should be identified. |
| information | Output K-M survival estimates using OUTSURV on PROC LIFETEST statement or SURVIVAL statement. Then calculate 1-K-M survival estimates as want to calculate probability of death over time. Then multiply |

Figure will run from 0% (no deaths) to 100% (all subjects have died) as the x-axis of time progresses from the

by 100 to obtain the percentage.

left to the right. Figure corresponds with Table 14.2.5.5.



# **LISTINGS**

Listing 16.2.1.1 Study Completion/Discontinuation Details

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Infusion<br>Administration<br>Start Date/Time | Infusion<br>Completion<br>Date/Time | Completion<br>Status | Reason for Early Termination<br>(Specify) | Date of Study<br>Completion/<br>Early<br>Termination |
|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | | DDMONYYYY/<br>XX:XX | Completed | (Death, Adverse Event(s), Withdrawal of Consent, Protocol Violation, Lost to Follow-up, Discretion of the Investigator, Discretion of the Sponsor, other) (provide details when reason for termination is other) | DDMONYYYY |
| | xx-xxx | F/33/B | | DDMONYYYY/<br>XX:XX | Withdrew | Other (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | DDMONYYYY |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.


## Listing 16.2.1.2 Eligibility/Randomization

| Treatment<br>Group | Subject No. | Sex/<br>Age/<br>Race <sup>1</sup> | Date/Time of<br>Written<br>Informed<br>Consent | Subject met all entry criteria? | Inclusion/Exclusion<br>Criteria Not Met | Subject<br>Randomized? | Date/Time of<br>Randomization |
|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | DDMONYYYY/<br>XX:XX | (Yes, No) | Inclusion Criteria 1 | (Yes, No) | DDMONYYYY/<br>XX:XX |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: All inc/exc criteria met comes from has the subject met all eligibility criteria? If date of randomization provided, subject is randomized set to Yes]


## Listing 16.2.1.3 Exclusions from Per Protocol Population

| Treatment Group | Subject No. | Sex/<br>Age/<br>Race <sup>1</sup> | Violation Code | Violation Description |
|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | xxxxxxx | *************************************** |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

Program: xxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Include violations with an NE (not evaluable) designation.]



#### Listing 16.2.3.1 Subject General Information

| | | | | | | | | Date or | Date/Time | | | _ | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treat- ment Subject Group No. | Subject<br>No. | Sex/<br>ct Age/<br>Race <sup>1</sup> | $\mathtt{mITT}^2$ | <sub>TT</sub> ² Safety/<br>Act Tmt | PP | Screened | Informed<br>Consent | Random-<br>ization | First Dose | Last<br>Dose | Study<br>Exit | Study<br>Outcome | Exit<br>Day <sup>3</sup> | Treatment<br>Duration<br>(hours) <sup>4</sup> | Compliance<br>Rate <sup>5</sup> |
| BHR- | xx-xxx | M/35/W | Yes | Yes | Yes | DDMONYYYY | DDMONYYYY/ | DDMONYYYY/ | DDMONYYYY/ | DDMONYYYY/ | DDMONYYYY | Completed | 182 | 120 | xxx.x |
| 100 | | F/33/B | Yes | Yes | Yes | DDMONYYYY | XX:XX<br>DDMONYYYY/<br>XX:XX | XX:XX<br>DDMONYYYY/<br>XX:XX | XX:XX<br>DDMONYYYY/<br>XX:XX | XX:XX<br>DDMONYYYY/<br>XX:XX | DDMONYYYY | Withdrew | 24 | 121 | xxx.x |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: List for BHR-100 and Placebo. Sort by subject number within treatment group. This note relates to all listings.]

<sup>&</sup>lt;sup>2</sup> mITT=Modified Intention-to-Treat, PP=Per Protocol.

 $<sup>^3</sup>$  Exit day = exit date (date of completion/date of early termination) - date of randomization + 1.

<sup>&</sup>lt;sup>4</sup> Treatment duration (hours) = (end of administration date/time - start of administration date/time + 1) - duration of any interruptions.

<sup>&</sup>lt;sup>5</sup> Compliance rate is calculated by dividing the hours of study medication taken by the number of hours that should have been taken during the treatment period multiplied by 100.

Version Date: 2.0 April 19, 2014 Protocol No. BHR-100-301

## Listing 16.2.3.2 Informed Consent

| | | | Date/Time | Did Subject Sig | n Informed Consent w | hen he/she regained consciousness? |
|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject No. | Sex/<br>Age/<br>Race <sup>1</sup> | of Written<br>Informed<br>Consent | Response | If Yes, Date<br>Subject Signed<br>Informed Consent | If No or N/A, Specify |
| BHR-100 | xx-xxx | M/35/W | DDMONYYYY/<br>XX:XX | (yes, no, N/A) | DDMONYYYY | ********** |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.



Listing 16.2.4.1 Demographic Characteristics

| Treatment<br>Group | Subject<br>No. | Date<br>of<br>Birth | Date of<br>Screening<br>Visit | Age<br>(years) <sup>1</sup> | Sex | Ethnicity <sup>2</sup> | Race <sup>3</sup><br>If other, Specify | Weight<br>(kg) | Region/Country <sup>4</sup> /Site |
|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | DDMONYYYY | DDMONYYYY | xx | (Male,<br>Female) | (HL, NHL,<br>NAL) | (W, B, P, A,<br>N, Z, O) | xx.x | xxxxxx/xx/xxxxx |
| | | | | | 10, | 111111111111111111111111111111111111111 | 11, 2, 0, | | (Region is North |
| | | | | | | | (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | America, Europe, or<br>Asia and South<br>America) |

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Weight is obtained from IWRS upload.]

 $<sup>^1</sup>$  Age is defined as (date of informed consent - date of birth + 1)/365.25.  $^2$  HL= Hispanic or Latino, NHL=Not Hispanic or Latino, NAL=Not Allowed to Obtain.

W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

<sup>&</sup>lt;sup>4</sup> This is the two letter country code: US=United States, AT=Austria, BE=Belgium, CZ=Czech Republic, FI=Finland, FR=France, DE=Germany, HU=Hungary, IL=Israel, IT=Italy, NL=Netherlands, RO=Romania, RU=Russia, GB=United Kingdom, ES=Spain, CN=China, MY=Malaysia, TW=Taiwan, Province of China, SG=Singapore, TH=Thailand, AR=Argentina.

Listing 16.2.4.2 Baseline Characteristics

| Treatment<br>Group | Subject | Sex/<br>Age/<br>Race <sup>1</sup> | Date of<br>Screening<br>Visit | Date/Time<br>of Injury | Start<br>Date/Time<br>of Study<br>Medication | Injury to<br>medication<br>intake<br>(hours) <sup>2</sup> | Cause of TBI <sup>3</sup> (If Other, Specify) | Exam | Status <sup>4</sup> |
|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | DDMONYYYY | DDMONYYYY/<br>XX:XX | DDMONYYYY/<br>XX:XX | 7 | Motor Vehicle | Head | Critical |
| | xx-xxx | F/33/W | DDMONYYYY | DDMONYYYY/<br>XX:XX | DDMONYYYY/<br>XX:XX | 8.5* | Other (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Abdomen | Serious |
| | xx-xxx | F/39/B | DDMONYYYY | DDMONYYYY/<br>XX:XX | DDMONYYYY/<br>XX:XX | 7 | (Motor Vehicle, Motorcycle, Fall, Sports/ Recreation, Pedestrian, Diving, Assault, Other) | (Head, Face,<br>Chest,<br>Abdomen,<br>Extremities,<br>Spine) | (None,<br>Minor,<br>Moderate,<br>Serious,<br>Severe,<br>Critical) |

•••

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

<sup>&</sup>lt;sup>2</sup> Injury to medication intake (hours) = start date/time of study medication - date/time of injury. A star (\*) will be added to indicate that the intake of study medication was greater than 8 hours after injury.

<sup>3</sup> TBI=Traumatic Brain Injury.

<sup>&</sup>lt;sup>4</sup> None=no treatment, moderate=requires only outpatient treatment, serious=requires non-ICU hospital admission, severe=requires ICU observation and/or basic treatment, critical=requires intubation, mechanical ventilation or vasopressors for blood.


Listing 16.2.4.3 Pre-Injury Narrative - Baseline Status - Part 1

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Interview<br>Date/Time | Occupational Status | Social Skills |
|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | DDMONYYY | ********** | ********** |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.


## Listing 16.2.4.3 Pre-Injury Narrative - Baseline Status - Part 2

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Interview<br>Date/Time | Activities of Daily Living | Mode of Transportation |
|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | DDMONYYY | ********** | ******** |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.


## Listing 16.2.4.3 Pre-Injury Narrative - Baseline Status - Part 3

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Interview<br>Date/Time | General | Source of Information |
|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | DDMONYYY | ********** | (Patient alone, Relative/Friend/Caretaker Alone, Patient plus Relative/Friend/Caretaker, Medical Personnel) |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.



Listing 16.2.4.4 Glasgow Coma Scale

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Study Day | Date/<br>Time of<br>Assessment | Stop<br>Date/<br>Time | Not<br>Done? | Eye Opening <sup>2</sup> (none due to severe facial swelling/damage) | Verbal<br>Response <sup>3</sup><br>(none due<br>to<br>intubation) | Motor<br>Response <sup>4</sup> | GCS<br>Score | Assessed By?<br>If Other,<br>Specify | Did<br>Neurological<br>Worsening<br>Occur? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| внк-100 | xx-xxx | M/30/W | (Screening Post-Resuscitation, Day 1, Day 2, Day 3, Day 4, Day 5, Day 6 Day 15) | DDMONYYYY/<br>XX:XX | DDMONYYYY/<br>XX:XX | (yes,<br>no) | (SPON,<br>SPEECH,<br>PAIN,<br>NONE)<br>(no, yes) | (O,<br>C,<br>INAPP,<br>INCOMP,<br>NONE) | (OC,<br>LP,<br>WNF,<br>ABF,<br>ABE,<br>NONE) | xx | (Neurosurgeon,<br>ER Physician,<br>Intensivist,<br>Other<br>(specify)) | <del>(yes, no)</del> |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.

 $<sup>^{2}</sup>$  SPON=Spontaneous, SPEECH=In response to speech, PAIN=In response to pain, NONE=None.

<sup>&</sup>lt;sup>3</sup> O=Oriented, C=Confused, INAPP=Inappropriate words, INCOM=Incomprehensible sounds, NONE=None.

<sup>4</sup> OC=Obeys Commands, LP=Localizes Pain, WNF=Withdrawal/Normal flexion, ABF=Abnormal flexion, ABE=Abnormal Extension, NONE=None.

Listing 16.2.4.5 Medical History

| Treatment<br>Group | Subject No. | Sex/<br>Age/<br>Race <sup>1</sup> | Date of<br>Diagnosis | System | Diagnosis or<br>Abnormality | Diagnosis<br>Active? | End Date |
|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | DDMONYYYY | (Skin, HEENT, Respiratory,) | xxxxxxxxxxxx | (Yes, No) | (DDMONYYYY, or missing if diagnosis is active) |

...

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.



## Listing 16.2.4.6 Prior and Concomitant Medications

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Preferred Drug Name/<br>Medication Name | Dose Per<br>Frequency | Units | Frequency | Route | Start Date | Ongoing? | Stop Date | Indication | P/<br>C <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| внк-100 | xx-xxx | M/35/W | ************************************** | xx | (mg, g,, Other) | (Day,<br>Week,<br>Month, As<br>needed,<br>One time) | (PO,<br>SC,<br>IM,<br>IV,<br>Other) | DDMONYYYY | (Yes,<br>No) | DDMONYYYY (Stop date will be missing if medication ongoing.) | xxxxxxxxxx | С |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

<sup>&</sup>lt;sup>2</sup> P=Prior Medication, C=Concomitant Medication, P&C=Prior and Concomitant Medication.


## Listing 16.2.4.7 Concomitant Procedures

| Treatment Group | Subject No. | Sex/<br>Age/<br>Race <sup>1</sup> | Procedure Date | Procedure | Indication/Reason |
|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | DDMONYYYY<br>Procedure Date | xxxxxxxxxxxxxx | xxxxxxxxxxxxx |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.


## Listing 16.2.4.8 Surgical Therapy

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Date of Surgery | Type of Surgery | Specify | Repeat<br>Procedure? |
|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | DDMONYYYY | (Intracranial Surgery,<br>Extracranial Surgery) | ((Aneurysm) if Intracranial Surgery,<br>(Maxillofacial) if Extracranial<br>Surgery, or Specify if Other) | (Yes, No) |
| | | | | | (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.



## Listing 16.2.4.9 Study Admission

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Was Subject Transferred from Another Facility? | Admission to<br>First Facility<br>Date/Time | Admission at<br>Study Center<br>Date/Time |
|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | (yes, no) | DDMONYYYY/ XX:XX | DDMONYYYY/ XX:XX |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.



## Listing 16.2.4.10 Subject Transfer

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Initial<br>Site<br>Number | Initial<br>Subject<br>Number | New<br>Site<br>Number | New<br>Subject<br>Number | Date Subject<br>First Seen at<br>New Site | Type of Visit<br>(Specify) |
|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | XX | xx-xxx | XX | xx-xxx | DDMONYYYY | (Day, 15, Day 30, Day 90,<br>Day 180, Other) |
| | | | | | | | | (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.



Listing 16.2.4.11 Facility Transfer

| | | | Subject Discharged/Transfe | erred From | Subject Discharged/Transferred to | /Admitted To |
|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Specify | Date | Specify | Date |
| BHR-100 | xx-xxx | M/35/W | (ICU, General Ward, Nursing Home/Long-Term Care, Other ICU, Other Hospital, Rehabilitation Unit, Home, Other) | DDMONYYYY | (ICU, General Ward, Nursing<br>Home/Long-Term Care, Other ICU,<br>Other Hospital, Rehabilitation<br>Unit, Home, Other) | DDMONYYYY |
| | | | (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.




# Listing 16.2.4.12 Intubation

| Treatment Group | Subject No. | Sex/<br>Age/<br>Race <sup>1</sup> | Date/Time of Intubation | Date/Time of Extubation |
|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | DDMONYYYY/<br>XX:XX | DDMONYYYY/<br>XX:XX |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.


## Listing 16.2.4.13 Daily Fluid

| Treatment Group | Subject No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Collection<br>Period Start<br>Date/Time | Collection<br>Period Stop<br>Date/Time | Total Fluid<br>Administered<br>(ml) | Total Fluid<br>Excreted<br>(ml) |
|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | Day 1 | DDMONYYYY/<br>XX:XX | DDMONYYYY/<br>XX:XX | xxxxx.x | xxxxx.x |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.



## Listing 16.2.5.1 Study Drug Administration - Part 1

| Treat-<br>ment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Dose/<br>Day/<br>Bottle/<br>Record | Start Date/<br>Time | Stop Date/<br>Time | Route | Infusion<br>Rate<br>(ml/hr) |
|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | (Loading,<br>Maintenance)/1<br>/1/1 | DDMONYYYY/<br>XX:XX | DDMONYYYY/<br>XX:XX | (Central line,<br>Peripheral<br>line) | xxxxx.x |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.



 $a_{\overline{\text{Version Date: 2.0 April 19, 2014}}}$ 

## Listing 16.2.5.1 Study Drug Administration - Part 2

| | | | | | Infusion Rate | | Infusion Rate Intern | rupted |
|---|---|---|---|---|---|---|---|---|
| Treat-<br>ment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Dose/<br>Day/<br>Bottle/<br>Record | Modified? | Reason<br>If Other, Specify | For more than 30 mins? | Reason<br>If Other, specify | Duration (mins) |
| BHR-100 | xx-xxx | M/35/<br>W | (Loading,<br>Maintenan<br>ce)/1/1/1 | (Yes, No) | (Adverse Event, I.V. access problem,, Other) | (Yes, No) | (Adverse Event, I.V. access problem,, Other) | xxx |
| | | | | | (^^^^^^^^ | | (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.



#### Listing 16.2.5.2 End of Treatment

| Treat-<br>ment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Did the Subject<br>Complete 5 Days<br>of Treatment? | Date/Time<br>Infusion<br>Completed | If No, Reason for Discon-<br>tinuation of Study Drug<br>(If Other, Specify) | Treatment<br>Duration<br>(hours) <sup>2</sup> |
|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | (Yes, No) | DDMONYYYY | (Adverse Event, Death, PI Decision,<br>Sponsor Decision, Consent Withdrawn, Other) | xxx |
| | | | | | (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.

<sup>&</sup>lt;sup>2</sup> Duration of study drug exposure (in hours) = date:hour of last study medication administered - date:hour of first study medication administered + 1 - sum of recorded durations of infusion rate interruptions.



Listing 16.2.6.1.1 Glasgow Outcome Scale, Questions

| Question | Details and Possible Responses |
|---|---|
| 1 | Has the subject resumed pre-injury occupational status? Yes/No. |
| | [If subject resumed pre-injury occupational status is "Yes"] Check one box on the right A, B, C or D, that is most specific to the subject: |
| | A: Subject has resumed pre-injury employment: (e.g. executive or skilled laborer that has returned to the same level of responsibility at the same number of hours worked each week at the same performance level equivalent to that of their pre-injury status, with or without the use of compensatory mechanisms.) B: Subject could have resumed pre-injury occupational status, but currently has a reduction in performance level due to outlying circumstances that are not brain related: (e.g. previous work place out of business so they are unemployed and job hunting or a physical injury such as leg amputation that prevents them from returning to work - these are not "Brain Related Injuries" and should not be rated as a No for these types of reasons.) C: Subject has resumed academic pursuits: (e.g. a student has resumed the same number of hours/classes at the same performance level equivalent to that of their pre-injury abilities - independently, without the need for special accommodations such as tutors, if they were not necessary prior to the injury.) D: Subject has resumed household responsibilities: (e.g. a subject that was previously a housewife, househusband, unemployed and/or volunteer that has returned to the same level of responsibility, same number of hours involved at the same performance level equivalent to that of pre-injury.) |
| 2 | Has the subject resumed at least half as often as the pre-injury level of social activities? Yes/No. |
| 3 | Has the subject resumed pre-injury level of independence in activities of daily living? Yes/No. |
| 4 | Is the subject able to be left alone at home and is able to care for her/himself at the same level of pre-injury? Yes/No. |
| 5 | Has the subject resumed independence in transportation? Yes/No. |
| 6 | Does the subject respond to verbal communication and/or obey commands? Yes/No. |

 $a_{ ext{Version Date: 2.0 April 19, 2014}}$ 


Listing 16.2.6.1.2 Glasgow Outcome Scale, Explanation of Categories

| Explanation |
|-----------------------------------------------------------------|
| If you answered YES to ALL questions (1-6). |
| If you answered NO to questions 1 and 2 and YES to 3, 4, 5 & 6. |
| If you answered NO to questions 3, 4, or 5 and YES to 6. |
| If you answered NO to Question 6. |



Listing 16.2.6.1.3 Glasgow Outcome Scale - Extended, Explanation of Categories

| GOS-E | |
|---|---|
| Rating | Explanation |
| Upper<br>Good | Return to normal life and NO current problems relating to the injury that affect daily life (dizziness, headache, and sensitivity to noise or light, slowness, memory failure, concentration problems). |
| Lower<br>Good | Return to normal life BUT current problems relating to the injury that affect daily life (dizziness, headache, and sensitivity to noise or light, slowness, memory failure, concentration problems). Social Activities: Resumed at least half as often as pre-injury. Disruption or Strain: Occasional (less than once per week). |
| Upper<br>Moderate | Work capacity: Reduced<br>Social Activities: Resumed less than half as often as pre-injury<br>Disruption or Strain: Frequent (once a week or more but tolerable) |
| Lower<br>Moderate | Work capacity: Unable to work or only able to work in sheltered workshop<br>Social Activities: Unable or rarely able to participate<br>Disruption or Strain: Constant (daily and intolerable) |
| Upper<br>Severe | Care: Does not require someone to be around at home most of the time (for at least 8 hours during the day, if necessary) Travel: Unable to travel locally without assistance Shopping: Unable to shop without assistance |
| Lower<br>Severe | Care: Requires frequent help of someone to be around at home most of the time |



#### Listing 16.2.6.1.4 Glasgow Outcome Scale

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Month | Interview<br>Date | Source of<br>Information | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | GOS Rating | GOS -<br>Extended<br>Rating |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | (3,6) | DDMONYYY | (Patient Alone,<br>Relative/Friend/<br>Caretaker Alone,<br>) | (Yes:<br>(A,B,C,D)<br>or No) | (Yes,<br>No) | (Yes,<br>No) | (Yes,<br>No) | (Yes,<br>No) | (Yes,<br>No) | (Good<br>Recovery,<br>Moderate<br>Disability,<br>Severe<br>Disability,<br>Vegetative<br>State,<br>Dead) | (Upper<br>Good,<br>Lower<br>Good,<br>Upper<br>Moderate,<br>Lower<br>Moderate,<br>Upper<br>Severe,<br>Lower<br>Severe) |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

[Note to Programmer: Dead is not an option on the GOS CRF page. This information can be read from the mortality or date of death details (for premature terminations due to death). This information should be combined for the derived datasets.]



Listing 16.2.6.1.5 Glasgow Outcome Scale, Glasgow Outcome Scale-Extended Narrative - Part 1

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Month | Interview<br>Date | Occupational Status | Summarize Subjects<br>Work Capacity |
|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | (3,6) | DDMONYYY | ************ | (Returned to normal level,<br>Reduced, Only able to work<br>in sheltered work shop or<br>unable to work) |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.



Listing 16.2.6.1.5 Glasgow Outcome Scale, Glasgow Outcome Scale-Extended Narrative - Part 2

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Month | Interview<br>Date | Social Skills | Has the subject resumed pre-<br>injury level of social<br>activities? |
|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | (3,6) | DDMONYYY | ************ | (At least half as often,<br>Less than half as often,<br>Unable to or rarely<br>participate) |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.



## Listing 16.2.6.1.5 Glasgow Outcome Scale, Glasgow Outcome Scale-Extended Narrative - Part 3

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Month | Interview<br>Date | Disruption or Strain | Summarize the subject's extent of disruption or strain: |
|---|---|---|---|---|---|---|
| BHR-100 | xx-xx | M/35/W | (3,6) | DDMONYYY | ************ | (Occasional (less than once per week), Frequent (once per week or more but tolerable), Constant (daily and intolerable)) |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.



Listing 16.2.6.1.5 Glasgow Outcome Scale, Glasgow Outcome Scale-Extended Narrative - Part 4

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Month | Interview<br>Date | Activities of Daily Living | Are the family able to leave subject home alone for >= 8 hours/day, if necessary? |
|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | (3,6) | DDMONYYY | ************ | (yes, no) |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.



## Listing 16.2.6.1.5 Glasgow Outcome Scale, Glasgow Outcome Scale-Extended Narrative - Part 5

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Month | Interview<br>Date | Mode of Transportation | Is subject able to drive or use public transport without assistance? | Is subject able to shop without assistance? |
|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | (3,6) | DDMONYYY | ****** | (yes, no) | (yes, no) |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.



Listing 16.2.6.1.5 Glasgow Outcome Scale, Glasgow Outcome Scale-Extended Narrative - Part 6

| Treatment<br>Group | Subject | Sex/<br>Age/<br>Race <sup>1</sup> | Month | Interview<br>Date | General | Are there any problems e.g. dizziness, that affect daily life after the head injury? |
|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | (3,6) | DDMONYYY | ************ | (yes, no) |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

Listing 16.2.6.1.6 Primary Efficacy, Covariates, and Subgroup Variables (Observed Values)

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | GOS Rating<br>at Month 6 | Region | GCS<br>Motor<br>Score | Pupil<br>Response | CT<br>Classification | Time to First Dose Relative to TBI (Hours) | Baseline<br>Hypoxia | Baseline<br>Hypo-<br>tension | Traumatic<br>Sub-<br>arachnoid<br>Hemorrhage |
|---|---|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/35/W | (Good<br>Recovery,<br>Moderate<br>Disability,<br>Severe<br>Disability,<br>Vegetative<br>State) | (North<br>America,<br>Europe,<br>Asia and<br>South<br>America) | (1-2,<br>3, 4,<br>5-6) | (Bilateral,<br>Unilateral,<br>No Reactive<br>Pupils, Not<br>Testable) | (II, III, IV, evacuated/non-evacuated mass lesion) | (0-<=4, >4-<=8, >8) | (Yes,<br>No) | (Yes,<br>No) | (Yes, No) |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.

Program: xxxxxxx.sas, Output: xxxxxxx.rtf, Generated on: DDMONYYYY xx:xx, Page x of x

Repeat this shell for

Listing 16.2.6.1.7 Primary Efficacy, Covariates, and Subgroup Variables (Missing Values Imputed)

Add

Note: Missing values are first imputed by carrying forward the Month 3 GOS assessment. If a subject has neither the 3 nor the 6 month G OS, the missing value is imputed based upon the primary proportional odds model. Missing covariates are imputed as the most common level over all subjects.


## Listing 16.2.6.2 Sliding Dichotomy

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Prognosis Group | GOS Group<br>(4-level) | GOS Group<br>(2-level) |
|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | Month 6 | (Best,<br>Intermediate,<br>Worst) | (Good Recovery, Moderate Disability, Severe Disability, Vegetative State/Dead) | (Favorable,<br>Unfavorable) |

<sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.



## Listing 16.2.6.3 Mortality

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Status<br>(If Other, Specify) | Patient Residence | Date of Death or<br>Date of Last<br>Contact | Time to Death<br>or Last Contact<br>(days) <sup>2</sup> |
|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | Month 1 | (Lost to Follow-up,<br>Consent Withdrawn,<br>Alive, Dead, Other<br>[specify]) | (At Home, Hospital, Rehab Unit, Nursing Home/Long-Term Care, Other[Specify]) | DDMONYYY | XX* |
| | | | Month 6 | | | | |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.

<sup>&</sup>lt;sup>2</sup> If subject has not died, they will be censored on their last date of contact for the Kaplan-Meier survival analysis.

<sup>\*</sup> Indicates that time to death or last contact is censored.




 $a_{rac{}{ ext{Version Date: 2.0 April 19, 2014}}}$ 

# Listing 16.2.6.4.1 SF-36, Explanation of Categories

| Question | Explanation |
|---|---|
| 1. In general, would you say your health is: | 1=Excellent, 2=Very Good, 3=Good, 4=Fair, 5=Poor. |
| 2. Compared to one year ago, how would you rate your health in general now? | 1=Much better now than one year ago, 2=Somewhat better now than one year ago, 3=About the same as one year ago, 4=Somewhat worse now than one year ago, 5=Much worse now than one year ago. |
| 3. The following questions are about activities you might do during a typical day. Does your health now limit you in these activities? If so, how much? | |
| a. Vigorous activities | 1=Yes, limited a lot, 2=Yes, limited a little, 3=No, not limited at all |
| b. Moderate activities | 1=Yes, limited a lot, 2=Yes, limited a little, 3=No, not limited at all |
| c. Lifting or carrying groceries | 1=Yes, limited a lot, 2=Yes, limited a little, 3=No, not limited at all |
| d. Climbing several flights of stairs | 1=Yes, limited a lot, 2=Yes, limited a little, 3=No, not limited at all |
| e. Climbing one flight of stairs | 1=Yes, limited a lot, 2=Yes, limited a little, 3=No, not limited at all |
| f. Bending, kneeling, or stooping | 1=Yes, limited a lot, 2=Yes, limited a little, 3=No, not limited at all |
| g. Walking more than one mile | 1=Yes, limited a lot, 2=Yes, limited a little, 3=No, not limited at all |
| h. Walking several hundred yards | 1=Yes, limited a lot, 2=Yes, limited a little, 3=No, not limited at all |
| i. Walking one hundred yards | 1=Yes, limited a lot, 2=Yes, limited a little, 3=No, not limited at all |
| j. Bathing or dressing yourself | 1=Yes, limited a lot, 2=Yes, limited a little, 3=No, not limited at all |
| 4. During the past 4 weeks, have you had any of the following problems with your work or other regular daily activities as a result of your physical health? | |
| a. | 1=All of the time, 2=Most of the time, 3=Some of the time, 4=A little |
| | of the time, 5=None of the time |
| b. | 1=All of the time, 2=Most of the time, 3=Some of the time, 4=A little |
| | of the time, 5=None of the time |
| c. | 1=All of the time, 2=Most of the time, 3=Some of the time, 4=A little |
| | of the time, 5=None of the time |
| d. | 1=All of the time, 2=Most of the time, 3=Some of the time, 4=A little |
| | of the time, 5=None of the time |



 $a_{rac{-}{ ext{Version Date: 2.0 April 19, 2014}}}$ 

## Listing 16.2.6.4.1 SF-36, Explanation of Categories

| Question | Explanation |
|---|---|
| 5. During the past 4 weeks, how much of the time have you had any of the following problems with your work or other regular daily activities as a result of any emotional problems (such as feeling depressed or anxious)? | |
| <ul> <li>a. Cut down on the amount of time spent on work or other<br/>activities.</li> </ul> | 1=All of the time, 2=Most of the time, 3=Some of the time, 4=A little of the time, 5=None of the time |
| b. Accomplished less than you would like | 1=All of the time, 2=Most of the time, 3=Some of the time, 4=A little of the time, 5=None of the time |
| c. Did work or other activities less carefully than usual | 1=All of the time, 2=Most of the time, 3=Some of the time, 4=A little of the time, 5=None of the time |
| 6. During the past 4 weeks, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? | 1=Not at all, 2=Slightly, 3=Moderately, 4=Quite a bit, 5=Extremely |
| 7. How much bodily pain have you had during the past 4 weeks? | 1=None, 2=Very mild, 3=Mild, 4=Moderate, 5=Severe, 6=Very severe |
| 8. During the past 4 weeks, how much did pain interfere with your normal work (including both work outside the home and housework)? | 1=Not at all, 2=Slightly, 3=Moderately, 4=Quite a bit, 5=Extremely |



 $a_{rac{}{ ext{Version Date: 2.0 April 19, 2014}}}$ 

# Listing 16.2.6.4.1 SF-36, Explanation of Categories

| Question | Explanation |
|---|---|
| 9. These questions are about how you feel and how things have been with you during the past 4 weeks. For each question, please give the one answer that comes closest to the way you have been feeling. How much of the time during the past 4 weeks | |
| a. Did you feel full of life? | 1 = All of the time, $2 = Most$ of the time, $3 = Some$ of the time, $4 = A$ little of the time, $5 = None$ of the time |
| b. Have you been very nervous? | 1 = All of the time, $2 = Most$ of the time, $3 = Some$ of the time, $4 = A$ little of the time, $5 = None$ of the time |
| c. Have you felt so down in the dumps that nothing could<br>cheer you up? | 1 = All of the time, $2 = Most$ of the time, $3 = Some$ of the time, $4 = A$ little of the time, $5 = None$ of the time |
| d. Have you felt calm and peaceful? | 1 = All of the time, $2 = Most$ of the time, $3 = Some$ of the time, $4 = A$ little of the time, $5 = None$ of the time |
| e. Did you have a lot of energy? | 1 = All of the time, $2 = Most$ of the time, $3 = Some$ of the time, $4 = A$ little of the time, $5 = None$ of the time |
| f. Have you felt downhearted and depressed? | 1 = All of the time, $2 = Most$ of the time, $3 = Some$ of the time, $4 = A$ little of the time, $5 = None$ of the time |
| g. Did you feel worn out? | 1 = All of the time, $2 = Most$ of the time, $3 = Some$ of the time, $4 = A$ little of the time, $5 = None$ of the time |
| h. Have you been happy? | 1 = All of the time, $2 = Most$ of the time, $3 = Some$ of the time, $4 = A$ little of the time, $5 = None$ of the time |
| i. Did you feel tired? | 1 = All of the time, $2 = Most$ of the time, $3 = Some$ of the time, $4 = A$ little of the time, $5 = None$ of the time |
| 10. During the past 4 weeks, how much of the time has your physical health or emotional problems interfered with your social activities (like visiting friends, relatives, etc.)? | |
| 11. How TRUE or FALSE is each of the following statements for you? | |
| a. I seem to get sick a little easier than other people | <pre>1 = Definitely true, 2 = Mostly true, 3 = Don't know, 4 = Mostly false, 5 = Definitely false</pre> |
| b. I am as healthy as anybody I know | <pre>1 = Definitely true, 2 = Mostly true, 3 = Don't know, 4 = Mostly false, 5 = Definitely false</pre> |
| c. I expect my health to get worse | <pre>1 = Definitely true, 2 = Mostly true, 3 = Don't know, 4 = Mostly false, 5 = Definitely false</pre> |
| d. My health is excellent | <pre>1 = Definitely true, 2 = Mostly true, 3 = Don't know, 4 = Mostly false, 5 = Definitely false</pre> |



## Listing 16.2.6.4.2 SF-36 (Individual Questions) - Part 1

| | | | | | Q1 | Q2 | | | | | | Q3 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Interview<br>Date | | | a | b | С | d | е | f | g | h | i | j_ |
| BHR-100 | xx-xxx | M/39/W | Month 3 | DDMONYYYY | (1-5) | (1-5) | | | | | ( | 1-3) | | | | |
| | | | Month 6 | | | | | | | | | | | | | |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.



Listing 16.2.6.4.2 SF-36 (Individual Questions) - Part 2

| | | G / | | _ | | Q4Q5 | | | Q6 | Q7 | Q8 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Interview<br>Date | a | b | С | d | a | b | С | | | |
| BHR-100 | xx-xxx | M/39/W | Month 3 | DDMONYYYY | | | (1-5) | | | (1-5) | ) | (1-5) | (1-5) | (1-5) |
| | | | Month 6 | | | | | | | | | | | |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.



#### Listing 16.2.6.4.2 SF-36 (Individual Questions) - Part 3

| | | | | | | | | | Q9 | | | | | Q10 | | ( | 211 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Interview<br>Date | a | b | С | d | е | f | g | h | i | | a | b | С | d |
| BHR-100 | xx-xxx | M/39/W | Month 3 | DDMONYYYY | | | | | (1-5 | ) | | | | (1-5) | | (: | 1-5) | |
| | | | Month 6 | | | | | | | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.



## Listing 16.2.6.4.3 SF-36 (Scales and Summary Scores) - Part 1

| Treatment<br>Group | Subject No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Interview<br>Date | Vitality | Physical<br>Functioning | Bodily<br>Pain | General<br>Health<br>Perceptions | Physical Role<br>Functioning |
|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | Month 3 | DDMONYYYY | xxx | xxx | xxx | XXX | XXX |
| | | | Month 6 | | | | | | |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.


Listing 16.2.6.4.3 SF-36 (Scales and Summary Scores) - Part 2

| Treatment Group | Subject No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Interview<br>Date | Emotional<br>Role<br>Functioning | Social Role<br>Functioning | Mental<br>Health | Physical<br>Composite | Mental<br>Composite |
|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | Month 3 | DDMONYYYY | XXX | XXX | xxx | xxx | xxx |
| | | | Month 6 | | | | | | |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.



 $a_{rac{}{ ext{Version Date: 2.0 April 19, 2014}}}$ 

## Listing 16.2.6.5.1 CT Scan and Classification - Part 1

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit/<br>Date/<br>Time | Admission CT<br>Scan / If No,<br>Study Day | Number of<br>Parenchymal<br>Hemorrhage<br>Lesions | Subarachnoid<br>Hemorrhage/<br>If Yes,<br>Specify | Basal<br>Cisterns | Midline<br>Shift<br>Size<br>(mm) | Total Volume of Largest Lesion (ml) | Parenchymal<br>Hemorrhage/ If<br>Yes, ≥ 25 ml? |
|---|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xx | M/30/W | Screen-<br>Ing<br>DDMONYYYY/<br>XX:XX | (Yes, No) / x | xx | (Yes, No)/<br>(Basal,<br>Convexity) | (Present,<br>Compressed,<br>Absent) | xx | xxxx.xx | (Yes,No)/<br>(Yes,No) |
| | | | Day 6<br>DDMONYYYY/<br>XX:XX | | | | | | | |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.



 $a rac{}{ ext{Version Date: 2.0 April 19, 2014}}$ 

## Listing 16.2.6.5.1 CT Scan and Classification - Part 2

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit/<br>Date/<br>Time | Cerebral Contusion / If Yes, ≥ 25 ml? | Subdural<br>Hemorrhage/<br>If Yes, ≥<br>25 ml? | Epidural<br>Hemorrhage/<br>If Yes, ≥<br>25 ml? | Intraventricular<br>Hemorrhage/ If<br>Yes, ≥ 25 ml? | Small Slit<br>Ventricles | Cerebral<br>Edema | Pneumocephalus |
|---|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | R-100 xx-xxx | M/30/W | Screen-<br>Ing<br>DDMONYYYY/<br>XX:XX | (Yes,No)/<br>(Yes,No) | (Yes,No)/<br>(Yes,No) | (Yes, No)/<br>(Yes, No) | (Yes, No)/<br>(Yes, No) | (Yes, No) | (Yes,<br>No) | (Yes, No) |
| | | | Day 6<br>DDMONYYYY/<br>XX:XX | | | | | | | |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.



Listing 16.2.6.5.1 CT Scan and Classification - Part 3

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit/<br>Date/<br>Time | Other<br>Intracranial<br>Findings/<br>Specify | Skull<br>Fracture,<br>Depressed | Skull<br>Fracture,<br>Basilar | Skull Fracture,<br>Other / Specify | Evacuated Mass or<br>Plans to Evacuate | CT<br>Classification |
|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xx | M/30/W | Screen-<br>Ing<br>DDMONYYYY/<br>XX:XX | (Yes,No)/<br>xxxxxxxx | (Yes, No) | (Yes, No) | (Yes, No) / | (Yes, No) | (1,2 6) |
| | | | Day 6<br>DDMONYYYY/<br>XX:XX | | | | | | |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.


## Listing 16.2.6.5.2 CT Scan Comparison - Part 1

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Date of<br>Comparison <sup>2</sup> | Parenchymal<br>Hemorrhage | Cerebral<br>Contusion | Subdural<br>Hematoma | Epidural<br>Hematoma | Subarachnoid<br>Hematoma | Intraventricular<br>Hemorrhage | Progressive<br>Intracranial<br>Pathology (PIP) |
|---|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | DDMONYYYY | (Not Applica | ble, Improve | ed, Worsene | ed, New Fin | dings, No Chan | ge) | (Not Applicable, Same, Worsened, Improved) |
| | | | DDMONYYYY | | | | | | | |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.

<sup>&</sup>lt;sup>2</sup> CT scans will be compared to the screening CT scan.



 $\mathcal{I}_{\overline{ ext{Version Date: 2.0 April 19, 2014}}}$ 

## Listing 16.2.6.5.2 CT Scan Comparison - Part 2

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Date of<br>Comparison <sup>2</sup> | Small Slit<br>Ventricles | Cerebral<br>Edema | Midline<br>Shift | Pneumo-<br>cephalus | Other<br>Intracranial<br>Findings<br>(specify) |
|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | DDMONYYYY | (3 | | Improved, Worngs, No Change) | | (Not Applicable, Improved, Worsened, New Findings, No Change) |
| BHR-100 | xx-xxx | M/31/W | DDMONYYYY | | | | | |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.

 $<sup>^{2}</sup>$  CT scans will be compared to the screening CT scan.



## Listing 16.2.6.5.2 CT Scan Comparison - Part 3

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Date of<br>Comparison <sup>2</sup> | Skull Fracture,<br>Depressed | Skull Fracture,<br>Basilar | Skull Fracture,<br>Other |
|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | DDMONYYYY | (Not | Applicable, Improved,<br>New Findings, No Cha | |
| BHR-100 | xx-xxx | M/31/W | DDMONYYYY | | | |

<sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.

 $<sup>^{2}</sup>$  CT scans will be compared to the screening CT scan.

 $a \overline{a}$  Version Date: 2.0 April 19, 2014

Listing 16.2.6.6.1 Intracranial Pressure

| Treatment Group | Subject No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Date | Time | Value |
|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | Screening | DDMONYYYY | xx.xx | xxx |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.



## Listing 16.2.6.6.2 Intracranial Pressure Monitoring

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Date/Time<br>ICP<br>Monitor<br>Placed | Device Used<br>(If Other, Specify) | End<br>Date/Time<br>ICP<br>Monitoring | Reason for Ending<br>ICP Monitoring<br>(If Other, Specify) |
|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | DDMONYYYY/<br>XX:XX | (Ventriculostomy,<br>Intraparenchymal, Epidural,<br>Subdural, Other) | DDMONYYYY/<br>XX:XX | (Clinically no longer required,<br>Monitor/catheter failure, Patient<br>considered unsalvageable, Patient<br>died, Other) |
| | | | | (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.



## Listing 16.2.6.7 Cerebral Perfusion Pressure

| Treatment Group | Subject No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Date | ICP<br>(mmHg) | Highest/<br>Lowest<br>ICP? | Pulse<br>Rate<br>(bpm) | Systolic<br>Blood<br>Pressure<br>(mmHg) | Diastolic<br>Blood<br>Pressure<br>(mmHg) | CPP<br>(mmHg) |
|---|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | Screen-<br>ing | DDMONYYYY | XXX | (H, L) | XXX | XXX | XXX | XXX |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.



Listing 16.2.6.8.1 Therapy Intensity Level - Part 1

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Date/<br>Time/<br>ICP <sup>2</sup> | Sedation | Paralysis<br>Induction | Ventricular<br>Drainage | Mannitol | Hypertonic<br>Saline |
|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | Screening | DDMONYYYY/<br>XX:XX/<br>(H, L, UNK) | (Yes, No) | (Yes, No) | (Yes, No) | (Yes, No) | (Yes, No) |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.

<sup>&</sup>lt;sup>2</sup> Was TIL recorded at highest (H), lowest (L) or unknown (UNK) ICP value. The therapies taken each study day through to day 6 can continue to be monitored after the ICP monitor is removed. For such cases the ICP measurement would be unknown.



## Listing 16.2.6.8.1 Therapy Intensity Level - Part 2

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Date/<br>Time/<br>ICP <sup>2</sup> | Pressor<br>Administration | Hyper-<br>ventilation | Hypothermia<br>for ICP<br>Reduction | Barbiturate<br>Induced<br>Coma | Surgical<br>Decompression | TIL<br>Score |
|---|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | Screening | DDMONYYYY/<br>XX:XX/<br>(H, L, UNK) | (Yes, No) | (Yes, No) | (Yes, No) | (Yes, No) | (Yes, No) | Х |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.

<sup>&</sup>lt;sup>2</sup> Was TIL recorded at highest (H), lowest (L) or unknown (UNK) ICP value. The therapies taken each study day through to day 6 can continue to be monitored after the ICP monitor is removed. For such cases the ICP measurement would be unknown.



#### Listing 16.2.7 Adverse Events

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Adverse Event/<br>Preferred Term/<br>SOC | Start Date/<br>Stop Date/<br>Day <sup>2</sup> / | Duration <sup>3</sup> /<br>Length of<br>Exposure<br>(hours) <sup>4</sup> | Intensity/<br>Relationship/<br>Outcome <sup>5</sup> | Action<br>Taken<br>with Study<br>Drug <sup>6</sup> | Treatment<br>for<br>AE?<br>(specify) <sup>7</sup> | Serious?/<br>(Reason for<br>Seriousness <sup>8</sup><br>)/<br>Treatment<br>Emergent? <sup>9</sup> |
|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | xxxxxxxxxxxx/<br>Xxxxxxxxxxxx/<br>xxxxxxxxxxx | DDMONYYYY/<br>DDMONYYYY/<br>xx | x/<br>x.xx | xxxxxxx/<br>x/<br>x | х | xxx/<br>(x) | xxx (xxx)/<br>xx |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.

<sup>&</sup>lt;sup>2</sup> Day is relative to the start date of study medication, event start date - administration start date + 1 if event start date is on or after the date of the start of study medication administration or event start date - administration start date if event date is before the date of the start of study medication administration.

<sup>&</sup>lt;sup>3</sup> Length of exposure is based on administration start date and administration end date during the study (end date - start date + 1).

<sup>&</sup>lt;sup>4</sup> Duration = AE end date - AE start date + 1.

<sup>&</sup>lt;sup>5</sup> Relationship: 1=Not related, 2=Possibly related, 3=Probably related, 4=Related. Outcome: 1=Recovered/resolved, 2=Recovering/resolving, 3=Not recovered/not resolved, 4=Recovered/resolved with sequelae, 5=Fatal, 6=Unknown.

<sup>6 1=</sup>Dose not changed, 2=Drug withdrawn, 3=Drug interrupted, 4=Dose reduced, 5=Dose increased, 6=Unknown, 7=Not applicable.

<sup>1 1=</sup>none, 2=Change in therapy intensity level, 3=procedure/surgery, 4=other (specify).

<sup>&</sup>lt;sup>8</sup> 1=Results in death, 2=Life threatening, 3=Results in persistent or significant disability/incapacity, 4=Requires or prolongs hospitalization, 5=Congenital abnormality/birth defect, 6=Other medically important event.

<sup>&</sup>lt;sup>9</sup> Treatment-emergent adverse events are defined as events that start on or after the first dose of study medication and up to 15 days and 6 months after the initiation of study treatment, for adverse events and serious adverse events respectively.

Listing 16.2.8.1.1 Laboratory (Coagulation) Results

| | | Sex/ | | | Sample | | Change | | Referen | nce Range | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject<br>No. | Age/<br>Race <sup>1</sup> | Test Name | Visit | Date/<br>Time | Result<br>(Unit) | from<br>Baseline | Range<br>Flag² | Low | High | Clin Sig? | Is this<br>an AE? |
| BHR-100 | xx-xxx | M/35/W | INR | Screening | DDMONYYYY/<br>XX:XX | xx.x g/L | xx.x | L | XX.X | xx.x | (Yes, No) | (Yes,<br>No) |
| | | | | Day 6 | DDMONYYYY/<br>XX:XX | xx.x g/L | xx.x | L | XX.X | XX.X | | |
| | | | | Day 15 | DDMONYYYY/<br>XX:XX | xx.x g/L | XX.X | L | XX.X | XX.X | | |
| | | | | | XX:XX | | | | | | | |

Note: The baseline value is defined as the last measurement taken prior to first administration of study drug (Day 1). For laboratory assessments this will be the screening visit.

[Note to Programmer: Do not include unscheduled results in this listing.]

<sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.  $^2$  N = Normal, L = Low, H = High.

[Use shell for Listing 16.2.8.1.1]


Listing 16.2.8.1.2 Laboratory (Hematology) Results
(Produce for Hemoglobin, Hematocrit, RBC, Reticulocyte Count, Platelet Count, WBC, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils)
Listing 16.2.8.1.3 Laboratory (Serum Chemistry) Results
(Produce for Sodium, Potassium, Chloride, Cholesterol, total, Triglycerides, ALT, AST, GGT, Alkaline Phosphatase, Total Protein, Glucose)
Listing 16.2.8.1.4 Laboratory (Urinalysis) Results
(Produce for pH, Specific Gravity, Protein, Glucose, Blood, WBC, RBC, Casts, Epithelial Cells, Bacteria)



Listing 16.2.8.1.5 Laboratory (Pregnancy Test) Results

| | | Sex/<br>Age/<br>Race <sup>1</sup> | Is Subject<br>Female of<br>Child-bearing<br>Potential? | If, Yes | | | |
|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject No. | | | Was Sample<br>Collected for<br>Pregnancy Test? | Pregnancy<br>Test Type | Date of<br>Collection | Pregnancy Test<br>Result |
| BHR-100 | xx-xxx | M/35/W | (yes, no) | (yes, no) | (Serum, Urine) | DDMONYYYY | (Positive,<br>Negative) |

...

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black, African American or of African Heritage, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, Z=Not Allowed to Obtain, O = Other.



## Listing 16.2.8.2 Vital Signs

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Date/Time | Pulse<br>Rate<br>(bpm) | Resp<br>Rate<br>(bpm) | SBP<br>(mmHg) | DBP<br>(mmHg) | Temp<br>(°C) | Weight<br>(kg) | Right<br>Pupil <sup>2</sup> | Left<br>Pupil <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | Screen-<br>ing | DDMONYYYY/<br>XX:XX | xxx | xx | xxx | xxx | xx.x | XX | (R,<br>NR,<br>UN) | (R,<br>NR,<br>UN) |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.

<sup>&</sup>lt;sup>2</sup> R=Reacts, NR=No Reaction, UN=Eyes Closed/Untestable.



aarrowsign Version Date: 2.0 April 19, 2014

## Listing 16.2.8.3 Physical Examinations

| Treatment<br>Group | Subject No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Date Exam<br>Performed | Body System | Status | Abnormalities |
|---|---|---|---|---|---|---|---|
| BHR-100 | xx-xxx | M/30/W | Screen-<br>ing | DDMONYYYY | Skin | Normal | |
| | | | | | HEENT | Abnormal | xxxxxxxxxxxxxxxxx |
| | | | | | Respiratory | Not Done | |
| | | | | | Cardiovascular | Not Done | |
| | | | | | Abdomen | Normal | |
| | | | | | Musculoskeletal | Normal | |
| | | | | | Neurological | Normal | |
| | | | | | Gastrointestinal | Normal | |
| | | | | | Genitourinary | Normal | |
| | | | | | Endocrine | | |
| | | | | | Lymph Nodes | | |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.



 $a ag{Version Date: 2.0 April 19, 2014}$ 

## Listing 16.2.8.4 12-Lead Electrocardiogram (ECG) - Part 1

| | | | | | Rhythm | | | | Conduction | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Heart<br>Rate<br>bpm) | Result | Specify | Clin<br>Sig | Result | Specify | Clin<br>Sig | QT<br>Prolongation<br>Interval |
| BHR-100 | xxx- | M/30/W | Screening | xx | (Normal,<br>Abnormal) | (Sinus Arrhythmia,, Other Arrhythmia [xxxxxxx]) | (Yes,<br>No) | (Normal,<br>Abnormal) | (LBBB,,<br>Other<br>[xxxxxx]) | (Yes,<br>No) | xxx |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.


## Listing 16.2.8.4 12-Lead Electrocardiogram (ECG) - Part 2

| | | Sex/ | | | QRS Complex | | _ |
|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject<br>No. | Age/<br>Race <sup>1</sup> | Visit | Result | Specify | Clin Sig | Comments |
| BHR-100 | xxx-xxxx | M/30/W | Screening | (Normal,<br>Abnormal) | (Non-specific ST changes,, other [xxxxx]) | (Yes,<br>No) | ****** |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.


## Listing 16.2.8.5 Arterial Blood Gas

| Treatment<br>Group | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Date/<br>Time | Line | рН | $PaCO_2$ (mmHg) | HCO <sub>3</sub> (mmol/L) | SaO <sub>2</sub> (%) | PaO <sub>2</sub><br>(mmHg) | FiO <sub>2</sub> (%) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| внк-100 | xx-xxx | M/30/W | Screening | DDMONYYYY/<br>XX:XX | (1.1,<br>2.2,<br>3.3,<br>4.4,<br>5.5,<br>6.6) | x.xx | xxx.x* | ххх.х | xxx.x | xxx.x | xx.xx* |

 $<sup>^{1}</sup>$  M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.

 $<sup>\</sup>mbox{\ensuremath{^{\star}}}$  Indicates the worst value of the day for a given parameter.



Listing 16.2.8.6 Neuroworsening - Part 1

| | | | | Ne | uroworsening | ? | | | or Neurolog | ic Worsenin | g | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Subject<br>No. | Sex/<br>Age/<br>Race <sup>1</sup> | Visit | Start<br>Date/<br>Time | Stop<br>Date/<br>Time | Contin-<br>uing? | Eye Opening <sup>2</sup> (none due to severe facial swelling/damage) | Verbal Response <sup>3</sup> (none due to intubation) | Motor<br>Response <sup>4</sup> | Right<br>Pupil<br>React-<br>ivity <sup>5</sup> | Left<br>Pupil<br>React-<br>ivity <sup>5</sup> | ICP(mmHg)/<br>SBP (mmHg)/<br>DBP (mmHg) |
| BHR-100 | xx-xxx | M/30/W | Day 1 | DDMONYYYY/<br>XX:XX | DDMONYYYY/<br>XX:XX | (yes, no) If no, a stop date should be provided in the previous column. | (SPON,<br>SPEECH,<br>PAIN,<br>NONE)<br>(no, yes) | (O,<br>C,<br>INAPP,<br>INCOMP,<br>NONE)<br>(yes, no) | (OC,<br>LP,<br>WNF,<br>ABF,<br>ABE,<br>NONE) | (R,<br>NR,<br>UN) | (R,<br>NR,<br>UN) | xxx/<br>xxx/<br>xxx |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.

<sup>&</sup>lt;sup>2</sup> SPON=Spontaneous, SPEECH=In response to speech, PAIN=In response to pain, NONE=None.

<sup>&</sup>lt;sup>3</sup> O=Oriented, C=Confused, INAPP=Inappropriate words, INCOM=Incomprehensible sounds, NONE=None.

<sup>4</sup> OC=Obeys Commands, LP=Localizes Pain, WNF=Withdrawal/Normal flexion, ABF=Abnormal flexion, ABE=Abnormal Extension, NONE=None.

<sup>&</sup>lt;sup>5</sup> R=Reacts, NR=No Reaction, UN=Untestable.



Listing 16.2.8.6 Neuroworsening - Part 2

| ubject | Sex/<br>Age/<br>Race <sup>1</sup> | Start<br>Date/<br>Time | Eye Opening <sup>2</sup> (none due to severe facial swelling/damage) | Verbal Response <sup>3</sup> (none due to intubation) | Motor<br>Response <sup>4</sup> | Right<br>Pupil<br>React-<br>ivity | Left<br>Pupil<br>React-<br>ivity | ICP(mmHg)/<br>SBP (mmHg)/<br>DBP (mmHg) | Primary Reason<br>for Deterioration<br>(If Other, Specify) |
|---|---|---|---|---|---|---|---|---|---|
| x-xxx | M/30/W | DDMONYYYY/<br>XX:XX | (SPON,<br>SPEECH,<br>PAIN,<br>NONE) | (O,<br>C,<br>INAPP,<br>INCOMP,<br>NONE) | (OC,<br>LP,<br>WNF,<br>ABF,<br>ABE, | (R,<br>NR,<br>UN) | (R,<br>NR,<br>UN) | xxx/<br>xxx/<br>xxx | (Increased Intracranial Volume Cerebral Ischemia, Seizures, Systemic Complication, Other [xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| 0 | • | bject Age/<br>. Race <sup>1</sup> | bject Age/ Date/ . Race¹ Time -xxx M/30/W DDMONYYYY/ | Sex/ Start (none due to bject Age/ Date/ severe facial swelling/damage) -xxx M/30/W DDMONYYYY/ (SPON, XX:XX SPEECH, PAIN, | Sex/ Start (none due to (none due bject Age/ Date/ severe facial to swelling/damage) intubation) -xxx M/30/W DDMONYYYY/ (SPON, (O, XX:XX SPEECH, C, PAIN, INAPP, NONE) INCOMP, NONE) | Sex/ Start (none due to (none due bject Age/ Date/ severe facial to Motor Race¹ Time swelling/damage) intubation) Response⁴ -xxx M/30/W DDMONYYYY/ (SPON, (O, (OC, XX:XX SPEECH, C, LP, PAIN, INAPP, WNF, NONE) INCOMP, ABF, NONE) ABE, | Sex/ Start (none due to (none due pupil bject Age/ Date/ severe facial to Motor React- Race¹ Time swelling/damage) intubation) Response⁴ ivity -xxx M/30/W DDMONYYYY/ (SPON, (O, (OC, (R, XX:XX SPEECH, C, LP, NR, PAIN, INAPP, WNF, UN) NONE) INCOMP, ABF, NONE) ABE, | Sex/ Start (none due to (none due Pupil Pupil bject Age/ Date/ severe facial to Motor React- React- Race¹ Time swelling/damage) intubation) Response⁴ ivity ivity -xxx M/30/W DDMONYYYY/ (SPON, (O, (OC, (R, (R, XX:XX SPEECH, C, LP, NR, NR, PAIN, INAPP, WNF, UN) UN) NONE) INCOMP, ABF, NONE) ABE, | Sex/ Start (none due to (none due Pupil Pupil ICP(mmHg)/ bject Age/ Date/ severe facial to Motor React- React- SBP (mmHg)/ . Race¹ Time swelling/damage) intubation) Response⁴ ivity ivity DBP (mmHg) -xxx M/30/W DDMONYYYY/ (SPON, (O, (OC, (R, (R, xxx/ XX:XX SPEECH, C, LP, NR, NR, xxx/ PAIN, INAPP, WNF, UN) UN) xxx NONE) INCOMP, ABF, NONE) ABE, |

<sup>&</sup>lt;sup>1</sup> M = Male, F = Female; W = White, B = Black or African American, P = Native Hawaiian or Other Pacific Islander, A = Asian, N = American Indian or Alaska Native, O = Other.

<sup>&</sup>lt;sup>2</sup> SPON=Spontaneous, SPEECH=In response to speech, PAIN=In response to pain, NONE=None.

<sup>&</sup>lt;sup>3</sup> O=Oriented, C=Confused, INAPP=Inappropriate words, INCOM=Incomprehensible sounds, NONE=None.

<sup>4</sup> OC=Obeys Commands, LP=Localizes Pain, WNF=Withdrawal/Normal flexion, ABF=Abnormal flexion, ABE=Abnormal Extension, NONE=None.

<sup>&</sup>lt;sup>5</sup> R=Reacts, NR=No Reaction, UN=Untestable.